# IPX203 (CARBIDOPA-LEVODOPA) EXTENDED-RELEASE CAPSULES

# IPX203-B16-02

# A RANDOMIZED CONTROLLED STUDY TO COMPARE THE SAFETY AND EFFICACY OF IPX203 WITH IMMEDIATE-RELEASE CARBIDOPALEVODOPA IN PARKINSON'S DISEASE PATIENTS WITH MOTOR FLUCTUATIONS

#### SPONSOR

Impax Laboratories, LLC 400 Crossing Boulevard, Third Floor Bridgewater, NJ 08807-2863

Original Protocol, May 18, 2017 Amendment 1, August 30, 2017 Amendment 2, October 23, 2017 Amendment 3, December 07, 2017 Amendment 4, September 28, 2018

#### CONFIDENTIALITY STATEMENT

All information provided is the property of Impax Laboratories, LLC and may not be divulged, published or otherwise disclosed without written consent of Impax. All information provided to the Investigator by the Sponsor, including clinical observations at the investigative site, shall be held strictly confidential and confined to the clinical personnel involved in conducting the study, under the supervision of the Investigator. This includes but is not limited to preclinical data, protocols, case report forms, and verbal or written communications. This information may be related in confidence to the Institutional Review Board or other committees functioning in a similar capacity. All reports, subject samples, data published or submitted to third parties will be identified by a coded number and initials only in order to maintain subject confidentiality.

#### SIGNATURE PAGE



Principal Investigator's printed name

# **INVESTIGATOR'S AGREEMENT**

| Protocol No.: | IPX203-B16-02 | | |
|---|---|---|---|
| Protocol Title: | Protocol Title: A Randomized Controlled Study to Compare the Safety and Efficacy of IPX203 with Immediate-Release Carbidopa-Levodopa in Parkinson's Disc Patients with Motor Fluctuations | | |
| obligations and re | equirements of clinical investi<br>armonization (ICH), Good Cli | the study as outlined herein, complying with igators and all other requirements of International Practice (GCP), and the appropriate | |
| me who assist in | the conduct of this clinical sture fully informed regarding the | rtinent information to all individuals responsible. I will discuss this material with them to the study medication, the conduct of the study | 0 |
| Principal Investig | ator's signature | <br>Date | |
| | | 2 | |

# STUDY CONTACT INFORMATION

Changes in Impax study personnel listed on this page do not require a protocol amendment.

| Role | Name and Contact Information |
|---|---|
| Sponsor | Impax Laboratories, LLC<br>400 Crossing Boulevard, Third Floor<br>Bridgewater, NJ 08807-2863<br>(732) 595-4600 |
| Medical Monitor | |
| Statistician | |
| Clinical Pharmacology | |
| Clinical Research Associates | |
| Serious Adverse Event<br>Reporting | FAX: (866) 954-2064 |

#### 1. SYNOPSIS

Name of Sponsor/Company: Impax Laboratories, LLC (Impax)

Name of Investigational Product: IPX203 (carbidopa-levodopa) Extended-Release Capsules

Name of Active Ingredients: carbidopa (CD), levodopa (LD)

**Protocol Title:** A Randomized Controlled Study to Compare the Safety and Efficacy of IPX203 with Immediate-Release Carbidopa-Levodopa in Parkinson's Disease Patients with Motor Fluctuations

Protocol No.: IPX203-B16-02
Study center(s): Multicenter

**Phase of Development:** Phase 3

**Objectives:** To evaluate the safety and efficacy of IPX203 in comparison to IR CD-LD in the treatment of CD-LD-experienced subjects with Parkinson's disease (PD) who have motor fluctuations.

**Methodology:** This is a multicenter, randomized, double-blind, double-dummy, active-controlled, parallel-group study. The study will consist of a 3-week, open-label IR CD-LD dose adjustment period; a 4-week, open-label period for conversion to IPX203; followed by a 13-week double-blind treatment period with subjects randomized in a 1:1 ratio, stratified by center, to receive either IPX203 (with matching IR CD-LD placebo) or IR CD-LD (with matching IPX203 placebo).

Subjects will continue to take permitted non-CD-LD-based PD medications throughout the study if documented in their prestudy regimen and if dosing regimens have been stable for at least 4 weeks prior to Visit 1. A "stable dosing regimen" means no change in dose or in dosing frequency.

- Within 4 weeks following the Screening visit, eligible subjects will complete their PD Diaries on each of the 3 consecutive days immediately prior to Visit 1.
- Following Visit 1, qualified subjects will enter a 3-week, open-label IR CD-LD treatment period allowing for dose adjustment. The dosing regimen of IR CD-LD may be adjusted during the dose adjustment period to minimize "Off" time without causing troublesome dyskinesia. The doses and regimens of the subject's other non-CD-LD PD medications (dopamine agonists, MAO-B inhibitors, amantadine, anticholinergics) should remain stable throughout this study. Any adjustments to the IR CD-LD dosing regimen will be done in consultation with the Investigator or qualified site personnel and will be recorded. The IR CD-LD dosing regimen should be stable for at least 5 days prior to returning for Visit 2. Rescue with additional or modified doses of concomitant PD medications or with use of CD-LD products other than the dispensed study medications is not permitted and will trigger discontinuation from the study. Subjects will complete their 3-day PD Diaries on each of the 3 consecutive days immediately prior to Visit 2.
- Following completion of the IR CD-LD dose adjustment period, subjects will begin a 4-week open-label period for conversion to IPX203. The initial dosing regimen of IPX203 will be based on the most frequent dose of the subject's dosing regimen of IR CD-LD at the end of the dose adjustment period (Visit 2). A 25-100 mg dose of IR CD-LD converts to a 70-280 mg CD-LD dose of IPX203 (2 capsules of 35-140 mg CD-LD IPX203), and a 12.5-50 mg dose of IR CD-LD converts to a 35-140 mg CD-LD dose of IPX203, but with a longer duration of effect. It is recommended that IPX203 should be dosed approximately every 8 hours with the exception that subjects who are currently receiving a total daily dose of less than 125-500 mg IR CD-LD at the end of the dose adjustment period will be initially administered every

12 hours. The dosing interval may be reduced to approximately every 8 hours if the subject does not achieve an acceptable duration of effect. The dosing regimen of IPX203 may be adjusted during the dose conversion period to achieve the optimal balance of efficacy and tolerability (minimize "Off" time without causing troublesome dyskinesia or other dopaminergic side effects). The doses and regimens of the subject's other non-CD-LD PD medications (dopamine agonists, MAO-B inhibitors, amantadine, anticholinergics) should remain stable throughout this study. The subject must be on a stable dosing regimen of IPX203 (no change in dose or in dosing frequency) for at least 5 days prior to returning for Visit 4. Any adjustments to the IPX203 dosing regimen will be done in consultation with the Investigator or qualified site personnel and will be recorded. Rescue with additional or modified doses of concomitant PD medications or with use of CD-LD products other than the dispensed study medications is not permitted and will trigger discontinuation from the study. Subjects will return to the clinic in 2 weeks for Visit 3 followed by Visit 4, 2 weeks later. Subjects will complete their 3-day PD Diaries on each of the 3 consecutive days immediately prior to Visit 4.

• Subjects who successfully complete the IPX203 dose conversion period will be randomized in 1:1 ratio, stratified by center, at Visit 4 into one of two parallel treatment arms of IPX203 (with matching IR CD-LD placebo) or IR CD-LD (with matching IPX203 placebo). The subjects will undergo 13 weeks of double-blind maintenance therapy with the stable dosing regimen established at the end of Week 3 (Visit 2) for IR CD-LD and at the end of Week 7 (Visit 4) for IPX203. Rescue with additional or modified doses of concomitant PD medications or with use of CD-LD products other than the dispensed study medications is not permitted and will trigger discontinuation from the study. Subjects will return to the clinic for 3 visits (Visits 5, 6, and 7) and will complete their 3-day PD Diaries on each of the 3 consecutive days immediately prior to each of these visits.

**Number of patients (planned):** Assuming approximately an 18% prerandomization drop-out, approximately 510 subjects will be enrolled to randomize 420 subjects.

#### Diagnosis and main criteria for inclusion:

#### Inclusion Criteria

- Male or female subjects diagnosed at age ≥ 40 years with PD, consistent with the United Kingdom Parkinson's Disease Society Brain Bank Diagnostic Criteria and who are being treated with stable regimens of CD-LD but experiencing motor fluctuations.
- Hoehn and Yahr Stages 1, 2, 3, or 4 in the "On" state (part of Movement Disorders Society version of the Unified Parkinson's Disease Rating Scale [MDS-UPDRS] Part III)
- Montreal Cognitive Assessment (MoCA) score ≥ 24 at Screening Visit in "On" state.
- By history, for the 4 weeks prior to Screening, the subject experiences daily "wearing-off" episodes with periods of bradykinesia in combination with at least one of rest tremor or rigidity, experiences an "Off" state upon awakening on most mornings, and reports an average of at least 2.5 cumulative hours per day of "Off" time during the waking hours.
- Able to differentiate "On" state from "Off" state as determined by at least 75% concordance with a
  trained rater in "On/Off" ratings for 8 ratings over a 4-hour training period. The concordance must
  include at least 1 "On" and 1 "Off" rating and must be achieved within two 4-hour training
  sessions.
- At Visit 1, review of the 3-day PD Diaries confirms the following: that the subject is able to properly complete the Diaries with valid entries; and that the subject has an <u>average of at least 2.5 hours</u> per day of "Off" time during waking hours over the 3 days with at least 1.5 hours of cumulative "Off" time on each day.

- Responsive to CD-LD therapy and currently being treated on a stable regimen with CD-LD for at least 4 weeks prior to Visit 1 and:
  - Requires at least 100 mg of LD from IR CD-LD for the first morning dose
  - Requires a total daily dose of at least 400 mg of LD and takes a maximum total daily dose of 2400 mg LD, from IR CD-LD alone or IR CD-LD in combination with a single daily bedtime dose of CR CD-LD
  - Has a dosing frequency of 4 to 9 times daily of CD-LD
  - By history, typically experiences an "On" response with the first dose of IR CD-LD of the day, but the efficacy of this dose typically lasts less than 4 hours.
- At Screening, the subject has predictable "Off" periods defined by a score of 1 or 2 on Item #4.5 (Complexity of Motor Fluctuations) of the MDS-UPDRS Part IV B (Motor Fluctuations).
- At Screening, the MDS-UPDRS Part III total score in the "Off" state is at least 20 units.

#### **Exclusion Criteria**

- Used any doses of controlled-release (CR) CD-LD apart from a single daily bedtime dose within 4 weeks prior to Visit 1.
- Used any dose of Rytary for the past 4 weeks prior to Visit 1 or were considered IPX066 or Rytary failures for reasons of efficacy or safety.
- Had prior neurosurgical treatment for PD or if such procedure is planned or anticipated during the study period.
- Allergic to any excipient in the study drugs.
- History of glaucoma with intraocular pressures that are elevated despite appropriate medical management.
- History of seizure or epilepsy and experienced at least 1 seizure during the past 12 months or has not been compliant with medically recommended therapy or visits.
- History of myocardial infarction with residual atrial, nodal, or ventricular arrhythmias that are not
  controlled with medical and/or surgical interventions. A recent (≤ 12 months) history of
  myocardial infarction with secondary arrhythmias is exclusionary regardless of the therapeutic
  control.
- Received within 4 weeks of Screening or planning to take during participation in the clinical study:
  - Any doses of a CR CD-LD apart from a single daily bedtime dose, any doses of Rytary, additional CD (eg, Lodosyn) or benserazide (eg, Serazide), or catechol-O-methyl transferase inhibitors (entacapone or tolcapone) or medications containing these inhibitors (Stalevo),
  - Nonselective monoamine oxidase inhibitors (MAOI), apomorphine, or antidopaminergic agents, including antiemetics.
- Subjects who have previously participated in an IPX203 study.

**Investigational product, dosage and mode of administration:** IPX203 (carbidopa-levodopa) Extended-Release capsules, containing 35-140 mg of CD-LD and matching placebo, for oral administration.

**Reference therapy, dosage and mode of administration:** Immediate-Release carbidopa-levodopa (IR CD-LD) tablets containing 25-100 mg of CD-LD, and matching placebo, for oral administration.

**Duration of treatment:** Approximately 24 weeks, including up to 4 weeks following Screening, 3 weeks of IR CD-LD dose adjustment, 4 weeks of IPX203 dose conversion, and 13 weeks of double-

blind therapy following randomization.

#### Criteria for evaluation:

Baseline is defined as assessments done at Visit 4 (randomization visit). Study Entry is defined as assessments done at Visit 1 (study entry visit).

#### Efficacy:

- Primary endpoint: Change from baseline in "Good on" time in hours per day, averaged over the PD Diary days, at the end of double-blind treatment period (Visit 7 or early termination). "Good on" time is derived from the 3-day PD Diaries and is defined as the sum of "On" time without dyskinesia and "On" time with nontroublesome dyskinesia.
- · Key secondary endpoints:
  - Change from baseline in "Off" time in hours per day, averaged over the PD Diary days at the end of double-blind treatment period (Visit 7 or early termination)
  - Proportion of subjects with either "much improved" or "very much improved" in Patient Global Impression of Change (PGI-C) scores at the end of double-blind treatment period (Visit 7 or early termination)
  - Change from baseline in the MDS-UPDRS Part III at the end of double-blind treatment period (Visit 7 or early termination)
  - Change from baseline in the sum of MDS-UPDRS Parts II and III at the end of doubleblind treatment period (Visit 7 or early termination)
- Additional endpoints:

The following endpoints will be evaluated (at the post-randomization visits) as change from baseline (Visit 4) as well as change from the study entry (Visit 1), when applicable, by visits:





 Safety: electrocardiograms (ECGs), clinical laboratory tests, physical examinations, Columbia-Suicide Severity Rating Scale (C-SSRS), and supine and standing orthostatic vital signs; adverse events and concomitant medications evaluated throughout the course of the study.

**Statistical methods:** For the primary endpoint, assuming a difference of 1 hour between IPX203 and IR CD-LD in "Good on" time and a standard deviation of the treatment difference to be 3.0 hours, a sample size of 210 per arm will be needed to ensure at least 90% power at a 0.05 significance level. Assuming approximately an 18% prerandomization drop-out, approximately 510 subjects would need to be enrolled to randomize 420 subjects.

The primary efficacy endpoint of change from baseline in "Good on" time will be analyzed using a mixed model for repeated measures (MMRM) model. The model will include baseline (Visit 4) "Good on" time as a covariate, treatment, visit, and pooled center as fixed effects, and a treatment-by-visit interaction. The model will employ an unstructured within subject covariance matrix and a restricted maximum likelihood (ReML) estimation method. The degree-of-freedom of the denominator will be estimated using the Kenward-Roger method.

The key secondary endpoints (change from baseline in "Off" time, change from baseline in MDS-UPDRS Part III, and change from baseline in the sum of the MDS-UPDRS Parts II and III) will be analyzed using MMRM models similar to the primary analysis model. The proportion of subjects with either "much improved" or "very much improved" on the PGI-C will be analyzed using Cochran-Mantel-Haenszel test to compare the two treatment groups with pooled center as a stratification factor.

In order to control the type I error rate, the primary and key secondary endpoints will be tested in a single hierarchical order: (1) change from baseline in "Good on" time, (2) change from baseline in "Off" time, (3) proportion of subjects with either "much improved" or "very much improved" in PGI-C, (4) change from baseline in the MDS-UPDRS Part III, (5) change from baseline in the sum of MDS-UPDRS Parts II and III.

Quantitative safety data will be summarized using descriptive statistics and frequency distributions. Qualitative safety data will be summarized by frequencies and percentages. All summaries will be presented by treatment arms.

# 2. TABLE OF CONTENTS, LIST OF TABLES, AND LIST OF FIGURES

# TABLE OF CONTENTS

| 1. | SYNOPSIS | 5 |
|---|---|---|
| 2. | TABLE OF CONTENTS, LIST OF TABLES, AND LIST OF FIGURES | 10 |
| 3. | LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS | 16 |
| 4. | INTRODUCTION | 19 |
| 5. | TRIAL OBJECTIVES | 23 |
| 6. | INVESTIGATIONAL PLAN | 24 |
| 6.1. | Overall Study Design. | 24 |
| 6.2. | Number of Subjects | 25 |
| 6.3. | Treatment Assignment | 26 |
| 6.4. | Dosing and Dose Determination Criteria | 26 |
| 6.4.1. | IR CD-LD Dose Adjustment Period | 26 |
| 6.4.2. | IPX203 Dose Conversion Period. | 26 |
| 6.4.3. | Double-Blind Maintenance Period | 28 |
| 6.5. | Criteria for Study Termination | 28 |
| 7. | SELECTION AND WITHDRAWAL OF SUBJECTS | 29 |
| 7.1. | Subject Inclusion Criteria | 29 |
| 7.2. | Subject Exclusion Criteria | 30 |
| 7.3. | Subject Withdrawal Criteria | 31 |
| 8. | STUDY PROCEDURES | 33 |
| 8.1. | Screening Visit. | 37 |
| 8.2. | Visit 1 – Start of IR CD-LD Dose Adjustment | 38 |
| 8.2.1. | Prior to Visit 1 | 38 |
| 8.2.2. | At Visit 1 | 38 |
| 8.2.3. | Post Visit 1 | 39 |
| 8.3. | Visits 2 (Week 3) and Visit 3 (Week 5) – IPX203 Dose Conversion | 39 |
| 8.3.1. | Prior to Visit 2 | 39 |
| 8.3.2. | Prior to Visit 3 | 39 |
| 833 | At Visits 2 and 3 | 39 |

| 8.3.4. | Post Visits 2 and 3 | 40 |
|--------|--------------------------------------------------|----|
| 8.4. | Visit 4 (Week 7) – Randomization | 40 |
| 8.4.1. | Prior to Visit 4 | 40 |
| 8.4.2. | At Visit 4. | 40 |
| 8.5. | Visit 5 (Week 10) and Visit 6 (Week 15) | 41 |
| 8.5.1. | Prior to Visit 5 and 6 | 41 |
| 8.5.2. | At Visit 5 and 6 | 41 |
| 8.6. | Visit 7 (Week 20) – End of Study/Study Exit | 42 |
| 8.6.1. | Prior to Visit 7 | 42 |
| 8.6.2. | At Visit 7 | 42 |
| 8.7. | Early Termination | 43 |
| 8.7.1. | Subjects Who Terminate Prior to Randomization | 43 |
| 8.7.2. | Subjects Who Terminate Early after Randomization | 44 |
| 8.8. | Blood Volume | 44 |
| 9. | TREATMENT OF SUBJECTS | 45 |
| 9.1. | Description of Study Drug. | 45 |
| 9.2. | Concomitant Medications | 45 |
| 9.2.1. | Permitted PD Medications | 45 |
| 9.2.2. | Prohibited Medications and Procedures | 45 |
| 9.2.3. | Rescue Medications | 46 |
| 9.3. | Treatment Compliance | 46 |
| 9.4. | Randomization and Blinding | 46 |
| 10. | STUDY DRUG MATERIALS AND MANAGEMENT | 47 |
| 10.1. | Study Drug | 47 |
| 10.2. | Study Drug Packaging and Labeling | 47 |
| 10.3. | Study Drug Storage | 47 |
| 10.4. | Study Drug Administration | 48 |
| 10.5. | Study Drug Dispensing and Accountability | 48 |
| 10.6. | Study Drug Handling and Disposal | 48 |
| 11. | ASSESSMENT OF EFFICACY | 49 |
| 11.1. | Parkinson's Disease Diary | 49 |
| 11.2. | Patient and Investigator Global Assessments | 49 |

| 11.3. | Movement Disorders Society Version of Unified Parkinson's Disease Rating Scale | 49 |
|---|---|---|
| 11.4. | Additional Assessments | 50 |
| 12. | ASSESSMENT OF SAFETY | 51 |
| 12.1. | Safety Parameters | 51 |
| 12.2. | Adverse Events | 51 |
| 12.2.1. | Definition of Adverse Event | 51 |
| 12.2.2. | Recording Adverse Events | 51 |
| 12.2.3. | Follow-up | 52 |
| 12.2.4. | Relationship to Study Drug | 52 |
| 12.2.5. | Assessment of Severity | 52 |
| 12.3. | Serious Adverse Events | 52 |
| 12.3.1. | Definition of Serious Adverse Event | 52 |
| 12.3.2. | Reporting Serious Adverse Events | 53 |
| 12.4. | Pregnancy | 53 |
| 12.5. | Other Safety Parameters and Related Information | 54 |
| 13. | STATISTICS | 55 |
| 13.1. | Study Design and Sample Size Estimation. | 55 |
| 13.2. | Demographics/Baseline Comparability | 55 |
| 13.3. | Efficacy Endpoints | 55 |
| 13.4. | Analysis of Efficacy Data | 57 |
| 13.4.1. | Primary Efficacy Endpoint | 57 |
| 13.4.2. | Key Secondary Efficacy Endpoints | 57 |
| 13.4.3. | Additional Efficacy Endpoints | 58 |
| 13.5. | Center Pooling Algorithm. | 58 |
| 13.6. | Sensitivity Analyses of the Primary Endpoint and Key Secondary Endpoints | 59 |
| 13.6.1. | Assessing Assumptions of the Mixed Model for Repeated Measures (MMRM) | 59 |
| 13.6.2. | Complete Case Analysis | 59 |
| 13.6.3. | Single LOCF/BLOCF Imputation | 59 |
| 13.6.4. | Pattern-Mixture Model | 60 |
| 13.7. | Subgroup Analyses | 61 |
| 13.8. | Multiplicity Adjustments | 61 |

| 13.9. | Analysis Populations | 62 |
|---|---|---|
| 13.9.1. | Safety Analysis Set | 62 |
| 13.9.2. | Intent-to-Treat Analysis Set. | 62 |
| 13.9.3. | Modified Intent-to-Treat Analysis Set | 62 |
| 13.9.4. | Completers Analysis Set. | 62 |
| 13.10. | Handling of Missing Data | 62 |
| 13.10.1. | Missing Data for PD Diaries. | |
| 13.10.2. | Missing Data for Global Assessments (PGI-C, | 63 |
| 13.10.3. | Missing Data for MDS-UPDRS | |
| 13.11. | Analysis of Safety | 64 |
| 14. | ADMINISTRATIVE PROCEDURES | 65 |
| 14.1. | Guidelines for Good Clinical Practice | 65 |
| 14.2. | Institutional Review Board Approval | 65 |
| 14.3. | Informed Consent | 65 |
| 14.4. | Study Monitoring | 65 |
| 14.5. | Protocol Amendments | 65 |
| 14.6. | Termination of Study | 66 |
| 14.7. | Case Report Forms | 66 |
| 14.8. | Investigator's Final Conduct Report | 66 |
| 14.9. | Records Retention | 66 |
| 15. | PUBLICATION POLICY | 67 |
| 16. | LIST OF REFERENCES. | 68 |
| 17. | APPENDICES | 70 |
| APPEND | IX A. PRESCRIBING INFORMATION FOR IR CD-LD | 70 |
| APPEND | IX B. INSTRUCTIONS FOR DOSE CONVERSION TO IPX203 | 82 |
| APPEND | IX C. UNITED KINGDOM PARKINSON'S DISEASE SOCIETY BRAIN BANK DIAGNOSTIC CRITERIA FOR PARKINSON'S DISEASE | 84 |
| APPEND | IX D. MONTREAL COGNITIVE ASSESSMENT (MOCA) | 85 |
| APPEND: | IX E. MOVEMENT DISORDERS SOCIETY VERSION OF UNIFIED PARKINSON'S DISEASE RATING SCALE (MDS-UPDRS) | 91 |
| APPEND | IX F. PATIENT GLOBAL IMPRESSION OF CHANGE (PGI-C) | 125 |

| APPENDIX K. | GASTROPARESIS CARDINAL SYMPTOM INDEX (GCSI) | 135 |
|-------------|--------------------------------------------------------|-----|
| APPENDIX O | COLUMBIA-SUICIDE SEVERITY RATING SCALE (C-SSRS) | 146 |
| | PARKINSON'S DISEASE DIARY | |
| | EXCIPIENTS IN IPX203, IPX203 PLACEBO, IR CD-LD, AND IR | 133 |
| | CEBO | 157 |
| APPENDIX R. | CLINICAL LABORATORY STUDIES | 158 |

# LIST OF TABLES

| Table 1: | Abbreviations and Specialist Terms | 16 |
|---|---|---|
| Table 2: | LD Dosage in Study IPX203-B14-02 | 20 |
| Table 3: | Recommended Starting IPX203 LD Dosing Regimen Based on the Dosing Regimen of IR CD-LD at the End of the Dose Adjustment Period | 27 |
| Table 4: | Events Schedule for Impax Study IPX203-B16-02 | 34 |
| Table 5: | Study Drugs for Study IPX203-B16-02 | 45 |
| | LIST OF FIGURES | |
| Figure 1: | Study Flow Chart | 25 |

# 3. LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

The following abbreviations and specialist terms are used in this study protocol.

Table 1: Abbreviations and Specialist Terms

| Abbreviation or Specialist Term | Explanation |
|---|---|
| AADC | aromatic amino acid decarboxylase |
| ADL | activities of daily living |
| AE | adverse event |
| ANCOVA | analysis of covariance |
| ANOVA | analysis of variance |
| BLOCF | baseline observation carried forward |
| BMI | body mass index |
| CD | carbidopa |
| CR | controlled release |
| CRF | case report form |
| C-SSRS | Columbia-Suicide Severity Rating Scale |
| ECG | electrocardiogram |
| ER | extended release |
| FDA | Food and Drug Administration |
| GCP | Good Clinical Practice |
| GCSI | Gastroparesis Cardinal Symptom Index |
| HIPAA | Health Insurance Portability and Accountability Act |
| ICF | informed consent form |
| ICH | International Conference on Harmonization |
| IEC | independent ethics committee |

| Abbreviation or Specialist Term | Explanation |
|---|---|
| IR | immediate release |
| IRB | institutional review board |
| IWRS | interactive web response system |
| LD | levodopa |
| LOCF | last observation carried forward |
| MAOI | monoamine oxidase inhibitors |
| MAR | missing at random |
| M-EDL | Motor Aspects of Experiences of Daily Living |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MDS-UPDRS | Movement Disorders Society version of the Unified Parkinson's Disease Rating Scale |
| mITT | modified intent-to-treat |
| MMRM | mixed model for repeated measures |
| MNAR | missing not at random |
| MoCA | Montreal Cognitive Assessment |
| nM-EDL | Non-Motor Aspects of Experiences of Daily Living |
| PD | Parkinson's disease |
| PGI-C | Patient Global Impression of Change |
| PK | pharmacokinetic (adjective)<br>pharmacokinetics (singular noun) |
| PI | principal investigator |

| Abbreviation or Specialist Term | Explanation |
|---------------------------------|----------------------------------|
| PMM | pattern-mixture models |
| ReML | restricted maximum likelihood |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SD | standard deviation |
| TEAE | treatment-emergent adverse event |
| US | United States |

#### 4. INTRODUCTION

Parkinson's disease (PD) is a progressive neurodegenerative disorder of the extrapyramidal nervous system. Levodopa (LD) used in combination with carbidopa (CD) is considered the gold standard for the symptomatic treatment of PD. LD is a dopamine precursor converted to dopamine by aromatic amino acid decarboxylase (AADC). Carbidopa is an AADC inhibitor that does not cross the blood-brain barrier. When used in combination with LD, CD increases the plasma half-life of LD from 50 minutes to 1.5 hours. Carbidopa inhibits the conversion of LD into dopamine in the periphery, thereby reducing the peripheral side-effects caused by dopamine and increasing the amount of LD available for transport into the brain. The administration of CD with LD reduces the dose of LD required to produce a dopaminergic response by about 75 percent (Sinemet prescribing information; Appendix A).

Due to its proven efficacy, LD is prescribed eventually to most subjects with PD. However, long-term use of LD is associated with certain complications, including "wearing-off" or "end-of-dose effect," where symptom control decreases causing the drug effects to wear off sooner. As the disease progresses further, motor complications, namely dyskinesias and motor "On/Off" fluctuations, develop in about 50% of the patients after 5 years of treatment (Fahn 1999). Such motor complications can be a significant source of disability and their management is a major unmet need in the treatment of PD.

Mechanisms underlying motor complications involving dyskinesias and "On/Off" fluctuations in PD are unclear. The pulsatile nature of standard orally administered LD is thought to contribute to the appearance of motor complications. Chronic intermittent pulsatile stimulation of the dopamine receptors that are under tonic control contributes to the development of dyskinesia in PD animal models as compared to animals treated with continuous infusion (Juncos et al 1989, Engber et al 1989, Blanchet et al 1995). In addition, unreliable absorption of LD potentially due to erratic gastric empting and variable in vivo dissolution of LD products is thought to contribute to the delay or inadequate response after oral dosing with standard CD-LD products (Melamed et al 1986, Kurlan et al 1988, Stocchi et al 1994). These findings suggest that motor complications in patients with PD may be less likely to develop with continuous dopaminergic stimulation.

Intraduodenal infusion of LD has been shown to significantly reduce motor complications and to reduce "Off" time. The findings of infusion studies in PD patients indicate that the maintenance of stable plasma LD concentrations and the avoidance of low trough levels are effective in reducing "Off" hours, increasing "On" hours without disabling dyskinesia, and reducing the severity of dyskinesia versus standard oral LD formulations (Mizuno 2007, Nilsson et al 2001, Nyholm et al 2005, Stocchi et al 2005). These findings provide a strong rationale for the development of an extended-release (ER) oral dosage form that delivers a constant LD plasma concentration in order to optimize relief of PD symptoms, and to minimize "Off" time and dyskinesia.

IPX203 is an investigational product containing CD-LD that is being developed by Impax Laboratories, LLC (Impax). The primary objective of the IPX203 program is to develop an extended-release product that can attain therapeutic LD plasma concentrations rapidly and

720

810

200

250

maintain constant LD plasma concentrations for a longer duration than currently approved products with minimal peak-to-trough fluctuations. IPX203 is designed to be dosed approximately every 8 hours.

Impax characterized the PK and pharmacodynamics of IPX203 in Study IPX203-B14-02, a single dose trial in subjects with advanced PD versus IR CD-LD and Rytary (carbidopa and levodopa) extended-release capsules. Twenty-six (26) subjects were randomized with 25 subjects completing all 3 treatments. One subject discontinued study early due to subject withdrawal. The doses of IPX203 and Rytary were determined on the basis of each subject's prestudy baseline morning dose of IR CD-LD (Table 2).

| Prestudy Baseline<br>Morning<br>IR LD (mg) | IR LD (mg) | Rytary<br>LD (mg) | IPX203<br>LD (mg) |
|---|---|---|---|
| 100 | 100 | 340 | 360 |
| 150 | 150 | 485 | 540 |

630

780

200

250

Table 2: LD Dosage in Study IPX203-B14-02

Administration of IPX203 yielded an initial increase in LD plasma concentrations that was similar to IR CD-LD but maintained LD concentrations for a longer duration than either IR CD-LD or Rytary. The bioavailability of LD (based on  $AUC_{\infty}$ ) from IPX203 was 88% relative to IR CD-LD and about 11% more than Rytary. Plasma exposure to LD ( $C_{max}$  and  $AUC_{\infty}$ ) following IPX203 increased in an approximately dose-proportional manner. Pharmacodynamic effects as measured by change from baseline scores on MDS-UPDRS Part III were consistent with the PK profiles of LD. Following IPX203 treatment, decrements in the Part III total score (reflecting improvements in motor symptoms) lasted for a longer duration than either IR CD-LD or Rytary. IPX203 provided a longer duration of effect compared with IR CD-LD and Rytary, including "Off" time and "Good on" time based on the Assessment of Subject's Motor State and on a range of improvement thresholds of the MDS-UPDRS Part III. The results were consistent with the prolonged LD plasma concentration profile with IPX203

compared to IR CD-LD or Rytary and support a dosing interval of approximately 8 hours.

Of the 26 subjects who received at least one of the 3 treatments, 9 (34.6%) reported at least one treatment-emergent adverse event (AE). None of these subjects reported a serious AE (SAE) nor did any subjects prematurely discontinue the study because of an AE. Adverse events were reported by more subjects during IR (28.0%) and IPX203 (19.2%) than during Rytary (8.0%) treatment. None of the reported AEs were classified as "severe." Adverse events reported by 2 or more subjects include: Dizziness (3 subjects), nausea (2 subjects), and hypertension (2 subjects). The numbers of subjects reporting these AEs during any single treatment period were small (0 to 2 subjects). Two subjects reported dizziness during IR CD-LD treatment and one subject each during IPX203 and Rytary treatments. Hypertension was reported by a total of 2 subjects, both reporting this AE during IPX203 and IR CD-LD treatments and 1 subject during Rytary treatment. Two subjects reported nausea only during the IR CD-LD treatment period. Of the 9 subjects reporting AEs, 6/26 (23.1%) of subjects reported AEs that were assessed as related to treatment, including all of the reports of dizziness, nausea, and dyskinesia (1 subject).

Study IPX203-B16-01 is a randomized, open-label, rater-blinded, multicenter, 2-treatment, 2-period, multiple-dose crossover study that has completed dosing. Twenty-eight (N=28) advanced PD subjects were randomized to 1 of 2 dosing sequences, with each treatment period lasting 15 days and separated by a 1-week wash-out period where subjects return to their usual stable pre-study CD-LD regimen. The objectives of this study are to compare the PK, pharmacodynamics, efficacy, and safety of IPX203 with IR CD-LD after single and multiple dosing. Subjects were permitted to take allowed non-CD-LD based PD medications throughout the study if dosing regimens had been stable for at least 4 weeks. Subjects were instructed to take their last dose of CD-LD no later than 10:00 PM on the evening prior to Day 1 of each treatment period and to withhold dosing for at least 5 hours before arriving at the site on Day 15 of each treatment period. On Day 1 of the IR CD-LD treatment period, subjects were started with a single dose of their usual prestudy first morning IR CD-LD dose. On Day 1 of the IPX203 treatment period, subjects were started with a single dose of IPX203 based on their usual prestudy first morning IR CD-LD dose using a LD conversion of 100 mg IR LD to 360 mg of IPX203 LD. During the IR CD-LD treatment period, the initial dosing regimen of IR CD-LD was the same as the subject's stable prestudy regimen. During the IPX203 treatment period, the IPX203 regimen for subsequent doses for the day was determined by identifying the most frequent prestudy IR LD dose in milligrams that the subject received in the afternoon and evening and administering IPX203 using a LD conversion of 100 mg IR LD to 270 mg of IPX203 LD. The protocol recommended that IPX203 be dosed approximately every 7 to 8 hours. During Days 1 through 9 of both treatment periods, investigators had the opportunity to adjust each subject's study medication regimen if necessary to optimize efficacy and safety. Pharmacokinetics and pharmacodynamics (MDS-UPDRS Part III and Assessments of Subject's Motor State) were periodically evaluated on Day 1 and Day 15 of each treatment period by qualified clinical staff who were blinded to dosing.

Data from this multiple-dose study confirmed the PK and pharmacodynamic results observed in the single dose study with IPX203:

- PK data from 27 subjects indicates IPX203 shows a rapid increase in LD concentrations followed by extended-release characteristics. Following IPX203; initial increases in LD concentrations were comparable to that from IR CD-LD. Bioavailability of LD following IPX203 was ~89% relative to IR CD-LD. LD plasma concentrations were sustained longer after IPX203 treatment than after IR CD-LD and support dosing every 8 hours. No accumulation of LD was evident at steady-state following IPX203 or IR CD-LD. Plasma LD concentrations following IPX203 were characterized by lower peak-to-trough fluctuation. No time-variant or time-dependent changes were noted in PK of CD or LD following IPX203.
- IPX203 demonstrated an onset of effect that was comparable to IR CD-LD in MDS-UPDRS Part III scores. IPX203 prolonged the duration over which MDS-UPDRS Part III scores were improved by prespecified threshold changes from baseline (≥4, ≥7, and ≥13 units).
- IPX203 provides a significant decrease in "Off" time and a significant increase in "Good on" time compared to IR CD-LD treatment on Day 1 and Day 15 when assessed by the Investigator's Assessment of Subject's Motor State. Subjects treated

with IPX203 did not experience a significant increase in "On" time with troublesome dyskinesia compared to IR CD-LD.

- Subjects achieved significant improvements in "Off" time, "Good on" time, and frequency of motor state fluctuations based on the 3-day PD Diaries.
- Twenty-eight subjects were enrolled in the multiple dose study and 27 subjects completed both treatments. Safety results were as follows:
  - One subject discontinued during the IPX203 treatment period due to an AE (orthostatic hypertension) that was considered possibly related to treatment.
  - A total of 39.3% (11/28) of treated subjects reported at least one treatment emergent AE, including 35.7% (10/28) during IPX203 treatment and 7.4% (2/27) during IR CD-LD treatment. Eight subjects reported AEs that were related to treatment (8 subjects during IPX203 treatment and 1 during IR CD-LD treatment).
  - Two subjects experienced serious adverse events (SAEs). One subject reported increased hypertension of mild severity during IPX203 treatment that was considered unrelated to treatment and resolved. A second subject reported moderate to severe dehydration, diarrhea, and atrial fibrillation during the washout period that were considered unrelated to treatment and resolved.
  - AEs reported in 2 or more subjects included nausea (2), dizziness (2), and dyskinesia (5), all of mild or moderate severity, and all during the IPX203 treatment.

The current protocol, Study IPX203-B16-02, is a multicenter, randomized, double-blind, double-dummy, active-controlled, parallel-group, Phase 3 study. It is designed to compare the efficacy, safety and tolerability of IPX203 with IR CD-LD following multiple doses over 13 weeks. The following IPX203 dosing guidelines will be utilized in the present study (IPX203-B16-02):

- The initial regimen of IPX203 is based on the most frequent dose of the subject's dosing regimen of IR CD-LD at the end of dose adjustment period (Visit 2);
- A 25-100 mg dose of IR CD-LD will be converted to a 70-280 mg CD-LD dose of IPX203;
- IPX203 will be administered approximately every 8 hours for most subjects;
- Investigators may adjust the IPX203 regimen during the dose conversion period to
  optimize the therapeutic effect (minimize "Off" time without causing troublesome
  dyskinesia or other dopaminergic side effects).

The proposed dose conversion scheme for this study has been developed based on a similar dose conversion from IR CD-LD to IPX203 that was studied in the completed Phase 2a study (IPX203-B14-02, n=25) and the Phase 2b study (IPX203-B16-01, n=28), both conducted in subjects with advanced PD using similar entry criteria to the present study. The doses of IPX203 are expected to be comparable to other ER CD-LD products, such as Rytary and Duopa.

# 5. TRIAL OBJECTIVES

To evaluate the safety and efficacy of IPX203 in comparison to IR CD-LD in the treatment of CD-LD experienced subjects with Parkinson's disease (PD) who have motor fluctuations.

#### 6. INVESTIGATIONAL PLAN

## 6.1. Overall Study Design

This is a multicenter, randomized, double-blind, double-dummy, active-controlled, parallel-group study. Subjects will continue to take permitted non-CD-LD-based PD medications throughout the study if documented in their prestudy regimen and if dosing regimens have been stable for at least 4 weeks prior to Visit 1. A "stable dosing regimen" means no change in dose or in dosing frequency. Within 4 weeks following the Screening visit, eligible subjects will complete their PD Diaries on each of the 3 consecutive days immediately prior to Visit 1.

Following Visit 1, qualified subjects will enter a 3-week, open-label IR CD-LD treatment period allowing for dose adjustment. During the IR CD-LD dose adjustment period, the initial dosing regimen of IR CD-LD will be the same as the subject's stable prestudy regimen unless the subject is taking a single daily bedtime dose of CR CD-LD, in which case, the CR CD-LD dose will be discontinued and substituted with a 1:1 milligram-equivalent dose of IR CD-LD. A "bedtime dose" is defined as the last daytime dose of CD-LD taken within 1 hour of onset of the subject's normal nighttime sleep period. The dosing regimen of IR CD-LD may be adjusted during the dose adjustment period to minimize "Off" time without causing troublesome dyskinesia. The doses and regimens of the subject's other non-CD-LD Parkinson's disease medications (dopamine agonists, MAO-B inhibitors, amantadine, anticholinergics) should remain stable throughout this study. Any adjustments to the IR CD-LD dosing regimen will be done in consultation with the Investigator or qualified site personnel and will be recorded. The subject must be on a stable dosing regimen (no change in dose or in dosing frequency) of IR CD-LD for at least 5 days prior to returning for Visit 2. Rescue with additional or modified doses of concomitant PD medications or with use of CD-LD products other than the dispensed study medications is not permitted and will trigger discontinuation from the study. Subjects will complete their 3-day PD Diaries on each of the 3 consecutive days immediately prior to Visit 1.

Following completion of the IR CD-LD dose adjustment period, subjects will begin a 4-week open-label period for conversion to IPX203. The initial dosing regimen of IPX203 during the conversion period will be based on the subject's dosing regimen of IR CD-LD at the end of the dose adjustment period (Visit 2) selecting the most frequent dose according to Table 3. A 25-100 mg dose of IR CD-LD converts to a 70-280 mg CD-LD dose of IPX203 but with a longer duration of effect. It is recommended that IPX203 should be dosed approximately every 8 hours with the exception that subjects who are currently receiving a total daily dose of less than 125-500 mg IR CD-LD at the end of the dose adjustment period will be initially administered IPX203 every 12 hours. The dosing interval may be reduced to approximately every 8 hours if the subject does not achieve an acceptable duration of effect. The dosing regimen of IPX203 may be adjusted during the dose conversion period to achieve the optimal balance of efficacy and tolerability (minimize "Off" time without causing troublesome dyskinesia or other dopaminergic side effects). Any adjustments to the IPX203 dosing regimen will be recorded. Rescue with additional or modified doses of concomitant PD medications or with use of CD-LD products other than the dispensed study medications is not permitted and will trigger discontinuation from the study. Subjects will return to the clinic in two weeks for Visit 3 followed by Visit 4 two weeks later. The subject must be on a stable dosing regimen of IPX203

(no change in dose or in dosing frequency) for at least 5 days prior to returning for Visit 4. Subjects will also be instructed to complete their 3-day PD Diaries on each of the 3 consecutive days immediately prior to Visit 4.

The study staff will call the subjects frequently (approximately every 1 to 3 days) during the IR CD-LD dose adjustment and IPX203 dose conversion periods. The calls are to ensure timely and appropriate dosing adjustments and to ensure that the subject is able to follow and adhere to the dosing instructions. The contacts may be less frequent after initial dose adjustments have been made. Any changes in the dosing regimen will be in consultation with the Investigator or qualified site personnel and will be documented.

Subjects who successfully complete the IPX203 dose conversion period will be randomized, stratified by center, in a 1:1 ratio at Visit 4 into one of two parallel treatment arms of IPX203 (with matching IR CD-LD placebo) or IR CD-LD (with matching IPX203 placebo). The subjects will undergo 13 weeks of double-blind, double-dummy maintenance therapy with the stable dosing regimen established at the end of Week 3 (Visit 2) for IR CD-LD and at the end of Week 7 (Visit 4) for IPX203. Subjects will return to the clinic for 3 visits (Visits 5, 6, and 7) and will be instructed to complete their 3-day PD Diaries on 3 consecutive days immediately prior to each of the 3 visits. Rescue with additional or modified doses of concomitant PD medications or use of CD-LD products other than the dispensed study medication is not permitted and will trigger discontinuation from the study.



Figure 1: Study Flow Chart

Abbreviations: IR=immediate-release, CD=carbidopa, LD=levodopa, ET=early termination

# 6.2. Number of Subjects

Assuming approximately an 18% prerandomization drop-out, approximately 510 subjects will be enrolled to randomize 420 subjects.

## 6.3. Treatment Assignment

Investigational product: IPX203 (carbidopa-levodopa) Extended-Release Capsules containing 35-140 mg of CD-LD, for oral administration.

Reference therapy: Immediate-Release carbidopa-levodopa (IR CD-LD) tablets containing 25-100 mg of CD-LD, for oral administration.

Subjects will be randomly assigned to one of two parallel treatment arms to receive either IPX203 (with matching IR CD-LD placebo) or IR CD-LD (with matching IPX203 placebo) during the double-blind maintenance therapy portion of the study.

# 6.4. Dosing and Dose Determination Criteria

IR CD-LD will be supplied as tablets containing 25-100 mg of CD-LD. IR CD-LD tablets may be split to achieve the required dose.

IPX203 will be supplied as capsules containing 35-140 mg of CD-LD. The suggested doses and regimen of IPX203 are intended to provide an onset of effect comparable to the subject's prestudy IR LD regimen and to extend the duration of effect. A 25-100 mg dose of IR CD-LD converts to a 70-280 mg CD-LD dose of IPX203.

#### 6.4.1. IR CD-LD Dose Adjustment Period

During the 3-week IR CD-LD dose adjustment period, the initial dosing regimen of IR CD-LD will be the same as the subject's stable prestudy regimen unless the subject is taking a single daily bedtime dose of CR CD-LD, in which case, the CR CD-LD dose will be discontinued and substituted with a 1:1 milligram-equivalent dose of IR CD-LD. A "bedtime dose" is defined as the last daytime dose of CD-LD taken within 1 hour of onset of the subject's normal nighttime sleep period. Subjects who were receiving IR CD-LD as a 1:10 CD-LD formulation will be started on IR CD-LD with a 1:4 ratio at the same frequency and LD dose. **The dosing regimen of IR CD-LD may be adjusted during the dose adjustment period** to minimize "Off" time without causing troublesome dyskinesia. The doses and regimens of the subject's other non-CD-LD Parkinson's disease medications (dopamine agonists, MAO-B inhibitors, amantadine, anticholinergics) should remain stable throughout this study. Any adjustments to the IR CD-LD dosing regimen will be done in consultation with the Investigator or qualified site personnel and will be recorded. The subject must be on a stable dosing regimen (no change in dose or in dosing frequency) of IR CD-LD for at least 5 days prior to returning for Visit 2.

#### 6.4.2. IPX203 Dose Conversion Period

During the 4-week IPX203 dose conversion period, the suggested initial dosing regimen of IPX203 will be based on the most frequent dose of the subject's <u>dosing regimen of IR CD-LD at</u> the end of the dose adjustment period (Visit 2). A 25-100 mg dose of IR CD-LD converts to a 70-280 mg CD-LD dose of IPX203, and a half tablet (12.5-50 mg dose of IR CD-LD) converts to a 35-140 mg CD-LD dose of IPX203. To facilitate conversion of subjects from IR CD-LD to IPX203, Table 3 presents recommended starting dose regimens. It is recommended that IPX203 should be dosed approximately every 8 hours with the exception that subjects who are currently receiving a total daily dose of less than 125-500 mg IR CD-LD at the end of the dose adjustment

period will be initially administered IPX203 every 12 hours. The dosing interval may be reduced to approximately every 8 hours if the subject does not achieve an acceptable duration of effect. **The dosing regimen of IPX203 may be adjusted during the dose conversion period** to achieve the optimal balance of efficacy and tolerability (minimize "Off" time without causing troublesome dyskinesia or other dopaminergic side effects). The maximum recommended daily dose of IPX203 is 600-2400 mg CD-LD. The doses and regimens of the subject's other non-CD-LD Parkinson's disease medications (dopamine agonists, MAO-B inhibitors, amantadine, anticholinergics) should remain stable throughout this study. The subject must be on a stable dosing regimen of IPX203 (no change in dose or in dosing frequency) for at least 5 days prior to returning for Visit 4.

Table 3: Recommended Starting IPX203 LD Dosing Regimen Based on the Dosing Regimen of IR CD-LD at the End of the Dose Adjustment Period

| Most Frequent IR CD-LD Unit Dose (mg) | Recommended Starting IPX203 Daily Dosing Regimen<br>CD-LD (mg) Every 8 Hours |
|---|---|
| 25-100 <sup>a</sup> | 70-280 mg (2 × 35-140 mg) |
| >25-100 – 37.5-150 | 105-420 mg (3 × 35-140 mg) |
| >37.5-150 – 50-200 | 140-560 mg (4 × 35-140 mg) |
| >50-200 | 175-700 mg (5 × 35-140 mg) |

<sup>&</sup>lt;sup>a</sup> Subjects who are on a total daily dose of less than 125-500 mg CD-LD from IR CD-LD should be advised to initially take IPX203 every 12 hours. The dosing interval may be reduced to approximately every 8 hours if the subject does not achieve an acceptable duration of effect.

During the dose conversion to IPX203, the Investigator or site staff are advised to be in frequent contact (every 1 to 3 days) with the subject especially during the initial dose conversion to assess the need for dosage adjustment with the goal of minimizing "Off" time without causing troublesome dyskinesia. Any changes to the dosing regimen should only be made by the Investigator or qualified site personnel. If the subject experiences troublesome dyskinesias during initial dose conversion, consider reducing the dose by one capsule (35-140 mg IPX203 CD-LD) before increasing the dosing interval. If turning "On" is slow following the first morning dose, consider taking the morning dose in the fasted state and/or increasing the dose by one capsule (35-140 mg IPX203 CD-LD). If turning "On" is slow later in the day or to reduce "end-of-dose" "Off" time, consider increasing the dose by one capsule (35-140 mg IPX203 CD-LD).

When two or more IR CD-LD doses correspond to the most frequent IR CD-LD dose, the suggested IPX203 conversion should be based on the higher of the IR CD-LD doses.

A summary of the instructions for dose conversion to IPX203 is provided in Appendix B.

#### 6.4.3. Double-Blind Maintenance Period

During the 13-week double-blind double-dummy maintenance period, subjects receive either IPX203 (with matching IR CD-LD placebo) or IR CD-LD (with matching IPX203 placebo) with the stable dosing regimen established at the end of Week 3 (Visit 2) for IR CD-LD and at the end of Week 7 (Visit 4) for IPX203.

# 6.5. Criteria for Study Termination

The Sponsor has the right to terminate this study and remove all study material from the study site at any time for medical or administrative reasons. The Sponsor will endeavor to give adequate notice to allow safe withdrawal of subjects from the study.

#### 7. SELECTION AND WITHDRAWAL OF SUBJECTS

Subjects must meet all of the following inclusion criteria to qualify for enrollment. Subjects who have any of the following exclusion criteria will not be enrolled in the study.

#### 7.1. Subject Inclusion Criteria

- Male or female subjects diagnosed at age ≥ 40 years with PD, consistent with the United Kingdom Parkinson's Disease Society Brain Bank Diagnostic Criteria (Appendix C) and who are being treated with stable regimens of CD-LD but experiencing motor fluctuations.
- 2. Able to provide written informed consent prior to the conduct of any study-specific procedures.
- 3. Female subjects of childbearing potential must have a negative urine pregnancy test at Screening Visit.
- 4. Negative urine screen for drugs of abuse and negative alcohol breath test at Screening.
- 5. Hoehn and Yahr Stages 1, 2, 3, or 4 in the "On" state (part of Movement Disorders Society version of the Unified Parkinson's Disease Rating Scale [MDS-UPDRS] Part III; Appendix E).
- 6. Agrees to use a medically acceptable method of contraception throughout the study and for 6 weeks after completing the study. Medically acceptable methods of contraception that may be used by the subject and/or partner include but are not limited to: abstinence, oral contraception, NuvaRing or transdermal systems, diaphragm with vaginal spermicide, intrauterine device, condom and partner using vaginal spermicide, surgical sterilization (6 months), progestin implant or injection, or postmenopausal female (no menstrual period for > 2 years) or vasectomy (> 6 months).
- 7. Montreal Cognitive Assessment (MoCA) score ≥ 24 at Screening Visit in "On" state (Appendix D).
- 8. By history, for the 4 weeks prior to Screening, the subject experiences daily "wearing-off" episodes with periods of bradykinesia in combination with at least one of rest tremor or rigidity, experiences an "Off" state upon awakening on most mornings, and reports an average of at least 2.5 cumulative hours per day of "Off" time during the waking hours.
- 9. Able to differentiate "On" state from "Off" state as determined by at least 75% concordance with a trained rater in "On/Off" ratings for 8 ratings over the 4-hour training period. The concordance must include at least 1 "On" and 1 "Off" rating and must be achieved within two 4-hour training sessions.
- 10. At Visit 1, review of the 3-day PD Diaries confirms the following: that the subject is able to properly complete the diaries with valid entries; and that the subject has an <u>average of at least 2.5 hours</u> per day of "Off" time during the waking hours over the 3 days with at least 1.5 hours of cumulative "Off" time on each day. Inability to properly complete the

diaries is indicated when more than 1 day of a diary is not returned or when more than 2 hours (4 half-hour periods) of one 24-hour diary day are missing (Appendix P).

- 11. Responsive to CD-LD therapy and currently being treated on a stable regimen with CD-LD for at least 4 weeks prior to Visit 1 and:
  - a. Requires at least 100 mg of LD from IR CD-LD for the first morning dose
  - b. Requires a total daily dose of at least 400 mg of LD and takes a maximum total daily dose of 2400 mg LD, from IR CD-LD alone or IR CD-LD in combination with a single daily bedtime dose of CR CD-LD
  - c. Has a dosing frequency of 4 to 9 times daily of CD-LD
  - d. By history, typically experiences an "On" response with the first dose of IR CD-LD of the day, but the efficacy of this dose typically lasts less than 4 hours.
- 12. At Screening, the subject has predictable "Off" periods defined by a score of 1 or 2 on Item #4.5 (Complexity of Motor Fluctuations) of the MDS-UPDRS Part IV B (Motor Fluctuations) (Appendix E).
- 13. At Screening, the MDS-UPDRS Part III total score in the "Off" state is at least 20 units.
- 14. Able and willing to comply with the protocol, including completion of diaries and availability for all study visits.

# 7.2. Subject Exclusion Criteria

- 1. Used any doses of controlled-release (CR) CD-LD apart from a single daily bedtime dose within 4 weeks prior to Visit 1.
- 2. Used any doses of Rytary for the past 4 weeks prior to Visit 1 or considered IPX066 or Rytary failures for reasons of efficacy or safety.
- 3. Received any investigational medications within 30 days or 5 times the half-life, whichever is longer, prior to Visit 1.
- 4. Female subjects who are currently breastfeeding or lactating.
- 5. Had prior neurosurgical treatment for PD or if such procedure is planned or anticipated during the study period.
- 6. Allergic to any excipient in the study drugs (See Appendix Q).
- 7. History of medical conditions or of a prior surgical procedure that would interfere with LD absorption, such as gastrectomy, proximal small-bowel resection, or bariatric surgery.
- 8. History of upper gastrointestinal hemorrhage in patients with peptic ulcer disease within the past 5 years.
- 9. History of glaucoma with intraocular pressures that are elevated despite appropriate medical management.
- 10. History of seizure or epilepsy and experienced at least 1 seizure during the past 12 months or has not been compliant with medically recommended therapy or visits.
- 11. History of myocardial infarction with residual atrial, nodal, or ventricular arrhythmias that are not controlled with medical and/or surgical interventions. A recent

- $(\leq 12 \text{ months})$  history of myocardial infarction with secondary arrhythmias is exclusionary regardless of the therapeutic control.
- 12. History of neuroleptic malignant syndrome or of nontraumatic rhabdomyolysis.
- 13. Liver enzyme values ≥ 2.5 times the upper limit of normal; or history of severe hepatic impairment.
- 14. Serum creatinine level  $\geq$  1.75 times the upper limit of normal; or requires dialysis at the time of Screening.
- 15. Subject with a history of malignant melanoma or with a suspicious undiagnosed skin lesion which in the opinion of the investigator could be melanoma.
- 16. History of drug or alcohol abuse within the 12 months prior to Screening.
- 17. Received within 4 weeks of Visit 1 or planning to take during participation in the clinical study:
  - a. any doses of a controlled-release (CR) LD apart from a single daily bedtime dose, any doses of Rytary, additional CD (eg, Lodosyn) or benserazide (eg, Serazide), or catechol-O-methyl transferase inhibitors (entacapone or tolcapone) or medications containing these inhibitors (Stalevo),
  - b. nonselective monoamine oxidase inhibitors (MAOI), apomorphine, or antidopaminergic agents, including antiemetics.
- 18. Treatment with any dopamine antagonist for the purposes of treating psychosis or bipolar disorder within the last 2 years or any history of psychosis within the past 10 years regardless of treatment. A brief, self-limited episode of psychosis precipitated by a medical intervention with return to normal mentation is not exclusionary. Mild PD-associated illusions are not exclusionary provided that they do not occur more than twice per week and the subject does not lose insight.
- 19. Employees or family members of the investigator, study site, or sponsor.
- 20. Subjects who have previously participated in an IPX203 study.
- 21. Subjects who, in the opinion of the clinical investigator, should not participate in the study.
- 22. Based on clinical assessment, subject does not adequately comprehend the terminology needed to complete the PD diary.

# 7.3. Subject Withdrawal Criteria

Site personnel should make every effort to conduct all protocol-specific procedures to complete the study. A subject may be discontinued from the study due to the following reasons:

- 1. Withdrawal by subject
- 2. Adverse event (AE)
- 3. Lack of efficacy
- 4. Study terminated by Sponsor

- 5. Protocol deviation
- 6. Noncompliance with study drug
- 7. Lost to follow-up
- 8. Death
- 9. Other

Subjects who withdraw early from the study will not be replaced. The reason or reasons for discontinuation will be specified and documented. Empty medication bottles and any unused study drug upon discontinuation will be collected. Study medication dispensed to a discontinued subject may not be redispensed to a different subject.

# 8. STUDY PROCEDURES

The procedures to be performed at each study visit are described below and summarized in Table 4.

Table 4: Events Schedule for Impax Study IPX203-B16-02

| | | 3 Weeks of<br>IR CD-LD<br>Dose<br>Adjustment | 4 Weeks of<br>IPX203 Dose Conversion | | | 13 Weeks of<br>Double-Blind Therapy | | |
|---|---|---|---|---|---|---|---|---|
| Assessment | Screening | Visit 1 | Visit 2 | Visit 3 | Visit 4<br>Randomization | Visit 5 | Visit 6 | Visit 7 / Study<br>Exit/Early<br>Termination <sup>b</sup> |
| Study Week <sup>a</sup> | -4 | 0 | 3 | 5 | 7 | 10 | 15 | 20 |
| ICF & HIPAA Authorization <sup>c</sup> | X | | | | | | | |
| Contact IWRS | X | X | X | X | X | X | X | X |
| Randomization | | | | | X | | | |
| Inclusion/Exclusion | X | X | | | | | | |
| Medical History | X | | | | | | | |
| Physical Examination | X | | | | | | | X |
| Vital Signs <sup>d</sup> | X | X | X | X | X | X | X | X |
| Height and Weight | X | | | | | X <sup>e</sup> | | X <sup>e</sup> |
| C-SSRS <sup>f</sup> | X | X | X | X | X | X | X | X |
| Clinical Laboratory Tests <sup>g</sup> | X | | | | | X | | X |
| Urine Pregnancy Test | X | | | | | | | |
| Urine Screen for Drug Abuse | X | | | | | | | |
| Alcohol Breath Test | X | | | | | | | |
| ECG | X | | | | | X | | X |
| MoCA <sup>h</sup> | X | | | | | | | |
| MDS-UPDRS Parts I-IV | Xi | X | X | | X | X | X | X |
| PGI-C <sup>j</sup> | | | | | | X | X | X |

| | | 3 Weeks of<br>IR CD-LD<br>Dose<br>Adjustment | 4 Weeks of<br>IPX203 Dose Conversion | | | 13 Weeks of<br>Double-Blind Therapy | | |
|---|---|---|---|---|---|---|---|---|
| Assessment | Screening | Visit 1 | Visit 2 | Visit 3 | Visit 4<br>Randomization | Visit 5 | Visit 6 | Visit 7 / Study<br>Exit/Early<br>Termination <sup>b</sup> |
| Study Week <sup>a</sup> | -4 | 0 | 3 | 5 | 7 | 10 | 15 | 20 |
| GCSI <sup>o</sup> | | X | | | | | | X |
| PD Diary Training; Perform<br>Concordance Testing at<br>Screening Only <sup>5</sup> | х | х | х | x | Х | X | х | |
| Dispense PD Diaries <sup>t</sup> | X | X | | X | X | X | X | |
| Review PD Diaries <sup>u</sup> | | X | X | | X | X | X | X |
| Reminder phone calls <sup>v,w</sup> | X <sup>v</sup> | X <sup>w</sup> | $X^{w}$ | $\mathbf{X}^{\mathbf{w}}$ | $X^{w}$ | X | X | X |
| Dispense study medication | | X | X | X | X | X | X | |
| Collect empty medication bottles<br>and any unused study<br>drug/Perform study drug<br>accountability | | | х | х | х | х | х | х |
| Adverse Events | X | X | X | X | X | X | X | X |
| Concomitant Medications | X | X | X | X | X | X | X | X |

C-SSRS = Columbia-Suicide Severity Rating Scale, ECG = electrocardiogram,
GCSI = Gastroparesis Cardinal Symptom Index, HIPAA = Health Insurance Portability and Accountability Act, ICF = informed consent form, IWRS = interactive web response
system, MDS-UPDRS = MDS version of Unified Parkinson's Disease Rating Scale, MoCA = Montreal Cognitive Assessment,

PD = Parkinson's
disease,
PGI-C =

Patient Global Impression of Change,

The interval between Screening and Visit 1 (Day 1) should not exceed 4 weeks. Study visits should occur within ± 3 days of their specified timing.

- Study Exit procedures to be conducted at the end of Visit 7 or during an early termination visit.
- Subjects enrolled at sites in the United States (US) must sign HIPAA authorization prior to the conduct of any study-specific procedures.
- d Record vital signs (blood pressure, heart rate, respiratory rate, and temperature [Screening and Study Exit only]) after subject has been resting supine for at least 5 minutes, then record orthostatic blood pressure and heart rate after subject has been standing for approximately 2 minutes. At Visits 1 and 4, orthostatic vital signs (blood pressure and heart rate) will be performed in triplicate, each set separated by at least 15 minutes from the previous set.
- e Weight only.
- f C-SSRS: Columbia Suicide Severity Rating Scale. See Appendix O.
- g See Appendix R.
- Montreal Cognitive Assessment in the "On" state: see Appendix D.
- At Screening MDS-UPDRS Parts I through IV will be done in both the "On" and "Off" state (see Appendix E).
- See Appendix F.

  See Appendix K.
- Train at Screening and then as needed at subsequent visits. Perform concordance testing at Screening.
- Dispense PD Diaries at Screening and Visits 1, 3, 4, 5, and 6. Call subjects 4 days prior to Visits 1, 2 and 4-7 to remind them to complete PD Diaries. Subjects record diary information for 3 consecutive days immediately prior to each of the visits (Days -3, -2, and -1). Call subjects the day prior to each visit to remind them to bring the PD Diaries, empty medication bottles, and any unused study drug to the office.
- <sup>u</sup> Review PD Diaries at Visits 1, 2, and 4-7.
- v Post-Screening reminder phone call: Notify individuals who successfully complete screening procedures following review of all study entry criteria and clinical laboratory results that they may continue in the study. The interval between Screening and Visit 1 should not exceed 4 weeks.
- W Reminder phone calls for Visits 1 through 4: In addition to the calls discussed above, make regular phone calls (approximately every 1 to 3 days) to subjects throughout the IR CD-LD dose-adjustment and IPX203 dose-conversion periods to evaluate each subject's adjustment to the study medication regimen.
## 8.1. Screening Visit

After the subject has signed the informed consent (and HIPAA authorization for US subjects only), complete the following procedures and assessments:

- Obtain an identification number from the Interactive Web Response System (IWRS).
   The IWRS will assign a 6-digit ID number to each subject, consisting of a 3-digit number representing the investigative site and a 3-digit sequential subject number.
- Review and record study entry criteria (Section 7).
- Perform urine pregnancy test for females of childbearing potential.
- Perform urine screen for drugs of abuse.
- Perform alcohol breath test.
- Complete medical history.
- Perform physical examination, including height and weight.
- Assess vital signs after subject is supine for at least 5 minutes (blood pressure, heart rate, temperature and respiratory rate) and then assess orthostatic blood pressure and heart rate after subject is standing (for approximately 2 minutes).
- Record current CD-LD regimen, other PD medications and their dosing schedule, and other concomitant medications.
- Record AEs.
- Perform a 12-lead ECG.
- Administer C-SSRS (Appendix O).
- Determine MoCA Score in the "On" state (Appendix D).
- Collect blood and urine samples for clinical laboratory studies (Appendix R).
- Determine Hoehn and Yahr staging of PD in the "On" state (part of MDS-UPDRS Part III Motor Examination) (Appendix E).
- Administer MDS-UPDRS Parts I through IV in the "On" and "Off" state (Appendix E).
- Train the subject how to complete the PD Diaries to assess his/her "On" and "Off" states, including assessment of any dyskinesia. After training the subject, perform the concordance testing. The subject's "On"/"Off" ratings must agree at least 75% of the time with the trained rater during the training sessions. That is, the subject's "On"/"Off" ratings must agree with the trained rater's ratings on at least 75% "On"/"Off" states in a single session to qualify for study inclusion. The 75% concordance rate must be based on 8 ratings, and must include at least one "On" and one "Off" state. The ratings should occur every 30 minutes and each session should last up to 4 hours. If the subject fails the first training session, the subject may be trained for one additional 4-hour training session. This repeat testing should not be

performed on the same day as the first session and can take place from 1 day to 3 weeks post Screening visit.

 Dispense PD Diaries and instruct the subject to complete the PD Diaries on 3 consecutive days immediately prior to Visit 1.

Notify individuals who successfully complete screening procedures following review of all study entry criteria and clinical laboratory results.

The interval between Screening and Visit 1 (Day 1) should not exceed 4 weeks.

# 8.2. Visit 1 – Start of IR CD-LD Dose Adjustment

#### 8.2.1. Prior to Visit 1

Contact the subject at least 4 days prior to Visit 1 to remind him/her to complete the 3-day PD Diaries starting 3 consecutive days immediately prior to Visit 1.

The day prior to Visit 1, remind subjects to:

• Bring their completed 3-day PD Diaries to the clinic.

#### 8.2.2. At Visit 1

For Visit 1 complete the following procedures:

- Collect and review the subject's 3-day PD Diaries. Ensure that the subject is averaging at least 2.5 hours per day of "Off" time over 3 days and at least 1.5 hours of "Off" time on each day based on the 3 day PD Diaries. If the subject cannot properly complete the diary, eg, if more than 1 day of the diary is not returned or if more than 1 day of the diary is not valid (ie, more than 2 hours [4 half periods] of the 24-hour diary are missing), he/she will not continue in the study.
- Review inclusion and exclusion criteria to ensure that the subject continues to meet these criteria.
- Review instruction of 3-day PD Diaries if needed.
- Measure vital signs (respiratory rate, blood pressure, and heart rate after supine for at least 5 minutes, and orthostatic pulse and blood pressure after standing for approximately 2 minutes). Orthostatic vital sign measurements (blood pressure and heart rate) will be performed in triplicate, each set separated by at least 15 minutes from the previous set.
- Administer C-SSRS (Appendix O).
- Administer MDS-UPDRS Parts I through IV (Appendix E).
- •
- •
- Complete GCSI (Appendix K).

- •
- Record any AEs and update changes in concomitant medication since the previous visit.
- Dispense PD Diaries.
- Contact IWRS and dispense study medication per IWRS instructions.

#### 8.2.3. **Post Visit 1**

Make regular phone calls (approximately every 1 to 3 days) while the IR CD-LD dose
is being adjusted. The IR CD-LD dosing regimen should be stable for at least 5 days
prior to returning for Visit 2.

# 8.3. Visits 2 (Week 3) and Visit 3 (Week 5) – IPX203 Dose Conversion

#### 8.3.1. Prior to Visit 2

- Call subjects 4 days prior to Visit 2 and remind them to complete their PD Diaries.
- Call subjects the day prior to Visit 2 to remind them to bring the PD Diaries, empty medication bottles, and any unused study drug to the office.

#### 8.3.2. Prior to Visit 3

• Call subjects the day prior to Visit 3 to remind them to bring back empty medication bottles and any unused study drug to the office.

#### 8.3.3. At Visits 2 and 3

For Visits 2 and 3 complete the following procedures:

- Measure vital signs (respiratory rate, blood pressure, and heart rate after supine for at least 5 minutes, and orthostatic pulse and blood pressure after standing for approximately 2 minutes).
- Administer C-SSRS (Appendix O).
- Collect empty medication bottles and any unused study drug; perform study drug accountability.
- Record and update AEs and concomitant medications.
- Contact IWRS and dispense study medication per IWRS instructions.

## **Additional Assessments at Visit 2 Only**

• Administer MDS-UPDRS Parts I through IV (Appendix E).

- Review PD Diaries. The subject will be terminated from the study if the subject does not average at least 2.5 hours per day of "Off" time over 3 days and at least 1.5 hours of "Off" time on each day based on the 3 day PD Diaries and/or if the subject cannot properly complete the diary, eg, if more than 1 day of the diary is not returned or if more than 1 day of the diary is not valid (ie, more than 2 hours [4 half periods] of the 24 hour diary are missing).
- Ensure that the subject has been on a stable dosing regimen for at least 5 days prior to dose conversion to IPX203. If the subject is not able to achieve a stable dosing regimen lasting at least 5 days, the subject will be discontinued.
- Conduct PD Diaries training, if needed.

## **Additional Activities at Visit 3 Only**

- Dispense PD Diaries.
- Review instruction of 3-day PD Diaries if needed.

#### **8.3.4.** Post Visits 2 and 3

Make regular phone calls (approximately every 1 to 3 days) to subjects throughout the dose conversion period, as needed, to evaluate each subject's adjustment to the study medication. The IPX203 dosing regimen should be stable for at least 5 days prior to returning for Visit 4.

## 8.4. Visit 4 (Week 7) – Randomization

#### **8.4.1.** Prior to Visit 4

- Call subjects 4 days prior to Visit 4 to remind them to complete their PD Diaries.
- Contact subjects 1 day prior to Visit 4 to remind them to bring back the PD Diaries, empty medication bottles, and any unused study drug to the office.

#### 8.4.2. At Visit 4

For Visit 4 complete the following procedures:

- Review PD Diaries. At least 1 day of valid diary data (ie, less than 2 hours [4 half periods] of the 24-hour diary are missing) must be available, otherwise the subject will be terminated from the study.
- Ensure that the subject has been on a stable dosing regimen for at least 5 days prior to randomization. If the subject is not able to achieve a stable dosing regimen lasting at least 5 days, the subject will be discontinued.
- Measure vital signs (respiratory rate, blood pressure, and heart rate after supine for at least 5 minutes, and orthostatic pulse and blood pressure after standing for approximately 2 minutes). Orthostatic vital sign measurements (blood pressure and heart rate) will be performed in triplicate, each set separated by at least 15 minutes from the previous set.
- Administer C-SSRS (Appendix O).

• Administer MDS-UPDRS Parts I through IV (Appendix E).



- Record and update AEs and concomitant medications.
- Conduct PD diaries training, if needed.
- Collect empty medication bottles and any unused study drug; perform study drug accountability.
- Contact IWRS for randomization and dispense medication per IWRS instructions.
- Dispense PD diaries.

## 8.5. Visit 5 (Week 10) and Visit 6 (Week 15)

#### 8.5.1. Prior to Visit 5 and 6

- Call subjects 4 days prior to Visits 5 and 6 to remind them to begin recording in their PD diaries on each of the 3 consecutive days immediately prior to each of these visits.
- Call the subjects the day prior to Visits 5 and 6 to remind the subjects to bring in their PD diaries, empty medication bottles, and any unused study drug to the office.

#### 8.5.2. At Visit 5 and 6

For Visits 5 and 6 complete the following procedures (note visit-specific tasks below):

- Measure vital signs (respiratory rate, blood pressure, and heart rate after supine for at least 5 minutes, and orthostatic pulse and blood pressure after standing for approximately 2 minutes).
- Administer C-SSRS (Appendix O).
- Administer MDS-UPDRS Parts I through IV (Appendix E).
- Complete PGI-C (Appendix F).
- Complete CGI-C (Appendix G).
- Review PD diaries.
- Conduct PD diaries training, if needed.
- Dispense PD diaries.

- Collect empty medication bottles and any unused study drug; perform study drug accountability.
- Contact IWRS and dispense study medication per IWRS instructions.
- Record any AEs and update changes in concomitant medication since the previous visit.

## Additional Activities at Visit 5 Only:

- Record weight.
- Perform a 12-lead ECG.
- Collect blood and urine samples for clinical laboratory studies (Appendix R).

## Additional Activities at Visit 6 Only:

- •
- •

# 8.6. Visit 7 (Week 20) – End of Study/Study Exit

#### **8.6.1. Prior to Visit** 7

- Call subjects 4 days prior to Visit 7 to remind them to begin recording in their PD Diaries on each of the 3 consecutive days immediately prior to Visit 7.
- Call the subjects the day prior to Visit 7 to remind the subjects to bring in their PD Diaries, empty medication bottles, and any unused study drug to the office.

#### 8.6.2. At Visit 7

All enrolled subjects must complete Study Exit procedures at the end of Visit 7 or during an early termination visit:

- Perform physical examination, including weight.
- Measure vital signs (temperature, respiratory rate, blood pressure, and heart rate after supine for at least 5 minutes, and orthostatic pulse and blood pressure after standing for approximately 2 minutes).
- Collect and review 3-day PD Diaries.
- Administer C-SSRS (Appendix O).
- Administer MDS-UPDRS Parts I through IV (Appendix E).
- Complete PGI-C (Appendix F).
- •

- Complete GCSI (Appendix K).
- Collect empty medication bottles and any unused study drug; perform study drug accountability.
- Record and update AEs and concomitant medications.
- Collect blood and urine samples for clinical laboratory studies (Appendix R).
- Perform a 12-lead ECG.
- Contact IWRS to record subject disposition.

## 8.7. Early Termination

## 8.7.1. Subjects Who Terminate Prior to Randomization

If the subject discontinues the study prior to randomization (Visit 4) the subject should complete the following assessments:

- Perform physical examination, including weight.
- Measure vital signs (temperature, respiratory rate, blood pressure, and heart rate after supine for at least 5 minutes, and orthostatic pulse and blood pressure after standing for approximately 2 minutes).
- Collect and review 3-day PD Diaries when available.
- Administer C-SSRS (Appendix O).
- Administer MDS-UPDRS Parts I through IV (Appendix E).
- Collect empty medication bottles and any unused study drug; perform study drug accountability.
- Record and update AEs and concomitant medications.
- Collect blood and urine samples for clinical laboratory studies (Appendix R).
- Perform a 12-lead ECG.
- Contact IWRS to record subject disposition.

# 8.7.2. Subjects Who Terminate Early after Randomization

If the subject discontinues the study after randomization (Visit 4), the subject should complete all assessments described in Section 8.6.2.

## 8.8. Blood Volume

Safety blood draws: Approximately 10 mL of blood will be drawn at Screening, Visit 5, and at Study Exit, for a combined total of 30 mL.

## 9. TREATMENT OF SUBJECTS

## 9.1. Description of Study Drug

Study drugs will be provided by Impax for this study:

- IPX203 (carbidopa-levodopa) Extended-Release Capsules containing 35-140 mg of CD-LD for oral administration. The CD-LD ratio is 1:4. In addition, matching placebo capsules will also be provided.
- Immediate-release carbidopa-levodopa (IR CD-LD) tablet containing 25-100 mg of CD-LD, for oral administration. In addition, matching placebo tablets will also be provided.

Table 5: Study Drugs for Study IPX203-B16-02

| Investigational Product | Dosage Strength (mg CD-LD) and Form |
|---|---|
| IPX203 (carbidopa-levodopa) Extended-<br>Release capsules | 35-140 mg<br>Capsules for oral administration |
| IR CD-LD (carbidopa-levodopa) tablets | 25-100 mg<br>Tablets for oral administration |
| IPX203 Placebo capsules | Capsules for oral administration |
| IR CD-LD Placebo tablets | Tablets for oral administration |

#### 9.2. Concomitant Medications

#### 9.2.1. Permitted PD Medications

Concomitant therapy with amantadine, selective monoamine oxidase (MAO) type B inhibitors (eg, selegiline, rasagiline), anticholinergic PD medications (eg, benztropine, trihexyphenidyl), and/or dopamine agonists (except apomorphine) is allowed provided the doses and regimens have been stable for at least 4 weeks prior to Visit 1 and the therapy is intended to be constant throughout the course of the study.

#### 9.2.2. Prohibited Medications and Procedures

Prohibited medications and procedures include the following:

Received within 4 weeks of Visit 1 or planning to take during participation in the
clinical study: any doses of a controlled-release (CR) CD-LD apart from a single
daily bedtime dose or any doses of Rytary, additional CD (eg, Lodosyn) or
benserazide (eg, Serazide), or catechol-O-methyl transferase inhibitors (entacapone or
tolcapone) or medications containing these inhibitors (Stalevo).

- Rescue with additional or modified doses of concomitant PD medications or with use
  of CD-LD products other than the dispensed study medications is not permitted and
  will trigger discontinuation from the study.
- Received within 4 weeks of Visit 1 or planning to take during participation in the clinical study: nonselective MAOI, selective MAO type A inhibitor (eg, phenelzine, moclobemide, pirlindole, bifemelane, toloxatone), apomorphine, or antidopaminergic agents including antiemetics.
- Treatment with any dopamine antagonist antipsychotic agents for the purposes of psychosis or bipolar disorder within the last 2 years. Use of antipsychotics to treat conditions other than psychosis or bipolar disorders may be allowed only after consultation with the medical monitor.
- Any neurosurgical procedure for the treatment of PD during the course of the study.

A subject who reports the use of any prohibited medications or procedure will be discontinued.

All medications taken within 30 days prior to signing the informed consent form (ICF) and all concomitant medications taken during the study will be recorded on the case report form (CRF).

#### 9.2.3. Rescue Medications

Rescue with additional or modified doses of concomitant non-CD-LD PD medications is not permitted and will trigger discontinuation from the study. During the dose adjustment and dose conversion periods, rescue with CD-LD products other than the dispensed study medications is not permitted and will trigger discontinuation from the study. No medication adjustments are allowed following randomization and during the double-blind phase of the study and will trigger discontinuation from the study.

## 9.3. Treatment Compliance

Study drug accountability and reconciliation will be performed by the study staff and the study monitor(s).

# 9.4. Randomization and Blinding

At Visit 4, subjects will be randomized, stratified by center, in a 1:1 ratio into one of two double-blind parallel treatment arms of IPX203 (and matching IR CD-LD placebo) or IR CD-LD (and matching IPX203 placebo).

## 10. STUDY DRUG MATERIALS AND MANAGEMENT

## 10.1. Study Drug

Study drugs include the investigational treatment IPX203 35-140 mg CD-LD (and matching placebo capsules) and the active comparator treatment IR 25-100 mg CD-LD, (and matching placebo tablets).

IPX203 is an extended-release (ER) capsule formulation of CD-LD. Impax will manufacture and provide the IPX203 and matching placebo.

IR CD-LD is commercially available and will be provided by Impax. Matching placebo tablets will be manufactured and provided by Impax.

## 10.2. Study Drug Packaging and Labeling

Impax or designee will provide study medications in bottles with appropriate labeling affixed. Labels on the study medication may include the following information:

- name, address, and phone number of the sponsor
- pharmaceutical dosage form/route of administration, quantity of dosage units, the name/identifier, and strength/potency
- batch and/or code number to identify the contents and packaging operation
- trial reference code (protocol number)
- trial subject identification number/treatment number and where relevant, the visit number
- name of investigator
- directions for use: Take tablet(s) or capsule(s) orally with water as directed.
- for clinical trial use only
- storage information: Store at 25°C (77°F), with excursions permitted to 15°C to 30°C (59°F to 86°F). Protect from light and moisture.
- period of use (use-by date, expiry date or retest date as applicable), in month/year format and in a manner that avoids any ambiguity.
- keep out of reach of children
- caution statement: Caution: New Drug—Limited by Federal (or United States) law to investigational use.

# 10.3. Study Drug Storage

The clinical site should store the study drug at 25°C (77°F), with excursions permitted to 15°C to 30°C (59°F to 86°F). The study drug should be stored in a tightly closed container, protected

from light and moisture. Storage temperature excursions above 30°C (86°F) should be reported by the clinical site to Impax or its designee.

## 10.4. Study Drug Administration

Subjects will be instructed to take their medications with approximately 240 mL of room-temperature water. The capsules or tablets should not be crushed or chewed.

IR CD-LD tablets may be split to achieve the required doses.

## 10.5. Study Drug Dispensing and Accountability

The Investigator must ensure that all study medication received at the study site is inventoried and accounted for, and that dispensed study medication is recorded in the subject's source documents, the CRF, and the study medication inventory log. Site personnel must not relabel or reassign study medication to other subjects or to individuals not enrolled in the study. The study monitor verifies medication accountability during monitoring visits.

# 10.6. Study Drug Handling and Disposal

The Investigator must retain and properly store all partially used and unused study medication until authorized by Impax regarding disposition.

## 11. ASSESSMENT OF EFFICACY

## 11.1. Parkinson's Disease Diary

Subjects are to record "asleep," "Off," and "On" without or with (nontroublesome or troublesome) dyskinesias during waking hours every 30 minutes over a 24-hour day. In the PD Diaries, subjects are instructed to indicate for each half-hour their predominant state during most of that period. "Off" is defined as the typical functional state when the medication is no longer providing benefit with regard to mobility, slowness, and stiffness in spite of taking medications. "On" is defined as the typical functional state when a subject has received medication and the medication is providing benefit with regard to mobility, slowness, and stiffness. Dyskinesias are defined as involuntary and irregular twisting and/or turning movements. Dyskinesia movements are usually an effect of medication and occur during "On" time. Nontroublesome dyskinesias do not interfere with function or do not cause meaningful discomfort. Troublesome dyskinesias do interfere with function or do cause meaningful discomfort.

## 11.2. Patient and Global Assessments

Patient Global Impression of Change (Appendix F): The patient will compare his/her condition from the start of the study on a 7-point scale ranging from "Very much worse" (1) to "Very much improved" (7) at the time of the assessment.



# 11.3. Movement Disorders Society Version of Unified Parkinson's Disease Rating Scale

The MDS-UPDRS has 4 parts:

Part I: Non-Motor Aspects of Experiences of Daily Living (nM-EDL) has
2 components. Component IA contains a number of behaviors assessed by the
investigator with all pertinent information from the patients and caregivers.
Component IB is completed by the patient with or without help from the caregiver but
independent of the investigator. These sections can be reviewed by the rater to ensure
all questions are answered clearly and the rater can help explain any ambiguities.

- Part II: Motor Aspects of Experiences of Daily Living (M-EDL) is a selfadministered questionnaire but can be reviewed by the investigator to ensure completeness and clarity.
- Part III: Motor Examination assesses the motor signs of PD and has instructions for the rater to give to or to demonstrate to the patient. It is completed by the rater.
- Part IV: Motor Complications integrates patient-derived information with the rater's
  clinical observations and judgements and is completed by the rater. It contains
  instructions for the rater and instructions to be read to the patient.

## 11.4. Additional Assessments



## 12. ASSESSMENT OF SAFETY

## 12.1. Safety Parameters

Safety will be assessed by the following parameters:

- Electrocardiograms (ECGs), clinical laboratory tests, physical examinations, the Columbia-Suicide Severity Rating Scale (C-SSRS), and vital signs, including supine and standing orthostatic blood pressure and heart rate.
- Adverse events and concomitant medications will be evaluated throughout the course of the study.

## 12.2. Adverse Events

## 12.2.1. Definition of Adverse Event

An adverse event (adverse experience) is any untoward medical occurrence in a patient or clinical trial subject administered a medicinal product and which does not necessarily have to have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign (eg, an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

All AEs and any clinically significant physical examination findings, 12-lead ECG abnormalities, or clinical laboratory measurements occurring during the study that were not present prior to administration of study medication and that continue at Study Exit should be followed and evaluated with additional tests, if necessary, until the AEs are medically stable or resolved. Follow-up on these AEs should be recorded on the source documents and reported to Impax.

#### 12.2.2. Recording Adverse Events

Elicit information about AEs with nonselective questions such as: "Have you experienced any changes in your health status since your last visit?" Encourage subjects to report AEs at onset.

Record information for any AE that emerges from the time the subject signs the ICF until Study Exit.

Monitor each subject closely for the development of AEs and record all such events on the AE page of the CRF. Whenever possible, group signs and symptoms that constitute a single diagnosis. For example, cough, rhinitis, and sneezing might be grouped as upper respiratory infection.

For each AE, record the onset date, severity, seriousness, relationship to study medication, date of resolution (or continuing), action taken, and outcome in the CRF. The Investigator is to make a causality assessment (relationship to study medication) for every AE.

#### **12.2.3.** Follow-up

The Investigator must follow each AE until resolved or medically stable.

## 12.2.4. Relationship to Study Drug

The Investigator documents his/her opinion of the relationship of the AE to the study medication as follows:

- Not Related—the experience can be readily explained by the subject's underlying
  medical condition or concomitant medications and no relationship exists between the
  study medication and the experience.
- Unlikely Related—the temporal relationship between the AE and the administration
  of the study medication is uncertain and it is likely that the AE can be explained by
  the subject's medical condition or other therapies.
- Possibly Related—there is some logical temporal relationship between the AE and the administration of the study medication and the experience is unlikely to be explained by the subject's medical condition or other therapies.
- Related—the temporal relationship is compelling between the administration of the study medication and the AE cannot be explained by the subject's medical condition or other therapies.

## 12.2.5. Assessment of Severity

Grade each AE for severity and note in the description of the AE. Determine the severity category of mild, moderate, or severe, as defined below, and enter the information on the AE page of the CRF.

- Mild—causing no limitation of usual activities
- Moderate—causing some limitation of usual activities
- · Severe—causing inability to carry out usual activities

#### 12.3. Serious Adverse Events

## 12.3.1. Definition of Serious Adverse Event

A serious adverse event (SAE) is any AE occurring at any dose that results in any of the following outcomes, regardless of relationship to the study medication:

- Death
- A life-threatening adverse drug experience
- Inpatient hospitalization or prolongation of existing hospitalization
- A persistent or significant disability/incapacity
- A congenital anomaly/birth defect

Important medical events that may not result in death, be life-threatening, or require
hospitalization may be considered an SAE when, based upon appropriate medical
judgment, they may jeopardize the subject and may require medical or surgical
intervention to prevent one of the outcomes listed in this definition.

## 12.3.2. Reporting Serious Adverse Events

Any SAE that occurs from the time the subject signs an ICF until 30 days after taking the final dose of study medication must be reported by the investigative staff to the Sponsor or the Sponsor's representative within 24 hours of knowledge of the event (see Study Contact Information).

An SAE form must be completed and sent to the Sponsor and/or the Sponsor's representative. All SAEs must also be recorded on the AE page of the CRF. Additionally, all SAEs must be reported to the institutional review board (IRB) per the IRB's requirements.

Those SAEs that are considered both serious and unexpected and related to the study drug are subject to expedited reporting. An "unexpected AE" is any AE where the nature or severity is not consistent with the current investigator brochure (IB) or if an IB is not required or available, the specificity or severity is not consistent with the provided risk information.

Unexpected fatal or life-threatening SAEs related to the study drug must be reported by the Sponsor to the appropriate regulatory authority in an expedited manner (ie, first report within 7 days of first knowledge by the Sponsor). The Sponsor will provide a final written report to that authority within 15 days of initial receipt of information on the event. The Sponsor or the Sponsor's representative will also inform all participating Investigators of the SAE.

Unexpected SAEs that are not fatal or life-threatening must be reported by the Sponsor to the appropriate regulatory authority as soon as possible but no later than 15 calendar days after first knowledge of the SAE by the Sponsor. The Sponsor or the Sponsor's representative also informs all participating Investigators of the SAE.

Subjects withdrawn from the study due to any SAE will be followed until the SAE is resolved or medically stable. Record all SAEs, regardless of severity and whether or not related to the study medication, on the appropriate page of the CRF.

The Investigator must determine whether the seriousness of the event warrants removal of the subject from the study. He/she should, in any case, institute appropriate diagnostic and therapeutic measures and keep the subject under observation for as long as is medically indicated, or refer the subject to appropriate health professionals.

# 12.4. Pregnancy

Any pregnancy that occurs from the time the subject signs an ICF until 30 days after taking the final dose of study medication must be reported within 24 hours to the Sponsor or the Sponsor's representative and the subject should be terminated from the study. All pregnancies will be followed through to delivery of the infant. If the subject experiences a termination of the pregnancy, it should be reported as defined in Section 12.3.2.

# 12.5. Other Safety Parameters and Related Information

Additional safety parameters (laboratory tests, 12-lead ECGs, physical examinations, and vital signs), the C-SSRS, the GCSI, and concomitant medications are collected as shown in the Schedule of Assessments in Table 4. Clinical laboratory assessments are listed in Appendix R.

## 13. STATISTICS

## 13.1. Study Design and Sample Size Estimation

This is a multicenter, randomized, double-blind, double-dummy, active-controlled, parallel-group study. Assuming a difference of 1 hour between IPX203 and IR CD-LD in "Good on" time and a standard deviation of the treatment differences to be 3.0 hours, a sample size of 210 subjects per arm will be needed to ensure at least 90% power at a 0.05 significance level.

Assuming approximately an 18% prerandomization drop-out, approximately 510 subjects would need to be enrolled to randomize 420 subjects.

## 13.2. Demographics/Baseline Comparability

The demographics and baseline characteristics will be summarized by treatment arms and overall using descriptive statistics. Demographics information includes age, sex, and race. Baseline disease characteristics include MDS-UPDRS Parts I, II, III, and IV, Hoehn and Yahr stage, MoCA scores, and age of onset of PD. Distributions of dosing information, including LD doses and years on LD, will also be summarized.

## 13.3. Efficacy Endpoints

- Primary endpoint: Change from baseline in "Good on" time in hours per day, averaged over the PD Diary days, at the end of double-blind treatment period (Visit 7 or early termination).
   "Good on" time is derived from the 3-day PD Diaries and is defined as the sum of "On" time without dyskinesia and "On" time with nontroublesome dyskinesia.
- Key secondary endpoints:
  - Change from baseline in "Off" time in hours per day, averaged over the PD Diary days at the end of double-blind treatment period (Visit 7 or early termination)
  - Proportion of subjects with either "much improved" or "very much improved" in Patient Global Impression of Change (PGI-C) scores at the end of double-blind treatment period (Visit 7 or early termination)
  - Change from baseline in the MDS-UPDRS Part III at the end of double-blind treatment period (Visit 7 or early termination)
  - Change from baseline in the sum of MDS-UPDRS Parts II and III at the end of double-blind treatment period (Visit 7 or early termination)

## Additional endpoints:

The following endpoints will be evaluated (at the post-randomization visits) as change from baseline (Visit 4) as well as change from the study entry (Visit 1), when applicable, by visits:





## 13.4. Analysis of Efficacy Data

In order to control the type I error rate, the primary efficacy endpoint and key secondary efficacy endpoints will be tested in a single hierarchical order as detailed in Section 13.8.

## 13.4.1. Primary Efficacy Endpoint

The primary efficacy endpoint is the mean change from baseline in "Good on" time in hours per day, averaged over the PD Diary days, at the end of the double-blind therapy (Visit 7 or early termination). "Good on" time is derived from the 3-day PD Diaries. For each day, "Good on" time is calculated by adding the number of half-hour intervals in which either an "On without dyskinesia" or "On with nontroublesome dyskinesia" is checked.

The primary efficacy endpoint will be analyzed using a mixed model for repeated measures (MMRM). The model will include baseline (Visit 4) "Good on" time as a covariate, treatment, visit, and pooled center as fixed effects, and a treatment-by-visit interaction. The model will employ an unstructured within subject covariance matrix and a restricted maximum likelihood (ReML) estimation method. The degree-of-freedom of the denominator will be estimated using the Kenward-Roger method (Kenward and Roger 1997). The primary analysis population will be the modified intent-to-treat as defined in Section 13.9. Missing data will be handled as in Section 13.10.

If the model fails to converge due to the unstructured covariance matrix, a simpler covariance matrix will be employed in the order of 1) heterogeneous Toeplitz [SAS PROC MIXED type = TOEPH], 2) heterogeneous autoregressive of order 1 [type = ARH(1)], 3) heterogeneous compound symmetry [type = CSH], 4) Toeplitz [type = TOEP], 5) autoregressive of order 1 [type = AR(1)], 6) compound symmetry [type = CS]. The first covariance structure that does not have a convergence problem will be the one used for the primary analysis.

## 13.4.2. Key Secondary Efficacy Endpoints

The first key secondary endpoint is the mean change from baseline in "Off" time in hours per day, averaged over the PD Diary days, at the end of the double-blind therapy (Visit 7 or early termination). "Off" time is derived from the 3-day PD Diaries. For each day, "Off" time is calculated by adding the number of half-hour intervals in which an "Off" is checked. This endpoint will be analyzed using a MMRM model with baseline (Visit 4) "Off" time as a covariate, treatment, visit, and pooled center as fixed effects, and a treatment-by-visit interaction. The model will employ an unstructured within subject covariance matrix and a restricted maximum likelihood (ReML) estimation method. The degree-of-freedom of the denominator will be estimated using the Kenward-Roger method (Kenward and Roger 1997).

The proportion of subjects with either "much improved" or "very much improved" in PGI-C scores at the end of the double-blind therapy (Visit 7 or early termination), the second key secondary endpoint, will be analyzed using a Cochran-Mantel-Haenszel test to compare the two treatment groups with pooled center as a stratification factor.

The mean change from baseline in the MDS-UPDRS Part III at the end of the double-blind therapy (Visit 7 or early termination) is the third key secondary endpoint. This endpoint will be analyzed using an MMRM model with baseline (Visit 4) MDS-UPDRS Part III as a covariate,

treatment, visit, and pooled center as fixed effects, and a treatment-by-visit interaction. The model will employ an unstructured within subject covariance matrix and a restricted maximum likelihood (ReML) estimation method. The degree-of-freedom of the denominator will be estimated using the Kenward-Roger method (Kenward and Roger 1997).

The mean change from baseline in sum of the MDS-UPDRS Parts II and III at the end of the double-blind therapy (Visit 7 or early termination) is the fourth key secondary endpoint. This endpoint will be analyzed using an MMRM model with baseline (Visit 4) MDS-UPDRS Parts II and III combined as covariates, treatment, visit, and pooled center as fixed effects, and a treatment-by-visit interaction. The model will employ an unstructured within subject covariance matrix and a restricted maximum likelihood (ReML) estimation method. The degree-of-freedom of the denominator will be estimated using the Kenward-Roger method (Kenward and Roger 1997).

For the 4 key secondary endpoints, the analysis population will be the modified intent-to-treat as defined in Section 13.9. Missing data will be handled as in Section 13.10.

## 13.4.3. Additional Efficacy Endpoints

In general, continuous endpoints will be summarized by standard descriptive statistics (mean, standard deviation, median, minimum, and maximum). Categorical endpoints will be summarized by frequencies and percentages. Comparisons between the two arms will be explored using appropriate statistical methodologies. Details will be provided in the SAP.

The primary endpoint, key secondary endpoints, as well as other efficacy endpoints will be presented by visit over the whole blinded treatment period from Baseline (Visit 4) to the end of the double-blind treatment period (Visit 7).

Other additional efficacy endpoints collected postrandomization will be analyzed by visit in a fashion similar to the primary and key secondary endpoints.

Additionally the PGI-C and will be analyzed using analysis of variance (ANOVA) with treatment and pooled center as factors.

# 13.5. Center Pooling Algorithm

The center pooling algorithm is as follows.

- 1. Sort centers from each country from smallest to largest based on the number of subjects in the modified intent-to-treat analysis set (mITT).
- Centers with less than 5 mITT subjects or at least one mITT subject per treatment group
  will be pooled with the next smallest center in the same country until the combined center
  (namely, pseudo-center) has more than 5 mITT subjects and at least one mITT subject
  per treatment group.
- 3. If after pooling within the same country, the pseudo-center still has less than 5 mITT subjects or still has zero subjects in one of the treatment group, that pseudo-center will be pooled with the next smallest center in the same geographical region (Western Europe, Eastern Europe, North America).

4. If after pooling within the same geographical region, the pseudo-center still has less than 5 mITT subjects or still has zero subjects in one of the treatment group, that pseudo-center will be pooled with the next smallest center in any region.

The process continues until all pooled pseudo-centers have at least 5 mITT subjects and at least one mITT subject per treatment group. These pooled centers will be used in analyses that adjust for pooled centers.

This pooling algorithm will be detailed in the Statistical Analysis Plan (SAP).

# 13.6. Sensitivity Analyses of the Primary Endpoint and Key Secondary Endpoints

Sensitivity analyses will be performed with respect to the primary efficacy endpoint and continuous key secondary endpoints ("Off" time, MDS-UPDRS Part III, and MDS-UPDRS Parts II and III combined) as follows.

#### 13.6.1. Assessing Assumptions of the Mixed Model for Repeated Measures (MMRM)

- a. The normality and homoscedasticity assumptions will be examined through residual analyses. The normality and homoscedasticity assumptions will further be tested via Shapiro-Wilk (Shapiro and Wilk 1965) and Levene (Levene 1960) tests, respectively, at a 0.05 level of significance. If normality and/or homoscedasticity assumption appears violated, then:
  - Nonparametric Wilcoxon Rank Sum test will be performed to compare the two treatment groups, with missing data imputed by the last observation carried forward (LOCF) method.
  - ii. Multiple imputation rank based analysis: instead of missing data imputed by the LOCF method, in this analysis, missing data at Visit 7 will be imputed multiple times to create 50 complete datasets. The multiple imputation procedure is described in Section 13.6.4 (part of the pattern-mixture model), using f = 0%. The Wilcoxon Rank Sum test will be performed on each of the 50 datasets. The results are then combined using Rubin's rule (Rubin 1987) via SAS PROC MIANALYZE.
- b. Missing at Random (MAR) assumption will be evaluated as discussed in Section 13.6.4.

#### 13.6.2. Complete Case Analysis

The primary endpoint will be analyzed using an ANCOVA model with "Good on" time at baseline (Visit 4) as a covariate, pooled center and treatment as factors. The model will be performed on subjects with <u>both</u> baseline "Good on" time and Visit 7 "Good on" time.

#### 13.6.3. Single LOCF/BLOCF Imputation

The primary efficacy endpoint will be analyzed using an ANCOVA model with "Good on" time at Visit 4 as a covariate, pooled center and treatment as factors. Missing data will be imputed by the LOCF and baseline observation carried forward (BLOCF) methods. These analyses will be performed on the mITT population.

#### 13.6.4. Pattern-Mixture Model

If an overall dropout rate postrandomization is > 15%, pattern-mixture models (PMM) will be employed to assess the robustness of the results under the missing not at random (MNAR) assumption. The pattern for PMM is defined by patients' last visit with an observed primary efficacy endpoint and the reason for dropout.

Multiple imputation with mixed missing data mechanism (MNAR for a missing data pattern and MAR for others) will be used to investigate the robustness of the primary result. Four specific data patterns will be examined:

- 1. Dropout at Visit 5 and reason = Lack of efficacy in IPX203 treatment arm,
- 2. Dropout at Visit 5 and reason = Lack of efficacy or adverse events in IPX203 treatment arm,
- 3. Dropout at Visit 6 and reason = Lack of efficacy in IPX203 treatment arm,
- 4. Dropout at Visit 6 and reason = Lack of efficacy or adverse events in IPX203 treatment arm.

The missing values will be imputed 50 times (multiple imputation) under the assumption that the distribution of the missing values is the same as that of the observed values. The PMM then investigates the departure from the MAR assumption by progressively decreasing the outcome (the "penalty") for those on IPX203 arm who fall into an assumed MNAR pattern above. For the dropout subjects on IPX203 arm that fall into one of the patterns above, the "penalty" is obtained by subtracting the imputed missing data after dropout by a factor f, with f starts from 0%, 5%, 10%, 15%, 20%, 25%, 30%, ..., 100% of the treatment difference seen in the primary model. This process continues until the conclusion from the primary analysis is overturned (a tipping point). In other words, if the dropout subject is from IPX203 arm and the dropout pattern falls into one of the 4 patterns above, then the subject's imputed value will be adjusted downward by a factor f, where f goes from 0% to 100% of the treatment difference seen in the primary model. Note that if 0% is used, the analysis is essentially multiple imputation under MAR assumption. On the other hand, if 100% is used, then the analysis is essentially a "jump to reference" where outcome on IPX203 arm is assumed to be the same as outcome on IR CD-LD. After imputations, the dataset will be analyzed using an MMRM model similar to the primary analysis model. The results will then be combined using the Rubin's rule (Rubin 1987) via SAS PROC MIANALYZE.

The procedure will be carried out in SAS as follows:

- a. Use Monte Carlo Markov Chain (MCMC) method in SAS PROC MI by treatment group to impute the intermittent missing data to form monotone missingness.
- Use MAR-based multiple imputation in SAS PROC MI to impute the missing data (SAS MONOTONE statement).
- c. For dropout subjects in IPX203 arm who fall into an MNAR pattern specified above, a delta which equals to f times the treatment difference obtained from the primary MMRM analysis at Visit 7 will be subtracted from their imputed values for all visits after the dropout ("penalizing" IPX203 arm).

- d. After imputation, use the MMRM model as in the primary analysis model to analyze the complete data along with the imputed data.
- e. Repeat steps a through d 50 times.

Combine results using Rubin's rule (Rubin 1987) via SAS PROC MIANALYZE.

## 13.7. Subgroup Analyses

The primary, key secondary endpoints, as well as overall summary of adverse events, will be examined for the following subgroups.

- Age:  $< 65, \ge 65$  years old at study entry
- Sex: Males, Females
- Race: Caucasians, non-Caucasians

Additionally, the following subgroups may be examined:

- Region
- Ethnicity
- Concomitant medications
- Weight
- Body mass index (BMI)
- PD duration
- Age of PD onset
- "Good On" time and "Off" time at study entry.

For all subgroup efficacy analyses, the same analysis methods as the primary and key secondary endpoints will be applied, unless the sample size in one of the subgroups becomes too small to hinder the statistical analysis. In that case, no inferential statistics will be provided for such a subgroup. The details for final subgroup analyses will be documented in the SAP.

# 13.8. Multiplicity Adjustments

The primary endpoint and 4 key secondary endpoints will be tested in a sequential hierarchical order as follows.

- 1. The primary endpoint, the mean change from baseline in "Good on" time (hours per day), will be tested first at a 0.05 level of significance.
- 2. If statistical significance is demonstrated, then the first key secondary endpoint, the mean change from baseline in "Off" time (hours per day), will be tested next at a 0.05 level of significance.
- 3. If statistical significance is demonstrated, then the second key secondary endpoint, the proportion of subjects with either "much improved" or "very much improved" on the PGI-C, will be tested next at a 0.05 level of significance.

- 4. If statistical significance is demonstrated, then the third key secondary endpoint, the mean change from baseline in the MDS-UPDRS Part III, will be tested at a 0.05 level of significance.
- 5. If statistical significance is demonstrated, then the fourth key secondary endpoint, the mean change from baseline in the sum of the MDS-UPDRS Parts II and III combined will be tested next at a 0.05 level of significance.

For the other efficacy endpoints, no adjustment will be made.

## 13.9. Analysis Populations

## 13.9.1. Safety Analysis Set

The Safety Analysis set will include all subjects who were treated with any study drug.

## 13.9.2. Intent-to-Treat Analysis Set

The Intent-to-treat Analysis Set will include all subjects who were randomized and treated with any study drug and have a baseline and at least one postbaseline efficacy assessment.

## 13.9.3. Modified Intent-to-Treat Analysis Set

The Modified Intent-to-treat Analysis Set will include all subjects who were randomized and treated and have a valid baseline PD Diary and at least one valid postrandomization PD Diary. This analysis set will be used for the primary analysis and key secondary analyses.

#### 13.9.4. Completers Analysis Set

The Completers Analysis Set will include all subjects who were randomized and treated and complete the study.

## 13.10. Handling of Missing Data

## 13.10.1. Missing Data for PD Diaries

An MMRM approach will be used to handle missing visit data. MMRM analysis will use all available valid visit data, including subjects with some missing visit data, in order to arrive at an estimate of the mean treatment effect.

A PD Diary is valid if at least 1 day of diary data is available using the rules defined below.

Imputation of missing data for a PD Diary day will be required if a PD Diary is not completed for a full day (6 am to 5:30 am). In this case, the method of imputation will be dependent upon the amount and pattern of missing data.

- For subjects with more than 1 day of diary data, the following rules will apply:
  - 1. If more than 4 half-hour time intervals are missing, then that particular day will not be included in the analysis. The missing data will be handled in the MMRM model.
  - 2. If a one-half hour time interval is missing and the observations on either side of the time interval are not missing, then the missing time interval will be imputed by

assigning a value of the previous measurement for the first 15 minutes and the value of the next measurement for the second 15 minutes.

- 3. If 2, 3, or 4 consecutive half-hour time intervals are missing, and these time intervals are available from other days of the visit then the following rules will be applied:
  - a. For missing time intervals on Day 1, data from Day 2 will be used for imputation for the same time intervals. If Day 2 data is also incomplete or not available, then Day 3 data will be used.
  - b. For missing time intervals on Day 2, data from Day 3 will be used for imputation if available; otherwise Day 1 data will be used.
  - c. Data from Day 2 will be used for imputing missing time intervals on Day 3. If data from Day 2 is not available, then Day 1 data will be used for imputation.
  - d. If data at the same time period are missing across all days, then the approach will be to split the individual missing half-hour intervals into 2 periods, with the first-half interval being imputed with data from the immediate previous nonmissing time period and the second-half interval being imputed with the next nonmissing time interval.
- For subjects with only 1 day of diary data, the following rules will apply:
  - 1. If more than 4 half-hour time intervals are missing, then that particular day will not be included in the analysis. The missing data will be handled in the MMRM model.
  - 2. If a one-half hour time interval is missing and the observations on either side of the time interval are not missing, then the missing time interval will be imputed by assigning a value of the previous measurement for the first 15 minutes and the value of the next measurement for the second 15 minutes.
  - 3. If 2, 3, or 4 consecutive half-hour intervals are missing, then the approach will be to split the individual missing half-hour intervals into 2 periods, with the first-half interval being imputed with data from the immediate previous nonmissing time period and the second-half interval being imputed with the next nonmissing time interval.

# 13.10.2. Missing Data for Global Assessments (PGI-C,

For subjects with missing PGI-C or for a particular visit, the data will be imputed as nonresponders (ie, not being "much improved").

## 13.10.3. Missing Data for MDS-UPDRS

If the MDS-UPDRS are missing for the particular visit, the missing data will be handled via the MMRM model.

If component questions are missing for a particular part of the MDS-UPDRS questionnaire, the missing items are assigned the average value for other items in that part as follows (Goetz 2015):

- For Part I (13 questions): up to 1 missing question will be imputed using the average value of the remaining 12 questions.
- For Part II (13 questions): up to 2 missing questions will be imputed using the average value of the remaining 11 questions.
- For Part III (33 questions): up to 7 missing questions will be imputed using the average value of the remaining 26 questions.
- Part IV (6 questions): no imputation is done.

If more component questions are missing than above for a particular part of the MDS-UPDRS questionnaire, the entire questionnaire will not be included in the analysis for that particular assessment. Missing data will be handled in a fashion similar to PD Diary data (Section 13.10.1) using the MMRM model.

For quality-of-life endpoints, missing responses within a questionnaire will not be imputed.

## 13.11. Analysis of Safety

The safety analysis will include all subjects who receive at least 1 dose of study medication. Reported AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). All AEs will be summarized by system organ class and preferred terms within system organ class. The severity, seriousness, and relationship to study medication will also be summarized by treatment arms. Each AE (based on preferred term) is counted once for a given subject. If the same AE occurred on multiple occasions, the highest severity and least complimentary relationship will be assumed.

The incidence of treatment-emergent AEs and serious AEs will be summarized by treatment arms.

Additionally, laboratory test data, physical examinations, vital signs, ECGs, C-SSRS, and GCSI will be summarized by treatment arms.

## 14. ADMINISTRATIVE PROCEDURES

#### 14.1. Guidelines for Good Clinical Practice

This study will be conducted in accordance with principles of Good Clinical Practice (GCP) as promulgated by the ICH. Good Clinical Practice is an international ethical and scientific quality standard for designing, conducting, recording, and reporting trials that involve the participation of human subjects. Compliance with this standard provides public assurance that the rights, safety, and well-being of human subjects are protected under current ethical principles, and that the clinical trial data are credible. Current GCP standards may be found in ICH Guidance E6 (Good Clinical Practice: Consolidated Guidance). This guidance describes the principles of GCP and the obligations of the institutional review board (IRB), the Investigator and the Sponsor in conducting this study in accordance with those principles.

## 14.2. Institutional Review Board Approval

The review of this protocol by an IRB and the performance of all aspects of the study, including the methods used for obtaining informed consent, must be in accordance with principles enunciated in the ICH and GCP Guidelines and by the appropriate regulatory authorities.

The Investigator is responsible for preparing documents for submission to the relevant IRB and obtaining written approval for this study. Institutional Review Board approval must be obtained prior to the initiation of the study. The Investigator's continued participation in the study is contingent on renewing approval with the IRB at least annually.

#### 14.3. Informed Consent

Site personnel should prepare an Informed Consent Form (ICF) incorporating the necessary elements of consent. The ICF is to be approved by Impax prior to submission to the IRB. The Investigator or his/her staff must explain the nature of the investigation and the risks involved to each subject prior to screening, and obtain a signed ICF. The subject should also be informed that he/she is free to voluntarily withdraw from the study at any time.

# 14.4. Study Monitoring

Impax representatives or designees will conduct site visits to the investigational facilities for the purpose of monitoring the study. The Investigator agrees to allow the monitor to inspect the drug storage area, study drug stocks, drug accountability records, subject charts and study source documents, and other records relevant to study conduct. The Investigator must permit access to such records if a regulatory or compliance audit is required.

#### 14.5. Protocol Amendments

All amendments to the protocol must be documented in writing, reviewed and approved by the Sponsor and Investigator, and submitted to the IRB for approval prior to implementation. If the protocol amendment substantially alters the study design or potential risk to the subject, a new

written ICF for continued participation in the study must be obtained from each subject affected by the change.

## 14.6. Termination of Study

The Sponsor has the right to terminate this study and remove all study material from the site at any time for medical or administrative reasons. In this event, the Sponsor will endeavor to give adequate notice to allow safe withdrawal of subjects from the study.

## 14.7. Case Report Forms

Site personnel should collect and record data for the study as source documents, and transfer the data into the CRF.

The Investigator must ensure that complete data for the clinical study are collected and accurately documented in the appropriate sections of the CRF and adequately supported by the appropriate source documentation. In addition, it is the Investigator's responsibility to provide signatures where requested indicating concurrence with data in the CRF.

## 14.8. Investigator's Final Conduct Report

At the completion of the study, the Investigator must provide Impax a copy of the final conduct report that was submitted to their IRB, including a review of AEs.

#### 14.9. Records Retention

International Conference on Harmonization, GCP, and US FDA guidelines require that essential documents be retained until at least 2 years after the last approval of a marketing application and until there are no pending or contemplated marketing applications, or at least 2 years have elapsed since the formal discontinuation of clinical development of the investigational product.

However, the essential documents should be retained for a longer period if required by the applicable regulatory requirements or by an agreement with the Sponsor. Records should never be destroyed without written approval from the Sponsor.

If an Investigator leaves the institution, he/she must transfer responsibilities for record retention to another individual willing to accept them. The Investigator must notify the Sponsor in writing of the transfer of study documents before the transfer of the study documents.

# 15. PUBLICATION POLICY

Study results may not be published without prior written approval from Impax.

## 16. LIST OF REFERENCES

Blanchet PJ, Calon F, Martel JC, et al. Continuous administration decreases and pulsatile administration increases behavioral sensitivity to a novel dopamine D2 agonist (U-91356A) in MPTP-exposed monkeys. J Pharmacol Exp Ther. 1995;272:854-859.

Engber TM, Susel Z, Juncos JL, Chase TN. Continuous and intermittent levodopa differentially affect rotation induced by D-1 and D-2 dopamine agonists. European Journal of Pharmacology. 1989;168:291-298.

Fahn S. Parkinson disease, the effect of levodopa, and the ELLDOPA trial. Earlier vs Later L DOPA. Arch Neurol. 1999 May;56(5):529-35.

Food and Drug Administration 2003. Guidance for Industry. Bioavailability and Bioequivalence Studies for Orally Administered Drug Products — General Considerations. U.S. Department of Health and Human Services. Food and Drug Administration. Center for Drug Evaluation and Research (CDER). March 2003.

Goetz CG, Luo S, Wang L, Tilley BC, LaPelle NR, Stebbins GT. Handling missing values in the MDS-UPDRS. Mov Disord. 2015 Oct;30(12):1632-8.

Juncos JL, Engber TM, Raisman R, et al. Continuous and intermittent levodopa differentially affect basal ganglia function. Ann Neurol. 1989;25:473-478.

Kenward MG and Roger JH. Small sample inference for fixed effects from restricted maximum likelihood. Biometrics. 1997;53:983-997.

Kurlan R, Rothfield KP, Woodward WR, Nutt JG, Miller C, Lichter D, et al. Erratic gastric emptying of levodopa may cause "random" fluctuations of parkinsonian mobility. Neurology. 1988;38(3):419-21.

Levene H. In contributions to probability and statistics: Essays in honor of Harold Hotelling, I. Olkin et al. eds. Stanford University Press. 1960: 278-292.

Melamed E, Bitton V, Zelig O. Delayed onset of responses to single doses of L-dopa in parkinsonian fluctuators on long-term L-dopa therapy. Clin Neuropharmacol. 1986;9(2):182-8.

Mizuno Y. Where do we stand in the treatment of Parkinson's disease? Neurology. 2007;254:13-18.

Nilsson D, Nyholm D, Aquilonius S-M. Duodenal levodopa infusion in Parkinson's diseaselong-term experience. Acta Neurologica Scandinavica. 2001;104:343-348.

Nyholm D, Nilsson Remahl AI, Dizdar N, et al. Duodenal levodopa infusion monotherapy vs oral polypharmacy in advanced Parkinson disease. Neurology. 2005;64:216-223.

Rubin DB. Multiple Imputation in Nonresponse in Surveys. San Francisco, CA: Wiley; 1987.

Shapiro SS and Wilk MB. An analysis of variance test for normality (complete samples). Biometrika. 1965;52(3-4): 591-611.

Sinemet (Carbidopa-Levodopa) Tablets Prescribing Information. Whitehouse Station, NJ: Manufactured by Merck & Co., Inc.; Marketed by Bristol-Myers Squibb Company; 2013.

Stocchi F, Quinn NP, Barbato L, Patsalos PN, O'Connel MT, Ruggieri S, et al. Comparison between a fast and a slow release preparation of levodopa and a combination of the two: a clinical and pharmacokinetic study. Clinical Neuropharmacol. 1994;17(1):38-44.

Stocchi F, Vacca L, et al. Intermittent vs continuous levodopa administration in patients with advanced Parkinson disease: a clinical and pharmacokinetic study. Arch Neurol. 2005:62(6):905-910.

# 17. APPENDICES

# APPENDIX A. PRESCRIBING INFORMATION FOR IR CD-LD

SINEMET - carbidopa and levodopa tablet Merck Sharp & Dohme Corp.

-----

SINEMET<sup>®</sup> (carbidopa levodopa) Tablets

#### DESCRIPTION

SINEMET $^{\$}$  (carbidopa levodopa) is a combination of carbidopa and levodopa for the treatment of Parkinson's disease and syndrome.

Carbidopa, an inhibitor of aromatic amino acid decarboxylation, is a white, crystalline compound, slightly soluble in water, with a molecular weight of 244.3. It is designated chemically as (—)-L- $\alpha$ -bydrazino- $\alpha$ -methyl- $\beta$ -(3,4-dihydroxybenzene) propanoic acid monohydrate. Its empirical formula is  $G_{10}H_{14}N_2O_4$ • $H_2O$ , and its structural formula is:

Tablet content is expressed in terms of anhydrous carbidopa which has a molecular weight of 226.3.

Levodopa, an aromatic amino acid, is a white, crystalline compound, slightly soluble in water, with a molecular weight of 197.2. It is designated chemically as (—)-L- $\alpha$ -amino- $\beta$ -(3,4-dihydroxybenzene) propanoic acid. Its empirical formula is  $C_9H_{11}NO_4$ , and its structural formula is:

SINEMET is supplied as tablets in three strengths:

SINEMET 25-100, containing 25 mg of carbidopa and 100 mg of levodopa.

SINEMET 10-100, containing 10 mg of carbidopa and 100 mg of levodopa.

SINEMET 25-250, containing 25 mg of carbidopa and 250 mg of levodopa.

Inactive ingredients are hydroxypropyl cellulose, pregelatinized starch, crospovidone, microcrystalline cellulose, and magnesium stearate. SINEMET 10-100 and 25-250 Tablets also contain FD&C Blue #2/Indigo Carmine AL. SINEMET 25-100 Tablets also contain D&C Yellow #10 Lake.

#### CLINICAL PHARMACOLOGY

#### Mechanism of Action

Parkinson's disease is a progressive, neurodegenerative disorder of the extrapyramidal nervous system affecting the mobility and control of the skeletal muscular system. Its characteristic features include resting tremor, rigidity, and bradykinetic movements. Symptomatic treatments, such as levodopa therapies, may permit the patient better mobility.

Current evidence indicates that symptoms of Parkinson's disease are related to depletion of dopamine in the corpus striatum. Administration of dopamine is ineffective in the treatment of Parkinson's disease apparently because it does not cross the blood-brain barrier. However, levodopa, the metabolic precursor of dopamine, does cross the blood-brain barrier, and presumably is converted to dopamine in the brain. This is thought to be the mechanism whereby levodopa relieves symptoms of Parkinson's disease.

#### **Pharmacodynamics**

When levodopa is administered orally, it is rapidly decarboxylated to dopamine in extracerebral tissues so that only a small portion of a given dose is transported unchanged to the central nervous system. For this reason, large doses of levodopa are required for adequate therapeutic effect, and these may often be accompanied by nausea and other adverse reactions, some of which are attributable to dopamine formed in extracerebral tissues.

Since levodopa competes with certain amino acids for transport across the gut wall, the absorption of levodopa may be impaired in some patients on a high protein diet.

Carbidopa inhibits decarboxylation of peripheral levodopa. It does not cross the blood-brain barrier and does not affect the metabolism of levodopa within the central nervous system.

The incidence of levodopa-induced nausea and vomiting is less with SINEMET than with levodopa. In many patients, this reduction in nausea and vomiting will permit more rapid dosage titration.

Since its decarboxylase inhibiting activity is limited to extracerebral tissues, administration of carbidopa with levodopa makes more levodopa available for transport to the brain.

#### **Pharmacokinetics**

Carbidopa reduces the amount of levodopa required to produce a given response by about 75% and, when administered with levodopa, increases both plasma levels and the plasma half-life of levodopa, and decreases plasma and urinary dopamine and homovanillic acid.

The plasma half-life of levodopa is about 50 minutes, without carbidopa. When carbidopa and levodopa are administered together, the half-life of levodopa is increased to about 1.5 hours. At steady state, the bioavailability of carbidopa from SINEMET tablets is approximately 99% relative to the concomitant administration of carbidopa and levodopa.

In clinical pharmacologic studies, simultaneous administration of carbidopa and levodopa produced greater urinary excretion of levodopa in proportion to the excretion of dopamine than administration of the two drugs at separate times.

Pyridoxine hydrochloride (vitamin  $B_6$ ), in oral doses of 10 mg to 25 mg, may reverse the effects of levodopa by increasing the rate of aromatic amino acid decarboxylation. Carbidopa inhibits this action of pyridoxine; therefore, SINEMET can be given to patients receiving supplemental pyridoxine (vitamin  $B_6$ ).

#### **Special Populations**

#### Geriatric

A study in eight young healthy subjects (21-22 yr) and eight elderly healthy subjects (69-76 yr) showed that the absolute bioavailability of levodopa was similar between young and elderly subjects following oral administration of levodopa and carbidopa. However, the systemic exposure (AUC) of levodopa was increased by 55% in elderly subjects compared to young subjects. Based on another study in forty patients with Parkinson's disease, there was a correlation between age of patients and the increase of AUC of levodopa following administration of levodopa and an inhibitor of peripheral dopa decarboxylase. AUC of levodopa was increased by 28% in elderly patients ( $\geq$  65 yr) compared to young patients ( $\leq$  65 yr). Additionally, mean value of Cmax for levodopa was increased by 24% in
elderly patients (≥ 65 yr) compared to young patients (< 65 yr) (see PRECAUTIONS, Geriatric Use).

The AUC of carbidopa was increased in elderly subjects (n=10, 65-76 yr) by 29% compared to young subjects (n=24, 23-64 yr) following IV administration of 50 mg levodopa with carbidopa (50 mg). This increase is not considered a clinically significant impact.

#### INDICATIONS AND USAGE

SINEMET is indicated in the treatment of Parkinson's disease, post-encephalitic parkinsonism, and symptomatic parkinsonism that may follow carbon monoxide intoxication or manganese intoxication.

Carbidopa allows patients treated for Parkinson's disease to use much lower doses of levodopa. Some patients who responded poorly to levodopa have improved on SINEMET. This is most likely due to decreased peripheral decarboxylation of levodopa caused by administration of carbidopa rather than by a primary effect of carbidopa on the nervous system. Carbidopa has not been shown to enhance the intrinsic efficacy of levodopa.

Carbidopa may also reduce nausea and vomiting and permit more rapid titration of levodopa.

#### CONTRAINDICATIONS

Nonselective monoamine oxidase (MAO) inhibitors are contraindicated for use with SINEMET. These inhibitors must be discontinued at least two weeks prior to initiating therapy with SINEMET. SINEMET may be administered concomitantly with the manufacturer's recommended dose of an MAO inhibitor with selectivity for MAO type B (e.g., selegiline HCl) (see PRECAUTIONS, Drug Interactions).

SINEMET is contraindicated in patients with known hypersensitivity to any component of this drug, and in patients with narrow-angle glaucoma.

## WARNINGS

When SINEMET is to be given to patients who are being treated with levodopa, levodopa must be discontinued at least twelve hours before therapy with SINEMET is started. In order to reduce adverse reactions, it is necessary to individualize therapy. See DOSAGE AND ADMINISTRATION section before initiating therapy.

The addition of carbidopa with levodopa in the form of SINEMET reduces the peripheral effects (nausea, vomiting) due to decarboxylation of levodopa; however, carbidopa does not decrease the adverse reactions due to the central effects of levodopa. Because carbidopa permits more levodopa to reach the brain and more dopamine to be formed, certain adverse central nervous system (CNS) effects, e.g., dyskinesias (involuntary movements), may occur at lower dosages and sooner with SINEMET than with levodopa alone.

All patients should be observed carefully for the development of depression with concomitant suicidal tendencies.

SINEMET should be administered cautiously to patients with severe cardiovascular or pulmonary disease, bronchial asthma, renal, hepatic or endocrine disease.

As with levodopa, care should be exercised in administering SINEMET to patients with a history of myocardial infarction who have residual atrial, nodal, or ventricular arrhythmias. In such patients, cardiac function should be monitored with particular care during the period of initial dosage adjustment, in a facility with provisions for intensive cardiac care.

As with levodopa, treatment with SINEMET may increase the possibility of upper gastrointestinal hemorrhage in patients with a history of peptic ulcer.

Falling Asleep During Activities of Daily Living and Somnolence

Patients taking SINEMET alone or with other dopaminergic drugs have reported suddenly falling asleep without prior warning of sleepiness while engaged in activities of daily living (includes operation of motor vehicles). Road traffic accidents attributed to sudden sleep onset have been reported. Although many patients reported somnolence while on dopaminergic medications, there have been reports of road traffic accidents attributed to sudden onset of sleep in which the patient did not perceive any warning signs, such as excessive drowsiness, and believed that they were alert immediately prior to the event. Sudden onset of sleep has been reported to occur as long as one year after the initiation of treatment.

Falling asleep while engaged in activities of daily living usually occurs in patients experiencing preexisting somnolence, although some patients may not give such a history. For this reason, prescribers should reassess patients for drowsiness or sleepiness especially since some of the events occur well after the start of treatment. Prescribers should be aware that patients may not acknowledge drowsiness or sleepiness until directly questioned about drowsiness or sleepiness during specific activities. Patients should be advised to exercise caution while driving or operating machines during treatment with SINEMET. Patients who have already experienced somnolence or an episode of sudden sleep onset should not participate in these activities during treatment with SINEMET.

Before initiating treatment with SINEMET, advise patients about the potential to develop drowsiness and ask specifically about factors that may increase the risk for somnolence with SINEMET such as the use of concomitant sedating medications and the presence of sleep disorders. Consider discontinuing SINEMET in patients who report significant daytime sleepiness or episodes of falling asleep during activities that require active participation (e.g., conversations, eating, etc.). If treatment with SINEMET continues, patients should be advised not to drive and to avoid other potentially dangerous activities that might result in harm if the patients become somnolent. There is insufficient information to establish that dose reduction will eliminate episodes of falling asleep while engaged in activities of daily living.

# Hyperpyrexia and Confusion

Sporadic cases of a symptom complex resembling neuroleptic malignant syndrome (NMS) have been reported in association with dose reductions or withdrawal of certain antiparkinsonian agents such as levodopa, carbidopa levodopa, or carbidopa levodopa extended release. Therefore, patients should be observed carefully when the dosage of levodopa is reduced abruptly or discontinued, especially if the patient is receiving neuroleptics.

NMS is an uncommon but life-threatening syndrome characterized by fever or hyperthermia. Neurological findings, including muscle rigidity, involuntary movements, altered consciousness, mental status changes; other disturbances, such as autonomic dysfunction, tachycardia, tachypnea, sweating, hyper- or hypotension; laboratory findings, such as creatine phosphokinase elevation, leukocytosis, myoglobinuria, and increased serum myoglobin have been reported.

The early diagnosis of this condition is important for the appropriate management of these patients. Considering NMS as a possible diagnosis and ruling out other acute illnesses (e.g., pneumonia, systemic infection, etc.) is essential. This may be especially complex if the clinical presentation includes both serious medical illness and untreated or inadequately treated extrapyramidal signs and symptoms (EPS). Other important considerations in the differential diagnosis include central anticholinergic toxicity, heat stroke, drug fever, and primary central nervous system (CNS) pathology.

The management of NMS should include: 1) intensive symptomatic treatment and medical monitoring and 2) treatment of any concomitant serious medical problems for which specific treatments are available. Dopamine agonists, such as bromocriptine, and muscle relaxants, such as dantrolene, are often used in the treatment of NMS; however, their effectiveness has not been demonstrated in controlled studies.

# PRECAUTIONS

General

As with levodopa, periodic evaluations of hepatic, hematopoietic, cardiovascular, and renal function are recommended during extended therapy.

Patients with chronic wide-angle glaucoma may be treated cautiously with SINEMET provided the intraocular pressure is well-controlled and the patient is monitored carefully for changes in intraocular pressure during therapy.

#### Dvs kines ia

Levodopa alone, as well as SINEMET, is associated with dyskinesias. The occurrence of dyskinesias may require dosage reduction.

## Hallucinations / Psychotic-Like Behavior

Hallucinations and psychotic-like behavior have been reported with dopaminergic medications. In general, hallucinations present shortly after the initiation of therapy and may be responsive to dose reduction in levodopa. Hallucinations may be accompanied by confusion and to a lesser extent sleep disorder (insomnia) and excessive dreaming.

SINEMET may have similar effects on thinking and behavior. This abnormal thinking and behavior may present with one or more symptoms, including paranoid ideation, delusions, hallucinations, confusion, psychotic-like behavior, disorientation, aggressive behavior, agitation, and delirium.

Ordinarily, patients with a major psychotic disorder should not be treated with SINEMET, because of the risk of exacerbating psychosis. In addition, certain medications used to treat psychosis may exacerbate the symptoms of Parkinson's disease and may decrease the effectiveness of SINEMET.

## Impulse Control / Compulsive Behaviors

Reports of patients taking dopaminergic medications (medications that increase central dopaminergic tone), suggest that patients may experience an intense urge to gamble, increased sexual urges, intense urges to spend money, binge eating, and/or other intense urges, and the inability to control these urges. In some cases, although not all, these urges were reported to have stopped when the dose was reduced or the medication was discontinued. Because patients may not recognize these behaviors as abnormal, it is important for prescribers to specifically ask patients or the caregivers about the development of new or increased gambling urges, sexual urges, uncontrolled spending or other urges while being treated with SINEMET. Physicians should consider dose reduction or stopping the medication if a patient develops such urges while taking SINEMET [see *Information for Patients*].

# Melanoma

Epidemiological studies have shown that patients with Parkinson's disease have a higher risk (2- to approximately 6-fold higher) of developing melanoma than the general population. Whether the increased risk observed was due to Parkinson's disease or other factors, such as drugs used to treat Parkinson's disease, is unclear.

For the reasons stated above, patients and providers are advised to monitor for melanomas frequently and on a regular basis when using SINEMET for any indication. Ideally, periodic skin examinations should be performed by appropriately qualified individuals (e.g., dermatologists).

# Information for Patients

The patient should be informed that SINEMET is an immediate-release formulation of carbidopa levodopa that is designed to begin release of ingredients within 30 minutes. It is important that SINEMET be taken at regular intervals according to the schedule outlined by the physician. The patient should be cautioned not to change the prescribed dosage regimen and not to add any additional antiparkinson medications, including other carbidopa levodopa preparations, without first consulting the physician.

Patients should be advised that sometimes a 'wearing-off' effect may occur at the end of the dosing interval. The physician should be notified if such response poses a problem to lifestyle.

Patients should be advised that occasionally, dark color (red, brown, or black) may appear in saliva, urine, or sweat after ingestion of SINEMET. Although the color appears to be clinically insignificant, garments may become discolored.

The patient should be advised that a change in diet to foods that are high in protein may delay the absorption of levodopa and may reduce the amount taken up in the circulation. Excessive acidity also delays stomach emptying, thus delaying the absorption of levodopa. Iron salts (such as in multivitamin tablets) may also reduce the amount of levodopa available to the body. The above factors may reduce the clinical effectiveness of the levodopa or carbidopa levodopa therapy.

Patients should be alerted to the possibility of sudden onset of sleep during daily activities, in some cases without awareness or warning signs, when they are taking dopaminergic agents, including levodopa. Patients should be advised to exercise caution while driving or operating machinery and that if they have experienced somnolence and/or sudden sleep onset, they must refrain from these activities. (See WARNINGS, Falling Asleep During Activities of Daily Living and Somnolence.)

There have been reports of patients experiencing intense urges to gamble, increased sexual urges, and other intense urges, and the inability to control these urges while taking one or more of the medications that increase central dopaminergic tone and that are generally used for the treatment of Parkinson's disease, including SINEMET. Although it is not proven that the medications caused these events, these urges were reported to have stopped in some cases when the dose was reduced or the medication was stopped. Prescribers should ask patients about the development of new or increased gambling urges, sexual urges or other urges while being treated with SINEMET. Patients should inform their physician if they experience new or increased gambling urges, increased sexual urges, or other intense urges while taking SINEMET. Physicians should consider dose reduction or stopping the medication if a patient develops such urges while taking SINEMET (See PRECAUTIONS, Impulse Control / Compulsive Behaviors).

# Laboratory Tests

Abnormalities in laboratory tests may include elevations of liver function tests such as alkaline phosphatase, SGOT (AST), SGPT (ALT), lactic dehydrogenase (LDH), and bilirubin. Abnormalities in blood urea nitrogen (BUN) and positive Coombs test have also been reported. Commonly, levels of blood urea nitrogen, creatinine, and uric acid are lower during administration of SINEMET than with levodopa.

SINEMET may cause a false-positive reaction for urinary ketone bodies when a test tape is used for determination of ketonuria. This reaction will not be altered by boiling the urine specimen. False-negative tests may result with the use of glucose-oxidase methods of testing for glucosuria.

Cases of falsely diagnosed pheochromocytoma in patients on carbidopa levodopa therapy have been reported very rarely. Caution should be exercised when interpreting the plasma and urine levels of catecholamines and their metabolites in patients on levodopa or carbidopa levodopa therapy.

#### **Drug Interactions**

Caution should be exercised when the following drugs are administered concomitantly with SINEMET.

Symptomatic postural hypotension occurred when SINEMET was added to the treatment of a patient receiving antihypertensive drugs. Therefore, when therapy with SINEMET is started, dosage adjustment of the antihypertensive drug may be required.

For patients receiving MAO inhibitors (Type A or B), see CONTRAINDICATIONS. Concomitant therapy with selegiline and carbidopa levodopa may be associated with severe orthostatic hypotension not attributable to carbidopa levodopa alone (see CONTRAINDICATIONS).

There have been rare reports of adverse reactions, including hypertension and dyskinesia, resulting from the concomitant use of tricyclic antidepressants and SINEMET.

Dopamine  $D_2$  receptor antagonists (e.g., phenothiazines, butyrophenones, risperidone) and isoniazid may reduce the therapeutic effects of levodopa. In addition, the beneficial effects of levodopa in Parkinson's disease have been reported to be reversed by phenytoin and papaverine. Patients taking these drugs with SINEMET should be carefully observed for loss of therapeutic response.

Use of SINEMET with dopamine-depleting agents (e.g., reserpine and tetrabenazine) or other drugs known to deplete monoamine stores is not recommended.

SINEMET and iron salts or multivitamins containing iron salts should be coadministered with caution. Iron salts can form chelates with levodopa and carbidopa and consequently reduce the bioavailability of carbidopa and levodopa.

Although metoclopramide may increase the bioavailability of levodopa by increasing gastric emptying, metoclopramide may also adversely affect disease control by its dopamine receptor antagonistic properties.

# Carcinogenesis, Mutagenesis, Impairment of Fertility

In a two-year bioassay of SINEMET, no evidence of carcinogenicity was found in rats receiving doses of approximately two times the maximum daily human dose of carbidopa and four times the maximum daily human dose of levodopa.

In reproduction studies with SINEMET, no effects on fertility were found in rats receiving doses of approximately two times the maximum daily human dose of carbidopa and four times the maximum daily human dose of levodopa.

# Pregnancy

No teratogenic effects were observed in a study in mice receiving up to 20 times the maximum recommended human dose of SINEMET. There was a decrease in the number of live pups delivered by rats receiving approximately two times the maximum recommended human dose of carbidopa and approximately five times the maximum recommended human dose of levodopa during organogenesis. SINEMET caused both visceral and skeletal malformations in rabbits at all doses and ratios of carbidopa/levodopa tested, which ranged from 10 times/5 times the maximum recommended human dose of carbidopa/levodopa to 20 times/10 times the maximum recommended human dose of carbidopa/levodopa.

There are no adequate or well-controlled studies in pregnant women. It has been reported from individual cases that levodopa crosses the human placental barrier, enters the fetus, and is metabolized. Carbidopa concentrations in fetal tissue appeared to be minimal. Use of SINEMET in women of childbearing potential requires that the anticipated benefits of the drug be weighed against possible hazards to mother and child.

# **Nursing Mothers**

Levodopa has been detected in human milk. Caution should be exercised when SINEMET is administered to a nursing woman.

#### Pediatric Use

Safety and effectiveness in pediatric patients have not been established. Use of the drug in patients below the age of 18 is not recommended.

# Geriatric Use

In the clinical efficacy trials for SINEMET, almost half of the patients were older than 65, but few were older than 75. No overall meaningful differences in safety or effectiveness were observed between

these subjects and younger subjects, but greater sensitivity of some older individuals to adverse drug reactions such as hallucinations cannot be ruled out. There is no specific dosing recommendation based upon clinical pharmacology data as SINEMET is titrated as tolerated for clinical effect.

## ADVERSE REACTIONS

The most common adverse reactions reported with SINEMET have included dyskinesias, such as choreiform, dystonic, and other involuntary movements, and nausea.

The following other adverse reactions have been reported with SINEMET:

Body as a Whole

Chest pain, asthenia.

Cardiovascular

Cardiac irregularities, hypotension, orthostatic effects including orthostatic hypotension, hypertension, syncope, phlebitis, palpitation.

Gastrointestinal

Dark saliva, gastrointestinal bleeding, development of duodenal ulcer, anorexia, vomiting, diarrhea, constipation, dyspepsia, dry mouth, taste alterations.

Hematologic

Agranulocytosis, hemolytic and non-hemolytic anemia, thrombocytopenia, leukopenia.

Hypersensitivity

Angioedema, urticaria, pruritus, Henoch-Schönlein purpura, bullous lesions (including pemphigus-like reactions).

Musculoskeletal

Back pain, shoulder pain, muscle cramps.

Nervous System/Psychiatric

Psychotic episodes including delusions, hallucinations, and paranoid ideation, bradykinetic episodes ("on-off" phenomenon), confusion, agitation, dizziness, somnolence, dream abnormalities including nightmares, insomnia, paresthesia, headache, depression with or without development of suicidal tendencies, dementia, pathological gambling, increased libido including hypersexuality, impulse control symptoms. Convulsions also have occurred; however, a causal relationship with SINEMET has not been established.

Respiratory

Dyspnea, upper respiratory infection.

Skin

Rash, increased sweating, alopecia, dark sweat.

Urogenital

Urinary tract infection, urinary frequency, dark urine.

Laboratory Tests

Decreased hemoglobin and hematocrit; abnormalities in alkaline phosphatase, SGOT (AST), SGPT (ALT), LDH, bilirubin, BUN, Coombs test; elevated serum glucose; white blood cells, bacteria, and blood in the urine.

Other adverse reactions that have been reported with levodopa alone and with various carbidopa

levodopa formulations, and may occur with SINEMET are:

Body as a Whole

Abdominal pain and distress, fatigue.

Cardiovascular

Myocardial infarction.

Gastrointestinal

Gastrointestinal pain, dysphagia, sialorrhea, flatulence, bruxism, burning sensation of the tongue, heartburn, hiccups.

Metabolic

Edema, weight gain, weight loss.

Musculoskeletal

Leg pain.

Nervous System/Psychiatric

Ataxia, extrapyramidal disorder, falling, anxiety, gait abnormalities, nervousness, decreased mental acuity, memory impairment, disorientation, euphoria, blepharospasm (which may be taken as an early sign of excess dosage; consideration of dosage reduction may be made at this time), trismus, increased tremor, numbness, muscle twitching, activation of latent Horner's syndrome, peripheral neuropathy.

Respiratory

Pharyngeal pain, cough.

Skin

Malignant melanoma, flushing.

Special Senses

Oculogyric crises, diplopia, blurred vision, dilated pupils.

Urogenital

Urinary retention, urinary incontinence, priapism.

Miscellaneous

Bizarre breathing patterns, faintness, hoarseness, malaise, hot flashes, sense of stimulation.

Laboratory Tests

Decreased white blood cell count and serum potassium; increased serum creatinine and uric acid; protein and glucose in urine.

#### OVERDOSAGE

Management of acute overdosage with SINEMET is the same as management of acute overdosage with levodopa. Pyridoxine is not effective in reversing the actions of SINEMET.

General supportive measures should be employed, along with immediate gastric lavage. Intravenous fluids should be administered judiciously and an adequate airway maintained. Electrocardiographic monitoring should be instituted and the patient carefully observed for the development of arrhythmias; if required, appropriate antiarrhythmic therapy should be given. The possibility that the patient may have taken other drugs as well as SINEMET should be taken into consideration. To date, no experience has been reported with dialysis; hence, its value in overdosage is not known.

Based on studies in which high doses of levodopa and/or carbidopa were administered, a significant proportion of rats and mice given single oral doses of levodopa of approximately 1500-2000 mg/kg are expected to die. A significant proportion of infant rats of both sexes are expected to die at a dose of 800 mg/kg. A significant proportion of rats are expected to die after treatment with similar doses of carbidopa. The addition of carbidopa in a 1:10 ratio with levodopa increases the dose at which a significant proportion of mice are expected to die to 3360 mg/kg.

#### DOSAGE AND ADMINISTRATION

The optimum daily dosage of SINEMET must be determined by careful titration in each patient. SINEMET tablets are available in a 1:4 ratio of carbidopa to levodopa (SINEMET 25-100) as well as 1:10 ratio (SINEMET 25-250 and SINEMET 10-100). Tablets of the two ratios may be given separately or combined as needed to provide the optimum dosage.

Studies show that peripheral dopa decarboxylase is saturated by carbidopa at approximately 70 to 100 mg a day. Patients receiving less than this amount of carbidopa are more likely to experience nausea and vomiting.

# Usual Initial Dosage

Dosage is best initiated with one tablet of SINEMET 25-100 three times a day. This dosage schedule provides 75 mg of carbidopa per day. Dosage may be increased by one tablet every day or every other day, as necessary, until a dosage of eight tablets of SINEMET 25-100 a day is reached.

If SINEMET 10-100 is used, dosage may be initiated with one tablet three or four times a day. However, this will not provide an adequate amount of carbidopa for many patients. Dosage may be increased by one tablet every day or every other day until a total of eight tablets (2 tablets q.i.d.) is reached.

# How to Transfer Patients from Levodopa

**Levo dopa must be discontinued at least twelve hours before starting SINEMET.** A daily dosage of SINEMET should be chosen that will provide approximately 25% of the previous levodopa dosage. Patients who are taking less than 1500 mg of levodopa a day should be started on one tablet of SINEMET 25-100 three or four times a day. The suggested starting dosage for most patients taking more than 1500 mg of levodopa is one tablet of SINEMET 25-250 three or four times a day.

#### Maintenance

Therapy should be individualized and adjusted according to the desired therapeutic response. At least 70 to 100 mg of carbidopa per day should be provided. When a greater proportion of carbidopa is required, one tablet of SINEMET 25-100 may be substituted for each tablet of SINEMET 10-100. When more levodopa is required, SINEMET 25-250 should be substituted for SINEMET 25-100 or SINEMET 10-100. If necessary, the dosage of carbidopa levodopa 25-250 may be increased by one-half or one tablet every day or every other day to a maximum of eight tablets a day. Experience with total daily dosages of carbidopa greater than 200 mg is limited.

Because both therapeutic and adverse responses occur more rapidly with SINEMET than with levodopa alone, patients should be monitored closely during the dose adjustment period. Specifically, involuntary movements will occur more rapidly with SINEMET than with levodopa. The occurrence of involuntary movements may require dosage reduction. Blepharospasm may be a useful early sign of excess dosage in some patients.

# Addition of Other Antiparkinsonian Medications

Standard drugs for Parkinson's disease, other than levodopa without a decarboxylase inhibitor, may be used concomitantly while SINEMET is being administered, although dosage adjustments may be

required.

# Interruption of Therapy

Sporadic cases of hyperpyrexia and confusion have been associated with dose reductions and withdrawal of SINEMET. Patients should be observed carefully if abrupt reduction or discontinuation of SINEMET is required, especially if the patient is receiving neuroleptics. (See WARNINGS.)

If general anesthesia is required, SINEMET may be continued as long as the patient is permitted to take fluids and medication by mouth. If therapy is interrupted temporarily, the patient should be observed for symptoms resembling NMS, and the usual daily dosage may be administered as soon as the patient is able to take oral medication.

## HOW SUPPLIED

No. 3916A — SINEMET 25-100 Tablets are yellow, round, uncoated tablets, that are coded "650" on one side and plain on the other. They are supplied as follows:

NDC 0006-3916-68 bottles of 100.

No. 3915 — SINEMET 10-100 Tablets are light dapple-blue, round, uncoated tablets, that are coded "647" on one side and plain on the other. They are supplied as follows:

NDC 0006-3915-68 bottles of 100.

No. 3917 — SINEMET 25-250 Tablets are light dapple-blue, round, uncoated tablets, that are coded "654" on one side and plain on the other. They are supplied as follows:

NDC 0006-3917-68 bottles of 100.

# Storage and Handling

Store at 25°C (77°F), excursions permitted to 15-30°C (59-86°F) [see USP Controlled Room Temperature]. Store in a tightly closed container, protected from light and moisture.

Dispense in a tightly closed, light-resistant container.

Manufactured for: Merck Sharp & Dohme Corp., a subsidiary of **MERCK & CO., INC.,** Whitehouse Station, NJ 08889, USA

Manufactured by:

Mylan Pharmaceuticals, Inc. Morgantown, WV 26505, USA

For patent information: www.merck.com/product/patent/home.html

Copyright © 1996-2018 Merck Sharp & Dohme Corp., a subsidiary of Merck & Co., Inc. All rights reserved.

Revised: 04/2018

uspi-mk0295b-t-1804r004

Rx Only

# APPENDIX B. INSTRUCTIONS FOR DOSE CONVERSION TO IPX203

The goal of the dose conversion period is to establish a dosing regimen for IPX203 that minimizes "Off" time without causing troublesome dyskinesias.

The initial dose of IPX203 is based on the subject's most frequent IR CD-LD dose established during the 3-week IR CD-LD dose adjustment period.

Table B-1 Recommended Starting IPX203 LD Dosing Regimen Based on the Dosing Regimen of IR CD-LD at the End of the Dose Adjustment Period

| Most Frequent IR CD-LD Unit<br>Dose (mg) | Recommended Starting IPX203 Daily Dosing Regimen<br>CD-LD (mg) Every 8 Hours |
|---|---|
| 25-100 <sup>a</sup> | 70-280 mg (2 × 35-140 mg) |
| >25-100 – 37.5-150 | 105-420 mg (3 × 35-140 mg) |
| >37.5-150 – 50-200 | 140-560 mg (4 × 35-140 mg) |
| >50-200 | 175-700 mg (5 × 35-140 mg) |

Subjects who are on a total daily dose of less than 125-500 mg CD-LD from IR CD-LD should be advised to initially take IPX203 every 12 hours. The dosing interval may be reduced to approximately every 8 hours if the subject does not achieve an acceptable duration of effect.

# Conversion Instructions:

- Convert the subject's most frequent daily dose of IR CD-LD to the corresponding dose of IPX203 according to the above table. It is recommended that the subject takes IPX203 doses approximately every 8 hours apart (for example, a subject may take IPX203 at 6 AM, 2 PM, and 10 PM). Some subjects may benefit from a shorter or longer dosing interval. The dosing interval may vary but should not be more frequent than every 6 hours. The maximum recommended daily dose of IPX203 is 600-2400 mg CD-LD.
- Subjects who are on a total daily dose of less than 125-500 mg CD-LD from IR CD-LD should be advised to initially take IPX203 every 12 hours. The dosing interval may be reduced to approximately every 8 hours if the subject does not achieve an acceptable duration of effect.
- 3. The Investigator or their staff are advised to be in telephone contact with the subject, especially during the initial dose conversion to assess the need for dosage adjustment with the goal of minimizing "Off" time without causing troublesome dyskinesia or other dopaminergic side effects. Calls to the subject can be reduced appropriately when the subject reaches a stable dosing regimen.
- 4. If dose adjustment is necessary, consider the following options recognizing that the number of capsules at each dose may be varied to achieve an optimal response.

- a. If turning "On" is slow following the first morning dose, consider taking the morning IPX203 dose in the fasted state and/or increasing the dose by one capsule (35-140 mg IPX203 CD-LD).
- b. If turning "On" is slow later in the day or to reduce "end-of-dose" "Off" time, consider increasing the dose by one capsule (35-140 mg IPX203 CD-LD) before reducing the dosing interval.
- 5. In case of troublesome dyskinesias, use the following guidelines:
  - a. Consider reducing the dose by one capsule (35-140 mg IPX203 CD-LD).
  - b. Consider increasing the dosing interval.
- 6. The subject must be on a stable dosing regimen of IPX203 (no change in dose or in dosing frequency) for at least 5 days prior to Visit 4 (randomization).

# APPENDIX C. UNITED KINGDOM PARKINSON'S DISEASE SOCIETY BRAIN BANK DIAGNOSTIC CRITERIA FOR PARKINSON'S DISEASE

# Step 1: Diagnosis of Parkinsonism

Bradykinesia and at least one of the following:

- Muscular rigidity
- 4–6 Hz resting tremor
- postural instability not caused by primary visual, vestibular, cerebellar or Proprioceptive dysfunction

# Step 2: Features tending to exclude Parkinson's disease as the cause of Parkinsonism

- History of repeated strokes with stepwise progression of parkinsonian features
- History of repeated head injury
- History of definite encephalitis
- Neuroleptic treatment at onset of symptoms
- >1 affected relatives
- Sustained remission
- Strictly unilateral features after 3 years
- Supranuclear gaze palsy
- · Cerebellar signs
- Early severe autonomic involvement
- Early severe dementia with disturbances of memory, language and praxis
- Babinski's sign
- Presence of a cerebral tumour or communicating hydrocephalus on computed tomography scan
- Negative response to large doses of levodopa (if malabsorption excluded)
- MPTP exposure

# Step 3: Features that support a diagnosis of Parkinson's disease (three or more required for diagnosis of definite Parkinson's disease)

- Unilateral onset
- Rest tremor present
- Progressive disorder
- · Persistent asymmetry affecting the side of onset most
- Excellent (70–100%) response to levodopa
- Severe levodopa-induced chorea
- Levodopa response for ≥5 years
- Clinical course of ≥10 years

# APPENDIX D. MONTREAL COGNITIVE ASSESSMENT (MOCA)

# Montreal Cognitive Assessment (MoCA)

## Administration and Scoring Instructions

The Montreal Cognitive Assessment (MoCA) was designed as a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. Time to administer the MoCA is approximately 10 minutes. The total possible score is 30 points; a score of 26 or above is considered normal.

#### 1. Alternating Trail Making:

Administration: The examiner instructs the subject: "Please draw a line, going from a number to a letter in ascending order. Begin here [point to (1)] and draw a line from 1 then to A then to 2 and so on. End here [point to (E)]."

Scoring: Allocate one point if the subject successfully draws the following pattern: 1 -A- 2- B- 3- C- 4- D- 5- E, without drawing any lines that cross. Any error that is not immediately self-corrected earns a score of 0.

# 2. Visuoconstructional Skills (Cube):

Administration: The examiner gives the following instructions, pointing to the cube: "Copy this drawing as accurately as you can, in the space below".

Scoring: One point is allocated for a correctly executed drawing.

- · Drawing must be three-dimensional
- · All lines are drawn
- No line is added
- Lines are relatively parallel and their length is similar (rectangular prisms are accepted)

A point is not assigned if any of the above-criteria are not met.

## 3. Visuoconstructional Skills (Clock):

Administration: Indicate the right third of the space and give the following instructions: "Draw a clock. Put in all the numbers and set the time to 10 past 11".

Scoring: One point is allocated for each of the following three criteria:

- Contour (1 pt.): the clock face must be a circle with only minor distortion acceptable (e.g., slight imperfection on closing the circle);
- Numbers (1 pt.): all clock numbers must be present with no additional numbers; numbers must be in the correct order and placed in the approximate quadrants on the clock face; Roman numerals are acceptable; numbers can be placed outside the circle contour;
- Hands (1 pt.): there must be two hands jointly indicating the correct time; the hour hand must be clearly shorter than the minute hand; hands must be centred within the clock face with their junction close to the clock centre.

A point is not assigned for a given element if any of the above-criteria are not met.

MoCA Version August 18, 2010 © Z. Nasreddine MD

#### 4. Naming:

Administration: Beginning on the left, point to each figure and say: "Tell me the name of this animal".

Scoring: One point each is given for the following responses: (1) lion (2) rhinoceros or rhino (3) camel or dromedary.

# 5. Memory:

Administration: The examiner reads a list of 5 words at a rate of one per second, giving the following instructions: "This is a memory test. I am going to read a list of words that you will have to remember now and later on. Listen carefully. When I am through, tell me as many words as you can remember. It doesn't matter in what order you say them". Mark a check in the allocated space for each word the subject produces on this first trial. When the subject indicates that (s)he has finished (has recalled all words), or can recall no more words, read the list a second time with the following instructions: "I am going to read the same list for a second time. Try to remember and tell me as many words as you can, including words you said the first time." Put a check in the allocated space for each word the subject recalls after the second trial.

At the end of the second trial, inform the subject that (s)he will be asked to recall these words again by saying, "Lwill ask you to recall those words again at the end of the test."

Scoring: No points are given for Trials One and Two.

# 6. Attention:

Forward Digit Span: Administration: Give the following instruction: "I am going to say some numbers and when I am through, repeat them to me exactly as I said them". Read the five number sequence at a rate of one digit per second.

Backward Digit Span: Administration: Give the following instruction: "Now I am going to say some more numbers, but when I am through you must repeat them to me in the <u>backwards</u> order." Read the three number sequence at a rate of one digit per second.

<u>Scoring</u>: Allocate one point for each sequence correctly repeated, (N.B.: the correct response for the backwards trial is 2-4-7).

<u>Vigilance: Administration:</u> The examiner reads the list of letters at a rate of one per second, after giving the following instruction: "I am going to read a sequence of letters. Every time I say the letter A, tap your hand once. If I say a different letter, do not tap your hand".

Scoring: Give one point if there is zero to one errors (an error is a tap on a wrong letter or a failure to tap on letter A).

MoCA Version August 18, 2010 © Z. Nasreddine MD

<u>Serial 7s: Administration</u>: The examiner gives the following instruction: "Now, I will ask you to count by subtracting seven from 100, and then, keep subtracting seven from your answer until I tell you to stop." Give this instruction twice if necessary.

<u>Scoring</u>: This item is scored out of 3 points. Give no (0) points for no correct subtractions, 1 point for one correction subtraction, 2 points for two-to-three correct subtractions, and 3 points if the participant successfully makes four or five correct subtractions. Count each correct subtraction of 7 beginning at 100. Each subtraction is evaluated independently; that is, if the participant responds with an incorrect number but continues to correctly subtract 7 from it, give a point for each correct subtraction. For example, a participant may respond "92 - 85 - 78 - 71 - 64" where the "92" is incorrect, but all subsequent numbers are subtracted correctly. This is one error and the item would be given a score of 3.

# 7. Sentence repetition:

Administration: The examiner gives the following instructions: "I am going to read you a sentence. Repeat it after me, exactly as I say it [pause]: I only know that John is the one to help today." Following the response, say: "Now I am going to read you another sentence. Repeat it after me, exactly as I say it [pause]: The cat always hid under the couch when dogs were in the room."

Scoring: Allocate 1 point for each sentence correctly repeated. Repetition must be exact. Be alert for errors that are omissions (e.g., omitting "only", "always") and substitutions/additions (e.g., "John is the one who helped today;" substituting "hides" for "hid", altering plurals, etc.).

# 8. Verbal fluency:

Administration: The examiner gives the following instruction: "Tell me as many words as you can think of that begin with a certain letter of the alphabet that I will tell you in a moment. You can say any kind of word you want, except for proper nouns (like Bob or Boston), numbers, or words that begin with the same sound but have a different suffix, for example, love, lover, loving. I will tell you to stop after one minute. Are you ready? [Pause] Now, tell me as many words as you can think of that begin with the letter F. [time for 60 sec]. Stop."

Scoring: Allocate one point if the subject generates 11 words or more in 60 sec. Record the subject's response in the bottom or side margins.

# 9. Abstraction:

Administration: The examiner asks the subject to explain what each pair of words has in common, starting with the example: "Tell me how an orange and a banana are alike". If the subject answers in a concrete manner, then say only one additional time: "Tell me another way in which those items are alike". If the subject does not give the appropriate response (fruit), say, "Yes, and they are also both fruit." Do not give any additional instructions or clarification. After the practice trial, say: "Now, tell me how a train and a bicycle are alike". Following the response, administer the second trial, saying: "Now tell me how a ruler and a watch are alike". Do not give any additional instructions or prompts.

MoCA Version August 18, 2010 © Z. Nasreddine MD

Scoring: Only the last two item pairs are scored. Give 1 point to each item pair correctly answered. The following responses are acceptable:

Train-bicycle = means of transportation, means of travelling, you take trips in both;

Ruler-watch = measuring instruments, used to measure.

The following responses are not acceptable: Train-bicycle = they have wheels; Ruler-watch = they have numbers.

#### 10. Delayed recall:

Administration: The examiner gives the following instruction: "I read some words to you earlier, which I asked you to remember. Tell me as many of those words as you can remember." Make a check mark ( $\sqrt{\phantom{a}}$ ) for each of the words correctly recalled spontaneously without any cues, in the allocated space.

Scoring: Allocate 1 point for each word recalled freely without any cues.

#### Optional:

Following the delayed free recall trial, prompt the subject with the semantic category cue provided below for any word not recalled. Make a check mark ( $\sqrt{\phantom{0}}$ ) in the allocated space if the subject remembered the word with the help of a category or multiple-choice cue. Prompt all non-recalled words in this manner. If the subject does not recall the word after the category cue, give him/her a multiple choice trial, using the following example instruction, "Which of the following words do you think it was, NOSE, FACE, or HAND?"

Use the following category and/or multiple-choice cues for each word, when appropriate:

FACE: category cue: part of the body
VELVET: category cue: type of fabric
CHURCH: category cue: type of building
DAISY: category cue: type of flower
RED: category cue: a colour

multiple choice: nose, face, hand
multiple choice: denim, cotton, velvet
multiple choice: church, school, hospital
multiple choice: rose, daisy, tulip
multiple choice: red, blue, green

Scoring: No points are allocated for words recalled with a cue. A cue is used for clinical information purposes only and can give the test interpreter additional information about the type of memory disorder. For memory deficits due to retrieval failures, performance can be improved with a cue. For memory deficits due to encoding failures, performance does not improve with a cue.

# 11. Orientation:

Administration: The examiner gives the following instructions: "Tell me the date today". If the subject does not give a complete answer, then prompt accordingly by saying: "Tell me the [year, month, exact date, and day of the week]." Then say: "Now, tell me the name of this place, and which city it is in."

<u>Scoring</u>: Give one point for each item correctly answered. The subject must tell the exact date and the exact place (name of hospital, clinic, office). No points are allocated if subject makes an error of one day for the day and date.

**TOTAL SCORE:** Sum all subscores listed on the right-hand side. Add one point for an individual who has 12 years or fewer of formal education, for a possible maximum of 30 points. A final total score of 26 and above is considered normal.

MoCA Version August 18, 2010 © Z. Nasreddine MD



# APPENDIX E. MOVEMENT DISORDERS SOCIETY VERSION OF UNIFIED PARKINSON'S DISEASE RATING SCALE (MDS-UPDRS)

START TIME \_\_\_:\_\_ (hh:mm, 24-hr clock)

# **MDS-UPDRS**

Given formatting concerns, this MDS-UPDRS source document does not track the Patient ID on each page of the assessment. DO NOT remove the staple binding this MDS-UPDRS packet.

July 1,2008

Copyright © 2008 international Parkinson and Movement Disorder Society. All rights reserved
This scale may not be copied, distributed or otherwise used in whole or in part without prior written consent of the international Parkinson and Movement
Disorder Society

# **MDS-UPDRS Permissions**

Permission is required to use the MDS-developed Rating Scales (with the exception of personal/individual use). Reproduction, translation, modification, sale, or distribution of any portion of the MDS Rating Scales is strictly prohibited. MDS Rating Scales may not be incorporated into clinical trials, training or certification programs or materials, software programs, or otherwise except through use of the <a href="Permissions Request Form">Permissions Request Form</a> and payment of applicable fees.

Continue to p. 3 to view the MDS-UPDRS

# MDS-UPDRS

The Movement Disorder Society (MDS)-sponsored new version of the UPDRS is founded on the critique that was formulated by the Task Force for Rating Scales in Parkinson's disease (Mov Disord 2003;18:738-750). Thereafter, the MDS recruited a Chairperson to organize a program to provide the Movement Disorder community with a new version of the UPDRS that would maintain the overall format of the original UPDRS, but address issues identified in the critique as weaknesses and ambiguities. The Chairperson identified subcommittees with chairs and members. Each part was written by the appropriate subcommittee members and then reviewed and ratified by the entire group. These members are listed below.

The MDS-UPDRS has four parts: Part I (non-motor experiences of daily living), Part II (motor experiences of daily living), Part III (motor examination) and Part IV (motor complications). Part I has two components: IA concerns a number of behaviors that are assessed by the investigator with all pertinent information from patients and caregivers, and IB is completed by the patient with or without the aid of the caregiver, but independently of the investigator. These sections can, however, be reviewed by the rater to ensure that all questions are answered clearly and the rater can help explain any perceived ambiguities. Part II is designed to be a self-administered questionnaire like Part IB, but can be reviewed by the investigator to ensure completeness and clarity. Of note, the official versions of Part IA, Part IB and Part II of the MDS-UPDRS do not have separate on or off ratings. However, for individual programs or protocols the same questions can be used separately for on and off. Part III has instructions for the rater to give or demonstrate to the patient; it is completed by the rater. Part IV has instructions for the rater and also instructions to be read to the patient. This part integrates patient-derived information with the rater's clinical observations and judgments and is completed by the rater.

The authors of this new version are:

Chairperson: Christopher G. Goetz

Part I: Werner Poewe (chair), Bruno Dubois, Anette Schrag Part II: Matthew B. Stern (chair), Anthony E. Lang, Peter A. LeWitt Part III: Stanley Fahn (chair), Joseph Jankovic, C. Warren Olanow

Part IV: Pablo Martinez-Martin (chair), Andrew Lees, Olivier Rascol, Bob van Hilten Development Standards: Glenn T. Stebbins (chair), Robert Holloway, David Nyenhuis

Appendices: Cristina Sampaio (chair), Richard Dodel, Jaime Kulisevsky Statistical Testing: Barbara Tilley (chair), Sue Leurgans, Jean Teresi,

Consultant: Stephanie Shaftman, Nancy LaPelle

Contact person: Christopher G. Goetz, MD Rush University Medical Center 1725 W. Harrison Street, Suite 755

Chicago, IL USA 60612

Telephone 312-942-8016 Email: cgoetz@rush.edu

July 1, 2008

# Part I: Non-Motor Aspects of Experiences of Daily Living (nM-EDL)

Overview: This portion of the scale assesses the non-motor impact of Parkinson's disease (PD) on patients' experiences of daily living. There are 13 questions. Part 1A is administered by the rater (six questions) and focuses on complex behaviors. Part 1B is a component of the self-administered Patient Questionnaire that covers seven questions on non-motor experiences of daily living.

#### Part 1A:

In administering Part IA, the examiner should use the following guidelines:

- Mark at the top of the form the primary data source as patient, caregiver, or patient and caregiver in equal proportion.
- The response to each item should refer to a period encompassing the prior week including the day on which the information is collected.
- 3. All items must have an integer rating (no half points, no missing scores). In the event that an item does not apply or cannot be rated (e.g., amputee who cannot walk), the item is marked UR for Unable to Rate.
- The answers should reflect the usual level of function and words such as "usually", "generally", "most of the time" can be used with patients.
- 5. Each question has a text for you to read (Instructions to patients/caregiver). After that statement, you can elaborate and probe based on the target symptoms outlined in the Instructions to examiner. You should NOT READ the RATING OPTIONS to the patient/caregiver, because these are written in medical terminology. From the interview and probing, you will use your medical judgment to arrive at the best response.
- Patients may have co-morbidities and other medical conditions that can affect their function. You and the patient must rate the problem as it exists and do not attempt to separate elements due to Parkinson's disease from other conditions.

#### **EXAMPLE OF NAVIGATING THROUGH THE RESPONSE OPTIONS FOR PART 1A**

Suggested strategies for obtaining the most accurate answer:

After reading the instructions to the patient, you will need to probe the entire domain under discussion to determine Normal vs. problematic: If your questions do not identify any problem in this domain, record 0 and move on to the next question.

If your questions identify a problem in this domain, you should work next with a reference anchor at the mid-range (option 2 or Mild) to find out if the patient functions at this level, better or worse. You will not be reading the choices of responses to the patient as the responses use clinical terminology. You will be asking enough probing questions to determine the response that should be coded.

Work up and down the options with the patient to identify the most accurate response, giving a final check by excluding the options above and below the selected response.



July 1, 2008 Copyright © 2008 International Parkinson and Movement Disorder Society. All rights reserved Page 3
This scale may not be copied, distributed or otherwise used in whole or in part without prior written consent of the International Parkinson and Movement Disorder Society

| MDS UPDRS Part I: Non-Motor Aspects of Experiences of Daily Living (nM-EDL) | | | |
|---|---|---|---|
| Part 1A: Complex | behaviors: [completed | by rater] | |
| Primary source of in | nformation: | | |
| ☐ Patient | ☐ Caregiver | ☐ Patient and Caregiver in Equal Proportion | |
| Some questions cor<br>areas, please choos<br>WEEK. If you are no | ncern common problems<br>se the best response tha | you six questions about behaviors that you may or may not exis and some concern uncommon ones. If you have a problem in t describes how you have felt MOST OF THE TIME during the n, you can simply respond NO. I am trying to be thorough, so I | n one of the<br>PAST |
| slowing, impaired re | niner: Consider all types | of altered level of cognitive function including cognitive deficits in attention and orientation. Rate their impact on batient and/or caregiver. | SCORE |
| following conversati | ions, paying attention, th | r the past week have you had problems remembering things,<br>inking clearly, or finding your way around the house or in<br>giver to elaborate and probes for information.] | |
| 0: Normal: | No cognitive impairme | nt. | |
| 1: Slight: | | d by patient or caregiver with no concrete interference with<br>carry out normal activities and social interactions. | |
| 2: Mild: | | itive dysfunction, but only minimal interference with<br>carry out normal activities and social interactions. | |
| 3; Moderate; | Cognitive deficits interiout normal activities ar | fere with but do not preclude the patient's ability to carry and social interactions. | |
| 4: Severe: | Cognitive dysfunction social interactions. | precludes the patient's ability to carry out normal activities and | |

July 1, 2008 Copyright © 2008 International Parkinson and Movement Disorder Society. All rights reserved. Page 4
This scale may not be copied, distributed or otherwise used in whole or in part without prior written consent of the International Parkinson and Movement Disorder Focusty

| 1.2 HALLUCINATI | ONS AND PSYCHOSIS | SCORE |
|---|---|---|
| (spontaneous false<br>and gustatory). Dete<br>impressions) as wel | niner: Consider both illusions (misinterpretations of real stimuli) and hallucinations sensations). Consider all major sensory domains (visual, auditory, tactile, olfactory ermine presence of unformed (for example sense of presence or fleeting false il as formed (fully developed and detailed) sensations. Rate the patient's insight into dentify delusions and psychotic thinking. | |
| | nts jand caregiver]: Over the past week have you seen, heard, smelled or felt things there? [If yes, examiner asks patient or caregiver to elaborate and probes for | |
| 0: Normal: | No hallucinations or psychotic behavior. | |
| 1: Slight: | Illusions or non-formed hallucinations, but patient recognizes them without loss of insight. | |
| 2: <b>M</b> il <b>d</b> : | Formed hallucinations independent of environmental stimuli. No loss of insight. | |
| 3: Moderate: | Formed hallucinations with loss of insight. | |
| 4: Severe: | Patient has delusions or paranoia. | |
| enjoyment. Determi | niner: Consider low mood, sadness, hopelessness, feelings of emptiness or loss of the inequality in the control of the control | |
| Instruction to the pa<br>to enjoy things? If y | to carry out daily routines and engage in social interactions. Internet (and caregiver): Over the past week have you felt low, sad, hopeless or unable es, was this feeling for longer than one day at a time? Did it make it difficult for you lactivities or to be with people? [If yes, examiner asks patient or caregiver to es for information.] | |
| 0: Normal: | No depressed mood. | |
| 1: Slight: | Episodes of depressed mood that are not sustained for more than one day at a time. No interference with patient's ability to carry out normal activities and social interactions. | |
| 2: Mild: | Depressed mood that is sustained over days, but without interference with normal activities and social interactions. | |
| 3: Moderate: | Depressed mood that interferes with, but does not preclude, the patient's ability to carry out normal activities and social interactions. | |
| | • | |
| 4: Severe; | Depressed mood precludes patient's ability to carry out normal activities and social interactions. | |

July 1, 2008 Copyright © 2008 International Parkinson and Movement Disorder Society. All rights reserved Page 5
This scale may not be copied, distributed or otherwise used in whole or in part without prior written consent of the International Parkinson and Movement Disorder Novety

| 1.4 ANX | (IOUS MO | ор | SCORE |
|---|---|---|---|
| over the | past week | niner: Determine nervous, tense, worried or anxious feelings (including panic attacks) and rate their duration and interference with the patient's ability to carry out daily e in social interactions. | |
| yes, was | this feeling<br>or to be w | ents <u>[and caregiver]</u> : Over the past week have you felt nervous, worried or tense? If<br>g for longer than one day at a time? Did it make it difficult for you to follow your usual<br>ith other people? [If yes, examiner asks patient or caregiver to elaborate and probes | |
| 0: 1 | Normal: | No anxious feelings. | |
| 1: 5 | | Anxious feelings present but not sustained for more than one day at a time. No interference with patient's ability to carry out normal activities and social interactions. | |
| 2: N | | Anxious feelings are sustained over more than one day at a time, but without interference with patient's ability to carry out normal activities and social interactions. | |
| 3: N | | Anxious feelings interfere with, but do not preclude, the patient's ability to carry out normal activities and social interactions. | |
| 4: 5 | | Anxious feelings preclude patient's ability to carry out normal activities and social interactions. | |
| 1.5 APA | THY | | |
| and rate t | the impact<br>r should att | <u>niner</u> : Consider level of spontaneous activity, assertiveness, motivation and initiative of reduced levels on performance of daily routines and social interactions. Here the tempt to distinguish between apathy and similar symptoms that are best explained by | |
| | | ents (and caregiver). Over the past week, have you felt indifferent to doing activities e? [If yes, examiner asks patient or caregiver to elaborate and probes for information.] | |
| 0: 1 | Normal: | No apathy. | |
| 1: 9 | Slight: | Apathy appreciated by patient and/or caregiver, but no interference with daily activities and social interactions. | |
| 2: N | Mild: | Apathy interferes with isolated activities and social interactions. | |
| 3: N | Moderate: | Apathy interferes with most activities and social interactions. | |
| 4: 5 | Severe: | Passive and withdrawn, complete loss of initiative. | |

July 1, 2008 Copyright © 2008 International Parkinson and Movement Disorder Society. All rights reserved Page 6
This scale may not be copied, distributed or otherwise used in whole or in part without prior written consent of the International Parkinson and Movement Disorder Novely

| Instructions to examiner: Co excessive gambling (e.g. ca interests (e.g., unusual inter other repetitive activities (e.g. extra non-prescribed medica impact of such abnormal act social relations (including nacredit cards, major family co activity). Instructions to patients fand urges that are hard to controhard to stop? [Give patient.] | onsider involvement in a variety of activities including atypical or sinos or lottery tickets), atypical or excessive sexual drive or rest in pornography, masturbation, sexual demands on partner), g. hobbies, dismantling objects, sorting or organizing), or taking ation for non-physical reasons (i.e., addictive behavior). Rate the tivities/behaviors on the patient's personal life and on his family and edd to borrow money or other financial difficulties like withdrawal of onflicts, lost time from work, or missed meals or sleep because of the licaregiver! Over the past week, have you had unusually strong of? Do you feel driven to do or think about something and find it examples such as gambling, cleaning, using the computer, taking about food or sex, all depending on the patients.] | SCORE |
|---|---|---|
| 1: Slight: Proble family/ 2: Mild: Proble and fai 3: Moderate: Proble and fai 4: Severe: Proble | blems present. In a are present but usually do not cause any difficulties for the patient or caregiver. In a are present and usually cause a few difficulties in the patient's personal mily life. In a are present and usually cause a lot of difficulties in the patient's personal mily life. In a are present and preclude the patient's ability to carry out normal es or social interactions or to maintain previous standards in personal and life. | |
| Other Sensation, Urinary | in Part I (Non-motor Experiences of Daily Living) [Sleep, Daytime Sleepiness,<br>Problems, Constipation Problems, Lightheadedness on Standing, and Fatigue<br>ionnaire along with all questions in Part II [Motor Experiences of Daily Living]. | |

July 1, 2008 Copyright © 2008 International Parkinson and Movement Disorder Society. All rights reserved Page 7
This scale may not be copied, distributed or otherwise used in whole or in part without prior written consent of the International Parkinson and Movement Disorder Novacy

| Patient Questionnaire: | | |
|---|---|---|
| Instructions: | | |
| This questionna | ire will ask you abou | t your experiences of daily living. |
| | | ng to be thorough, and some of these questions may<br>er. If you do not have the problem, simply mark 0 for NO. |
| Please read ead applies to you. | ch one carefully and i | read all answers before selecting the one that best |
| patients can do | things better at one tach question, so plea | r usual function over the past week including today. Some time of the day than at others. However, only one answer se mark the answer that best describes what you can |
| | | ons besides Parkinson's disease. Do not worry about nother conditions. Just answer the question with your |
| Use only 0, 1, 2 | 2, 3, 4 for answers, no | othing else. Do not leave any blanks. |
| | nurse can review the<br>her alone or with thei | questions with you, but this questionnaire is for patients r caregivers. |
| Who is filling ou | it this questionnaire ( | check the best answer): |
| ☐ Patient | ☐ Caregiver | ☐ Patient and Caregiver in Equal Proportion |

July 1, 2008 Copyright © 2008 International Parkinson and Movement Disorder Society. All rights reserved Page 8
This scale may not be copied, distributed or otherwise used in whole or in part without prior written consent of the International Parkinson and Movement Disorder Novelle

| .7 SI | LEEP PROB | BLEMS | SCOR |
|---|---|---|---|
| | | k, have you had trouble going to sleep at night or staying asleep<br>Consider how rested you felt after waking up in the morning. | |
| 0: | Normal: | No problems. | |
| 1: | Slight: | Sleep problems are present but usually do not cause trouble getting a full night of sleep. | |
| 2: | Mild: | Sleep problems usually cause some difficulties getting a full night of sleep. | |
| 3: | Moderate: | Sleep problems cause a lot of difficulties getting a full night of sleep, but I still usually sleep for more than half the night. | |
| 4: | Severe: | I usually do not sleep for most of the night. | |
| | AYTIME SLI | | |
| ver t | | EEPINESS k, have you had trouble staying awake during the daytime? No daytime sleepiness. | |
| over t | he past weel | k, have you had trouble staying awake during the daytime? | |
| 0:<br>0:<br>1: | he past weel | k, have you had trouble staying awake during the daytime? No daytime sleepiness. | |
| 0:<br>1:<br>2: | he past weel<br>Normal:<br>Slight: | k, have you had trouble staying awake during the daytime? No daytime sleepiness. Daytime sleepiness occurs but I can resist and I stay awake. Sometimes I fall asleep when alone and relaxing. For example, | |
| 0:<br>1:<br>2:<br>3: | he past weel<br>Normal:<br>Slight:<br>Mild: | k, have you had trouble staying awake during the daytime? No daytime sleepiness. Daytime sleepiness occurs but I can resist and I stay awake. Sometimes I fall asleep when alone and relaxing. For example, while reading or watching TV. I sometimes fall asleep when I should not. For example, while | |

July 1, 2008 Copyright © 2008 International Parkinson and Movement Disorder Society. All rights reserved Page S
This scale may not be copied, distributed or otherwise used in whole or in part without prior written consent of the International Parkinson and Movement Disorder Novacy

| PAIN AND O | THER SENSATIONS | SCORE |
|---|---|---|
| er the past wee<br>gling or cramps | k, have you had uncomfortable feelings in your body like pain, aches? | |
| 0: Normal: | No uncomfortable feelings. | |
| 1: Slight: | I have these feelings. However, I can do things and be with other people without difficulty. | |
| 2: Mild: | These feelings cause some problems when I do things or am with other people. | |
| 3: Moderate: | These feelings cause a lot of problems, but they do not stop me from doing things or being with other people. | |
| 4: Severe: | These feelings stop me from doing things or being with other people. | |
| 0 URINARY P | ROBLEMS | |
| er the past wee | ROBLEMS k, have you had trouble with urine control? For example, an urgent need to urinate too often, or urine accidents? | |
| er the past wee | k, have you had trouble with urine control? For example, an urgent | |
| er the past wee<br>ed to urinate, a | k, have you had trouble with urine control? For example, an urgent need to urinate too often, or urine accidents? | |
| er the past wee<br>ed to urinate, a<br>0: Normal: | k, have you had trouble with urine control? For example, an urgent need to urinate too often, or urine accidents? No urine control problems. I need to urinate often or urgently. However, these problems do | |
| er the past wee<br>ed to urinate, a<br>0: Normal:<br>1: Slight: | k, have you had trouble with urine control? For example, an urgent need to urinate too often, or urine accidents? No urine control problems. I need to urinate often or urgently. However, these problems do not cause difficulties with my daily activities. Urine problems cause some difficulties with my daily activities. | |
| er the past wee<br>ed to urinate, a<br>0: Normal:<br>1: Slight:<br>2: Mild: | k, have you had trouble with urine control? For example, an urgent need to urinate too often, or urine accidents? No urine control problems. I need to urinate often or urgently. However, these problems do not cause difficulties with my daily activities. Urine problems cause some difficulties with my daily activities. However, I do not have urine accidents. Urine problems cause a lot of difficulties with my daily activities, | |
| er the past wee ed to urinate, a 0: Normal: 1: Slight: 2: Mild: 3: Moderate: | k, have you had trouble with urine control? For example, an urgent need to urinate too often, or urine accidents? No urine control problems. I need to urinate often or urgently. However, these problems do not cause difficulties with my daily activities. Urine problems cause some difficulties with my daily activities. However, I do not have urine accidents. Urine problems cause a lot of difficulties with my daily activities, including urine accidents. I cannot control my urine and use a protective garment or have a | |
| er the past wee ed to urinate, a 0: Normal: 1: Slight: 2: Mild: 3: Moderate: | k, have you had trouble with urine control? For example, an urgent need to urinate too often, or urine accidents? No urine control problems. I need to urinate often or urgently. However, these problems do not cause difficulties with my daily activities. Urine problems cause some difficulties with my daily activities. However, I do not have urine accidents. Urine problems cause a lot of difficulties with my daily activities, including urine accidents. I cannot control my urine and use a protective garment or have a | |

July 1, 2009 Copyright © 2008 International Parkinson and Movement Disorder Society. All rights reserved: Page 10
This scale may not be copied, distributed or otherwise used in whole or in part without prior written consent of the International Parkinson and Movement Disorder Society.

| 1.11 CONSTIPATI | ON PROBLEMS | SCORE |
|---|---|---|
| Over the past week moving your bowels | have you had constipation troubles that cause you difficulty s? | |
| 0: Normal: | No constipation. | |
| 1: Slight: | I have been constipated. I use extra effort to move my bowels.<br>However, this problem does not disturb my activities or my being comfortable. | |
| 2: Mild: | Constipation causes me to have some troubles doing things or being comfortable. | |
| 3: Moderate: | Constipation causes me to have a lot of trouble doing things or being comfortable. However, it does not stop me from doing anything. | |
| 4: Severe: | I usually need physical help from someone else to empty my bowels. | |
| 1.12 LIGHT HEAD | EDNESS ON STANDING | |
| Over the past week or lying down? | , have you felt faint, dizzy or foggy when you stand up after sitting | |
| 0: Normal: | No dizzy or foggy feelings. | |
| 1: Slight: | Dizzy or foggy feelings occur. However, they do not cause me troubles doing things. | |
| 2: Mild: | Dizzy or foggy feelings cause me to hold on to something, but I do not need to sit or lie back down. | |
| 3: Moderate: | Dizzy or foggy feelings cause me to sit or lie down to avoid fainting or falling. | |
| 4: Severe: | Dizzy or foggy feelings cause me to fall or faint. | |

July 1. 2008 Copyright © 2008 International Parkinson and Movement Disorder Society. All rights reserved Page 1
This scale may not be copied, distributed or otherwise used in whole or in part without prior written consent of the International Parkinson and Movement Disorder Novacy

| 1.13 FATIGUE | | SCORE |
|---|---|---|
| Over the past week, his sleepy or sad. | nave you usually felt fatigued? This feeling is not part of being | |
| 0: Normal: No | lo fatigue. | |
| | atigue occurs. However it does not cause me troubles doing nings or being with people. | |
| | atigue causes me some troubles doing things or being with eople. | |
| | atigue causes me a lot of troubles doing things or being with eople. However, it does not stop me from doing anything. | |
| 4: Severe: Fa | atigue stops me from doing things or being with people. | |
| Part II: Mo | otor Aspects of Experiences of Daily Living (M-EDL) | |
| 2.1 SPEECH | | |
| Over the past week, h | nave you had problems with your speech? | |
| 0: Normal: No | lot at all (no problems). | |
| | My speech is soft, slurred or uneven, but it does not cause others ask me to repeat myself. | |
| | ly speech causes people to ask me to occasionally repeat myself, but not everyday. | |
| 1 | ly speech is unclear enough that others ask me to repeat myself very day even though most of my speech is understood. | |
| 4: Severe: M | lost or all of my speech cannot be understood. | |

July 1, 2008 Copyright © 2008 International Parkinson and Movement Disorder Society. All rights reserved. Page 12
This scale may not be copied, distributed or otherwise used in whole or in part without prior written consent of the International Parkinson and Movement Disorder Society.

| 2.2 SALIVA AND DROOLING | | SCORE |
|---|---|---|
| Over the past week, have you usua awake or when you sleep? | ally had too much saliva during when you are | |
| 0: Normal: Not at all (no p | roblems). | |
| 1: Slight: I have too mud | ch saliva, but do not drool. | |
| 2: Mild: I have some d | rooling during sleep, but none when I am awake. | _ |
| 3: Moderate: I have some ditissues or a ha | rooling when I am awake, but I usually do not need indkerchief. | |
| | n drooling that I regularly need to use tissues or a o protect my clothes. | |
| 2.3 CHEWING AND SWALLOWII | NG | |
| | ally had problems swallowing pills or eating meals?<br>ed or your meals to be made soft, chopped or | |
| 0: Normal: No problems. | | |
| | slowness in my chewing or increased effort at it I do not choke or need to have my food specially | |
| | my pills cut or my food specially prepared because swallowing problems, but I have not choked over | |
| 3: Moderate. I choked at lea | st once in the past week. | |
| 4: Severe: Because of ch tube. | ewing and swallowing problems, I need a feeding | |

July 1, 2009 Copyright © 2008 International Parkinson and Movement Disorder Society. All rights reserved: Page 13
This scale may not be copied, distributed or otherwise used in whole or in part without prior written consent of the International Parkinson and Movement Disorder Society.

| 2.4 EATING TASK | KS . | SCORE |
|---|---|---|
| | k, have you usually had troubles handling your food and using or example, do you have trouble handling finger foods or using his, chopsticks? | |
| 0: Normal: | Not at all (no problems). | |
| 1: Slight: | I am slow, but I do not need any help handling my food and have not had food spills while eating. | |
| 2: Mild: | I am slow with my eating and have occasional food spills. I may need help with a few tasks such as cutting meat. | |
| 3: Moderate: | I need help with many eating tasks but can manage some alone. | |
| 4: Severe: | I need help for most or all eating tasks. | |
| 2.5 DRESSING | | |
| | k, have you usually had problems dressing? For example, are you dhelp with buttoning, using zippers, putting on or taking off your | |
| 0: Normal: | Not at all (no problems). | |
| 1: Slight: | am slow but I do not need help. | |
| 2: Mild: | am slow and need help for a few dressing tasks (buttons, bracelets). | |
| 3: Moderate: | I need help for many dressing tasks. | |
| 4: Severe: | I need help for most or all dressing tasks. | |

July 1, 2008 Copyright © 2008 International Parkinson and Movement Disorder Society. All rights reserved: Page 1
This scale may not be copied, distributed or otherwise used in whole or in part without prior written consent of the International Parkinson and Novement Disorder Novety.

| 2.6 HYGIENE | SCORE | E |
|---|---|---|
| Over the past week, have you usually been slow or do you need help with washing, bathing, shaving, brushing teeth, combing your hair or with other personal hygiene? | | |
| 0: Normal: Not at all (no | problems). | |
| 1: Slight: am slow but | t I do not need any help. | ] |
| 2: Mild: I need somed | one else to help me with some hygiene tasks. | J |
| 3: Moderate: I need help for | or many hygiene tasks. | |
| 4: Severe: I need help fo | or most or all of my hygiene tasks. | |
| 2.7 HANDWRITING | | |
| Over the past week, have people usually had trouble reading your handwriting? | | |
| 0: Normal: Not at all (no | problems). | |
| 1: Slight: My writing is: | slow, clumsy or uneven, but all words are clear. | 1 |
| 2: Mild: Some words | are unclear and difficult to read. | |
| 3: Moderate: Many words | are unclear and difficult to read. | |
| 4: Severe: Most or all wo | ords cannot be read. | |
| 2.8 DOING HOBBIES AND OTHER ACTIVITIES | | |
| Over the past week, have you usually had trouble doing your hobbies or other things that you like to do? | | |
| 0: Normal: Not at all (no | problems). | |
| 1: Slight: am a bit slo | w but do these activities easily. | 1 |
| 2: Mild: I have some | difficulty doing these activities. | ] |
| 3: Moderate: I have major | problems doing these activities, but still do most. | |
| 4: Severe: am unable t | o do most or all of these activities. | |

July 1. 2008 Copyright © 2008 International Parkinson and Movement Disorder Society. All rights reserved Page 1
This scale may not be copied, distributed or otherwise used in whole or in part without prior written consent of the International Parkinson and Movement Disorder Novacy

| 2.9 | Τl | JRNING IN E | BED | SCORE |
|---|---|---|---|---|
| Over the past week, do you usually have trouble turning over in bed? | | | | |
| | <ul><li>0: Normal: Not at all (no problems).</li><li>1: Slight: have a bit of trouble turning, but do not need any help.</li></ul> | | | |
| | 2: Mild I have a lot of trouble turning and need occasional help from someone else. | | | |
| | 3: | Moderate: | To turn over I often need help from someone else. | |
| | 4: | Severe: | am unable to turn over without help from someone else. | |
| 2.10 TREMOR | | | | |
| Over the past week, have you usually had shaking or tremor? | | | | |
| | 0: | Normal: | Not at all. I have no shaking or tremor. | |
| | 1: | Slight: | Shaking or tremor occurs but does not cause problems with any activities. | |
| | 2: | Mild: | Shaking or tremor causes problems with only a few activities. | |
| | 3: | Moderate: | Shaking or tremor causes problems with many of my daily activities. | |
| | 4: | Severe: | Shaking or tremor causes problems with most or all activities. | |
| 2.11 GETTING OUT OF BED, A CAR, OR A DEEP CHAIR | | | | |
| Over the past week, have you usually had trouble getting out of bed, a car seat, or a deep chair? | | | | |
| | 0: | Normal: | Not at all (no problems). | |
| | 1: | Slight: | am slow or awkward, but I usually can do it on my first try. | |
| | 2: | Mild: | need more than one try to get up or need occasional help. | |
| | 3: | Moderate: | I sometimes need help to get up, but most times I can still do it on my own. | |
| | 4: | Severe: | need help most or all of the time. | |

July 1. 2008 Copyright © 2008 International Parkinson and Movement Disorder Society. All rights reserved Page 16
This scale may not be copied, distributed or otherwise used in whole or in part without prior written consent of the International Parkinson and Movement Disorder Society.
| 2.12 WALKING AND | BALANCE | SCORE |
|---|---|---|
| Over the past week, h | nave you usually had problems with balance and walking? | |
| 0: Normal: N | lot at all (no problems). | |
| 1: Slight: | am slightly slow or may drag a leg. I never use a walking aid. | |
| | occasionally use a walking aid, but I do not need any help from nother person. | |
| fa | usually use a walking aid (cane, walker) to walk safely without alling. However, I do not usually need the support of another person. | |
| | usually use the support of another person to walk safely without alling. | |
| 2.13 FREEZING | | |
| as if your feet are stud | on your usual day when walking, do you suddenly stop or freeze ck to the floor. | |
| 0: Normal: N | lot at all (no problems). | |
| h | briefly freeze but I can easily start walking again. I do not need telp from someone else or a walking aid (cane or walker) because if freezing. | |
| s | freeze and have trouble starting to walk again, but I do not need comeone's help or a walking aid (cane or walker) because of reezing. | |
| b | When I freeze I have a lot of trouble starting to walk again and, because of freezing, I sometimes need to use a walking aid or need someone else's help. | |
| | decause of freezing, most or all of the time, I need to use a walking aid or someone's help. | |
| This completes the questionnaire. We may have asked about problems you do not even have, and may have mentioned problems that you may never develop at all. Not all patients develop all these problems, but because they can occur, it is important to ask all the questions to every patient. Thank you for your time and attention in completing this questionnaire. | | |

July 1, 2008 Copyright © 2008 International Parkinson and Movement Disorder Society. All rights reserved Page 17.
This scale may not be copied, distributed or otherwise used in whole or in part without prior written consent of the International Parkinson and Movement Disorder Society.

| Part III: Motor Examination |
|---|
| Overview: This portion of the scale assesses the motor signs of PD. In administering Part III of the MDS-UPDRS the examiner should comply with the following guidelines: |
| At the top of the form, mark whether the patient is on medication for treating the symptoms of Parkinson's disease and, if on levodopa, the time since the last dose. |
| Also, if the patient is receiving medication for treating the symptoms of Parkinson's Disease, mark the patient's clinical state using the following definitions: ON is the typical functional state when patients are receiving medication and have a good response. OFF is the typical functional state when patients have a poor response in spite of taking medications. |
| The investigator should "rate what you see". Admittedly, concurrent medical problems such as stroke, paralysis, arthritis, contracture, and orthopedic problems such as hip or knee replacement and scoliosis may interfere with individual items in the motor examination. In situations where it is absolutely impossible to test (e.g., amputations, plegia, limb in a cast), use the notation " <b>UR</b> " for Unable to Rate. Otherwise, rate the performance of each task as the partient performs in the context of co-morbidities. |
| All items must have an integer rating (no half points, no missing ratings). |
| Specific instructions are provided for the testing of each item. These should be followed in all instances. The investigator demonstrates while describing tasks the patient is to perform and rates function immediately thereafter. For Global Spontaneous Movement and Rest Tremor items (3.14 and 3.17), these items have been placed purposefully at the end of the scale because clinical information pertinent to the score will be obtained throughout the entire examination. |
| At the end of the rating, indicate if dyskinesia (chorea or dystonia) was present at the time of the examination, and if so, whether these movements interfered with the motor examination. |
| 3a Is the patient on medication for treating the symptoms of Parkinson's Disease? $\square$ No $\square$ Yes |
| 3b If the patient is receiving medication for treating the symptoms of Parkinson's Disease,<br>mark the patient's clinical state using the following definitions; |
| ON: On is the typical functional state when patients are receiving medication and have a good response. |
| ☐ OFF: Off is the typical functional state when patients have a poor response in spite of taking medications. |
| 3c Is the patient on Levodopa? |

July 1, 2008 Copyright © 2008 International Parkinson and Movement Disorder Society. All rights reserved Page 1. This scale may not be copied, distributed or otherwise used in whole or in part without prior written consent of the International Parkinson and Movement Disorder Society.

| SPEECH | | SCO |
|---|---|---|
| essary. Sugges<br>tor's office. Eva | miner: Listen to the patient's free-flowing speech and engage in conversation if sted topics: ask about the patient's work, hobbies, exercise, or how he got to the fluate volume, modulation (prosody) and clarity, including slurring, palilalia (repetition chyphemia (rapid speech, running syllables together). | |
| 0: Normal: | No speech problems. | |
| 1: Slight: | Loss of modulation, diction or volume, but still all words easy to understand. | |
| 2: Mild: | Loss of modulation, diction, or volume, with a few words unclear, but the overall sentences easy to follow. | |
| 3: Moderate: | Speech is difficult to understand to the point that some, but not most, sentences are poorly understood. | |
| 4: Severe: | Most speech is difficult to understand or unintelligible. | |
| FACIAL EXPE | RESSION | |
| | miner: Observe the patient sitting at rest for 10 seconds, without talking and also | |
| | erve eye-blink frequency, masked facies or loss of facial expression, spontaneous of lips. | |
| 0: Normal: | | |
| 0: Normal:<br>1: Slight: | of lips. | |
| | of lips. Normal facial expression. | |
| 1: Slight:<br>2: Mild: | of lips. Normal facial expression. Minimal masked facies manifested only by decreased frequency of blinking. In addition to decreased eye-blink frequency, Masked facies present in the lower face as well, namely fewer movements around the mouth, such as less | |
| 1: Slight:<br>2: Mild: | of lips. Normal facial expression. Minimal masked facies manifested only by decreased frequency of blinking. In addition to decreased eye-blink frequency, Masked facies present in the lower face as well, namely fewer movements around the mouth, such as less spontaneous smiling, but lips not parted. | |
| <ol> <li>Slight:</li> <li>Mild:</li> <li>Moderate:</li> </ol> | of lips. Normal facial expression. Minimal masked facies manifested only by decreased frequency of blinking. In addition to decreased eye-blink frequency, Masked facies present in the lower face as well, namely fewer movements around the mouth, such as less spontaneous smilling, but lips not parted. Masked facies with lips parted some of the time when the mouth is at rest. | |

July 1. 2008 Copyright © 2008 International Parkinson and Movement Disorder Society. All rights reserved Page 15
This scale may not be copied, distributed or otherwise used in whole or in part without prior written consent of the International Parkinson and Movement Disorder Novety

| 3.3 RIGIDITY | | SCORE |
|---|---|---|
| Instructions to examiner: Rigidity is judged on slow passive movement of major joints with the patient in a relaxed position and the examiner manipulating the limbs and neck. First, test without an activation maneuver. Test and rate neck and each limb separately. For arms, test the wrist and elbow joints simultaneously. For legs, test the hip and knee joints simultaneously. If no rigidity is detected, use an activation maneuver such as tapping fingers, fist opening/closing, or heel tapping in a limb not being tested. Explain to the patient to go as limp as possible as you test for rigidity. | | Neck |
| 0: Normal: | No rigidity. | |
| 1: Slight: | Rigidity only detected with activation maneuver. | |
| 2: <b>M</b> il <b>d</b> : | Rigidity detected without the activation maneuver, but full range of motion is easily achieved. | RUE |
| 3: Moderate: | Rigidity detected without the activation maneuver; full range of motion is achieved with effort. | |
| 4: Severe: | Rigidity detected without the activation maneuver and full range of motion not achieved. | LUE |
| | | RLE |
| | | LLE |
| 3.4 FINGER TAPP | ING | |
| perform the task wh<br>thumb 10 times as | niner: Each hand is tested separately. Demonstrate the task, but do not continue to life the patient is being tested. Instruct the patient to tap the index finger on the quickly AND as big as possible. Rate each side separately, evaluating speed, ns, halts and decrementing amplitude. | |
| 0: Normal: | No problems. | |
| 1: Slight: | Any of the following: a) the regular rhythm is broken with one or two interruptions or hesitations of the tapping movement; b) slight slowing; c) the amplitude decrements near the end of the 10 taps. | R |
| 2: Mild: | Any of the following: a) 3 to 5 interruptions during tapping; b) mild slowing; c) the amplitude decrements midway in the 10-tap sequence. | |
| 3: Moderate: | Any of the following: a) more than 5 interruptions during tapping or at least one longer arrest (freeze) in ongoing movement; b) moderate slowing; c) the amplitude decrements starting after the 1st tap. | L |
| 4: Severe: | Cannot or can only barely perform the task because of slowing, interruptions or decrements. | |

July 1, 2008 Copyright © 2008 International Parkinson and Movement Disorder Society. All rights reserved Page 20
This scale may not be copied, distributed or otherwise used in whole or in part without prior written consent of the International Parkinson and Movement Disorder Society.

| 3.5 HAND MOVE | MENTS | SCORE |
|---|---|---|
| perform the task will<br>bent at the elbow's<br>AND as quickly as | miner. Test each hand separately. Demonstrate the task, but do not continue to nile the patient is being tested. Instruct the patient to make a tight fist with the arm to that the palm faces the examiner. Have the patient open the hand 10 times as fully possible. If the patient fails to make a tight fist or to open the hand fully, remind him/each side separately, evaluating speed, amplitude, hesitations, halts and itude. | |
| 0: Normal: | No problem. | |
| 1: Slight: | Any of the following: a) the regular rhythm is broken with one or two interruptions or hesitations of the movement; b) slight slowing; c) the amplitude decrements near the end of the task. | R |
| 2: Mild: | Any of the following: a) 3 to 5 interruptions during the movements; b) mild slowing; c) the amplitude decrements midway in the task. | |
| 3: Moderate: | Any of the following: a) more than 5 interruptions during the movement or at least one longer arrest (freeze) in ongoing movement; b) moderate slowing; c) the amplitude decrements starting after the 1st open-and-close sequence. | L |
| 4: Severe: | Cannot or can only barely perform the task because of slowing, interruptions or decrements. | |
| perform the task with the his/her body with the | niner: Test each hand separately. Demonstrate the task, but do not continue to nile the patient is being tested. Instruct the patient to extend the arm out in front of ne palms down; then to turn the palm up and down alternately 10 times as fast and as ate each side separately, evaluating speed, amplitude, hesitations, halts and litude. | |
| 0: Normal: | No problems. | |
| 1: Slight: | Any of the following: a) the regular rhythm is broken with one or two interruptions or hesitations of the movement; b) slight slowing; c) the amplitude decrements near the end of the sequence. | |
| 2: Mild: | Any of the following: a) 3 to 5 interruptions during the movements; b) mild slowing; c) the amplitude decrements midway in the sequence. | R |
| 3: Moderate: | Any of the following: a) more than 5 interruptions during the movement or at least one longer arrest (freeze) in ongoing movement; b) moderate slowing c) the amplitude decrements starting after the 1st supination-pronation sequence. | |
| 4; Severe: | Cannot or can only barely perform the task because of slowing, interruptions or decrements. | L |

July 1, 2008 Copyright © 2008 International Parkinson and Movement Disorder Society. All rights reserved: Page 21
This scale may not be copied, distributed or otherwise used in whole or in part without prior written consent of the International Parkinson and Movement Disorder Novety

| 3.7 TOE TAPPING | | SCORE |
|---|---|---|
| Test each foot separ<br>patient is being teste<br>then tap the toes 10 | tiner: Have the patient sit in a straight-backed chair with arms, both feet on the floor. rately. Demonstrate the task, but do not continue to perform the task while the ed. Instruct the patient to place the heel on the ground in a comfortable position and times as big and as fast as possible. Rate each side separately, evaluating speed, hs, halts and decrementing amplitude. | |
| <ul><li>0: Normal:</li><li>1: Slight:</li><li>2: Mild:</li><li>3: Moderate:</li><li>4: Severe:</li></ul> | No problem. Any of the following: a) the regular rhythm is broken with one or two interruptions or hesitations of the tapping movement; b) slight slowing; c) amplitude decrements near the end of the ten taps. Any of the following: a) 3 to 5 interruptions during the tapping movements; b) mild slowing; c) amplitude decrements midway in the task. Any of the following: a) more than 5 interruptions during the tapping movements or at least one longer arrest (freeze) in ongoing movement; b) moderate slowing; c) amplitude decrements after the first tap. Cannot or can only barely perform the task because of slowing, interruptions or decrements. | R |
| have both feet comfo<br>continue to perform<br>ground in a comforta | tiner: Have the patient sit in a straight-backed chair with arms. The patient should ortably on the floor. Test each leg separately. Demonstrate the task, but do not the task while the patient is being tested. Instruct the patient to place the foot on the able position and then raise and stomp the foot on the ground 10 times as high and Rate each side separately, evaluating speed, amplitude, hesitations, halts and tude. No problems. Any of the following: a) the regular rhythm is broken with one or two interruptions or hesitations of the movement; b) slight slowing; c) amplitude decrements near the end of the task. Any of the following: a) 3 to 5 interruptions during the movements; b) mild slowness; c) amplitude decrements midway in the task. Any of the following: a) more than 5 interruptions during the movement or at least one longer arrest (freeze) in ongoing movement; b) moderate slowing in speed; c) amplitude decrements after the first tap. Cannot or can only barely perform the task because of slowing, interruptions or decrements. | R L |

July 1, 2008 Copyright © 2008 International Parkinson and Movement Disorder Society. All rights reserved Page 2.
This scale may not be copied, distributed or otherwise used in whole or in part without prior written consent of the International Parkinson and Movement Disorder Society.

| 3.9 ARISING F | ROM CHAIR | SCORE |
|---|---|---|
| floor and sitting I<br>across the chest<br>to two more time<br>folded across the<br>push off using hi | Arising is slower than normal; or may need more than one attempt; or may need to move forward in the chair to arise. No need to use the arms of the chair. Pushes self up from arms of chair without difficulty. te: Needs to push off, but tends to fall back; or may have to try more than one time using arms of chair, but can get up without help. | |
| towards the exa<br>simultaneously.<br>the examiner. T<br>heel strike durin | Independent walking with minor gait impairment. Independent walking but with substantial gait impairment. | |

July 1, 2008 Copyright © 2008 International Parkinson and Movement Disorder Society. All rights reserved. Page 2
This scale may not be copied, distributed or otherwise used in whole or in part without prior written consent of the International Parkinson and Movement Disorder Novatje

| 3.11 FREEZING OF G | AIT | SCORE |
|---|---|---|
| episodes. Observe for the end of the task. To assessment. 0; Normal: 1: Slight: 2: Mild: 3: Moderate: | er: While assessing gait, also assess for the presence of any gait freezing start hesitation and stuttering movements especially when turning and reaching of the extent that safety permits, patients may NOT use sensory tricks during the No freezing. Freezes on starting, turning or walking through doorway with a single halt during any of these events, but then continues smoothly without freezing during straight walking. Freezes on starting, turning or walking through doorway with more than one halt during any of these activities, but continues smoothly without freezing during straight walking. Freezes once during straight walking. Freezes multiple times during straight walking. | |
| a quick, forceful pull on comfortably apart and put the patient on what is a falling. There should be observation of the numpurposely milder and patient to flex the body backwards or falling. Latings begin with three test so that the rating is | er: The test examines the response to sudden body displacement produced by the shoulders while the patient is standing erect with eyes open and feet parallel to each other. Test retropulsion. Stand behind the patient and instruct about to happen. Explain that s/he is allowed to take a step backwards to avoid a solid wall behind the examiner, at least 1-2 meters away to allow for the liber of retropulsive steps. The first pull is an instructional demonstration and is of rated. The second time the shoulders are pulled briskly and forcefully towards up force to displace the center of gravity so that patient MUST take a step inter needs to be ready to catch the patient, but must stand sufficiently back so as or the patient to take several steps to recover independently. Do not allow the abnormally forward in anticipation of the pull. Observe for the number of steps up to and including two steps for recovery is considered normal, so abnormal a steps. If the patient falls to understand the test, the examiner can repeat the shaded on an assessment that the examiner feels reflects the patient's limitations anding or lack of preparedness. Observe standing posture for item 3.13 No problems: Recovers with one or two steps. 3-5 steps, but subject recovers unaided. More than 5 steps, but with absence of postural response; falls if not caught by examiner. Very unstable, tends to lose balance spontaneously or with just a gentle pull on the shoulders. | |

July 1, 2009 Copyright © 2008 International Parkinson and Movement Disorder Society. All rights reserved: Page 24
This scale may not be copied, distributed or otherwise used in whole or in part without prior written consent of the International Parkinson and Movement Disorder Society.

| 3.13 POSTURE | | SCORE |
|---|---|---|
| during walking, and while to stand up straight and se | Posture is assessed with the patient standing erect after arising from a chair, being tested for postural reflexes. If you notice poor posture, tell the patient ee if the posture improves (see option 2 below). Rate the worst posture seen points. Observe for flexion and side-to-side leaning. | |
| 0: Normal: No j | problems. | |
| 1: Slight: Not | quite erect, but posture could be normal for older person. | |
| | finite flexion, scoliosis or leaning to one side, but patient can correct posture normal posture when asked to do so. | |
| | oped posture, scoliosis or leaning to one side that cannot be corrected tionally to a normal posture by the patient. | |
| 4: Severe: Flex | xion, scoliosis or leaning with extreme abnormality of posture. | |
| 3.14 GLOBAL SPONTAN | NEITY OF MOVEMENT (BODY BRADYKINESIA) | |
| small amplitude and pover<br>the legs. This assessmen | This global rating combines all observations on slowness, hesitancy, and rty of movement in general, including a reduction of gesturing and of crossing it is based on the examiner's global impression after observing for itle sitting, and the nature of arising and walking. | |
| 0: Normal: No | problems. | |
| 1: Slight: Slig | ght global slowness and poverty of spontaneous movements. | |
| 2: Mild: Mil | ld global slowness and poverty of spontaneous movements. | |
| 3: Moderate: Mo | oderate global slowness and poverty of spontaneous movements. | |
| 4: Severe: Se | evere global slowness and poverty of spontaneous movements. | |
| 3.15 POSTURAL TREMO | OR OF THE HANDS | |
| | All tremor, including re-emergent rest tremor, that is present in this posture is | |
| to be included in this rating. Rate each hand separately. Rate the highest amplitude seen. Instruct the patient to stretch the arms out in front of the body with palms down. The wrist should be straight and the fingers comfortably separated so that they do not touch each other. Observe this posture for 10 seconds | | |
| 0: Normal: No | tremor. | R |
| 1: Slight: Tre | emor is present but less than 1 cm in amplitude. | |
| 2: Mild: Tre | emor is at least 1 but less than 3 cm in amplitude. | |
| 3: Moderate: Tre | emor is at least 3 but less than 10 cm in amplitude. | Ļ |
| 4: Severe: Tre | emor is at least 10 cm in amplitude. | L |

July 1, 2008 Copyright © 2008 International Parkinson and Movement Disorder Society. All rights reserved. Page 25
This scale may not be copied, distributed or otherwise used in whole or in part without prior written consent of the International Parkinson and Movement Disorder Society.

| 3.16 KINETIC TREMOR OF THE HANDS | SCORE |
|---|---|
| Instructions to examiner: This is tested by the finger-to-nose maneuver. With the arm starting from the outstretched position, have the patient perform at least three finger-to-nose maneuvers with each hand reaching as far as possible to touch the examiner's finger. The finger-to-nose maneuver should be performed slowly enough not to hide any tremor that could occur with very fast arm movements. Repeat with the other hand, rating each hand separately. The tremor can be present throughout the movement or as the tremor reaches either target (nose or finger). Rate the highest amplitude seen. | |
| 0: Normal: No tremor. | |
| 1: Slight: Tremor is present but less than 1 cm in amplitude. | R |
| 2: Mild: Tremor is at least 1 but less than 3 cm in amplitude. | |
| 3: Moderate: Tremor is at least 3 but less than 10 cm in amplitude. | |
| 4: Severe: Tremor is at least 10 cm in amplitude. | L |
| 3.17 REST TREMOR AMPLITUDE | |
| Instructions to examiner: This and the next item have been placed purposefully at the end of the examination to allow the rater to gather observations on rest tremor that may appear at any time during the exam, including when quietly sitting, during walking and during activities when some body parts are moving but others are at rest. Score the maximum amplitude that is seen at any time as the final score. Rate only the amplitude and not the persistence or the intermittency of the tremor. As part of this rating, the patient should sit quietly in a chair with the hands placed on the arms of the chair (not in the lap) and the feet comfortably supported on the floor for 10 seconds with no other directives. Rest tremor is assessed separately for all four limbs and also for the lip/jaw. Rate only the maximum amplitude that is seen at any time as the final rating. | RUE |
| Extremity ratings | |
| 0: Normal: No tremor. | LUE |
| 1: Slight: ≤ 1 cm in maximal amplitude. | |
| 2: Mild: > 1 cm but < 3 cm in maximal amplitude. | |
| 3: Moderate: 3 - 10 cm in maximal amplitude. | RLE |
| 4: Severe: > 10 cm in maximal amplitude. | RLE |
| Lip/Jaw ratings | |
| 0: Normal: No tremor. | LLE |
| 1: Slight: ≤1 cm in maximal amplitude. | |
| 2: Mild: > 1 cm but ≤ 2 cm in maximal amplitude. | |
| 3: Moderate: > 2 cm but ≤ 3 cm in maximal amplitude. | Lip/Jaw |
| 4: Severe: > 3 cm in maximal amplitude. | |

July 1, 2008 Copyright © 2008 International Parkinson and Movement Disorder Society. All rights reserved. Page 26
This scale may not be copied, distributed or otherwise used in whole or in part without prior written consent of the International Parkinson and Movement Disorder Society.

| rest tremor during | ner: This item receives one rating for all rest tremor and focuses on the constancy the examination period when different body parts are variously at rest. It is rated ad of the examination so that several minutes of information can be coalesced into No tremor. Tremor at rest is present ≤ 25% of the entire examination period. |
|---|---|
| 1: Slight:<br>2: Mild: | |
| 2: Mild: | Tremor at rest is present ≤ 25% of the entire examination period. |
| 3: Moderate: | Tremor at rest is present 26-50% of the entire examination period. |
| 5. Moderate. | Tremor at rest is present 51-75% of the entire examination period. |
| 4: Severe: | Tremor at rest is present > 75% of the entire examination period. |
| YSKINESIA IMPAC | T ON PART III RATINGS |
| A. Were dyskin | esias (chorea or dystonia) present during examination? |
| B. If yes, did the | ese movements interfere with your ratings? |
| DEHN AND YAHR | STAGE |
| 0: Asymptomatic | |
| 1: Unilateral inve | olvement only |
| 2: Bilateral invol | vement without impairment of balance. |
| | ate involvement; some postural instability but physically independent; needs recover from pull test. |
| 4: Severe disabi | lity, still able to walk or stand unassisted. |
| 5: Wheelchair bo | ound or bedridden unless aided. |

July 1, 2008 Copyright © 2008 International Parkinson and Movement Disorder Society. All rights reserved. Page 27
This scale may not be copied, distributed or otherwise used in whole or in part without prior written consent of the International Parkinson and Movement Disorder Novett

### Part IV: Motor Complications

Overview and Instructions: In this section, the rater uses historical and objective information to assess two motor complications, dyskinesias and motor fluctuations that include OFF-state dystonia. Use all information from patient, caregiver, and the examination to answer the six questions that summarize function over the past week including today. As in the other sections, rate using only integers (no half points allowed) and leave no missing ratings. If the item cannot be rated, place UR for Unable to Rate. You will need to choose some answers based on percentages, and therefore you will need to establish how many hours generally are awake hours and use this figure as the denominator for "OFF" time and dyskinesias. For "OFF dystonia", the total "Off" time will be the denominator. Operational definitions for examiner's use.

Dyskinesias: Involuntary random movements

Words that patients often recognize for dyskinesias include "irregular jerking", "wiggling", "twitching". It is essential to stress to the patient the difference between dyskinesias and tremor, a common error when patients are assessing dyskinesias.

Dystonia: contorted posture, often with a twisting component:

Words that patients often recognize for dystonia include "spasms", "cramps", "posture".

Motor fluctuation: Variable response to medication:

Words that patients often recognize for motor fluctuation include "wearing out", "wearing off", "roller-coaster effect", "on-off", "uneven medication effects".

OFF: Typical functional state when patients have a poor response in spite of taking mediation or the typical functional response when patients are on NO treatment for parkinsonism. Words that patients often recognize include "low time", "bad time", "shaking time", "slow time", "time when my medications don't work."

ON: Typical functional state when patients are receiving medication and have a good response: Words that patients often recognize include "good time", "walking time", "time when my medications work."

#### A. DYSKINESIAS [exclusive of OFF-state dystonia]

| | SCORE |
|---|---|
| 4.1 TIME SPENT WITH DYSKINESIAS | |
| Instructions to examiner: Determine the hours in the usual waking day and then the hours of dyskinesias. Calculate the percentage. If the patient has dyskinesias in the office, you can point them out as a reference to ensure that patients and caregivers understand what they are rating. You may also use your own acting skills to enact the dyskinetic movements you have seen in the patient before or show them dyskinetic movements typical of other patients. Exclude from this question early morning and nighttime painful dystonia. | |
| Instructions to patient [and caregiver]: Over the past week, how many hours do you usually sleep on a daily basis, including nighttime sleep and daytime napping? Alright, if you sleep hrs, you are awake hrs. Out of those awake hours, how many hours in total do you have wiggling, twitching or jerking movements? Do not count the times when you have tremor, which is a regular back and forth shaking or times when you have painful foot cramps or spasms in the early morning or at nighttime. I will ask about those later. Concentrate only on these types of wiggling, jerking and irregular movements. Add up all the time during the waking day when these usually occur. How many hours (use this number for your calculations). | |
| 0: Normal: No dyskinesias. | |
| 1: Slight: ≤ 25% of waking day. | |
| 2: Mild: 26 - 50% of waking day. 1. Total Hours Awake: | |
| 3: Moderate: 51 - 75% of waking day. 2. Total Hours with Dyskinesia: | |
| 4: Severe: > 75% of waking day. 3. % Dyskinesia = ((2/1)*100): | |

July 1, 2008 Copyright © 2008 International Parkinson and Movement Disorder Society. All rights reserved Page 28
This scale may not be copied, distributed or otherwise used in whole or in part without prior written consent of the International Parkinson and Movement Disorder Society

| 4.2 FUNCTIONAL IMPACT OF DYSKINESIAS | | |
|---|---|---|
| Instructions to examiner: Determine the degree to which dyskinesias impact on the patient's daily function in terms of activities and social interactions. Use the patient's and caregiver's response to your question and your own observations during the office visit to arrive at the best answer. | | |
| Instructions to patient [and caregiver]: Over the past week, did you usually have trouble doing things or being with people when these jerking movements occurred? Did they stop you from doing things or from being with people? | | |
| 0: Normal: | No dyskinesias or no impact by dysl | kinesias on activities or social interactions. |
| 1: Slight: | | es, but the patient usually performs all al interactions during dyskinetic periods. |
| 2: Mild: | | es, but the patient usually performs all<br>al interactions during dyskinetic periods. |
| 3: Moderat | | he point that the patient usually does not usually participate in some social activities |
| 4: Severe: | Dyskinesias impact on function to tr<br>perform most activities or participate<br>dyskinetic episodes. | ne point that the patient usually does not<br>e in most social interactions during |
| | B. MOTOR FLU | ICTUATIONS |
| 4.3 TIME SPEN | T IN THE OFF STATE | |
| Instructions to examiner: Use the number of waking hours derived from 4.1 and determine the hours spent in the "OFF" state. Calculate the percentage. If the patient has an OFF period in the office, you can point to this state as a reference. You may also use your knowledge of the patient to describe a typical OFF period. Additionally you may use your own acting skills to enact an OFF period you have seen in the patient before or show them OFF function typical of other patients. Mark down the typical number of OFF hours, because you will need this number for completing 4.6. | | |
| Instructions to patient [and caregiver]: Some patients with Parkinson's disease have a good effect from their medications throughout their awake hours and we call that "ON" time. Other patients take their medications but still have some hours of low time, bad time, slow time or shaking time. Doctors call these low periods "OFF" time. Over the past week, you told me before that you are general awake hrs each day. Out of these awake hours, how many hours in total do you usually have this type of low level or OFF function (use this number for your calculations). | | |
| 0: Normal: | No OFF time. | |
| 1: Slight: | ≤ 25% of waking day. | |
| 2: Mild: | 26 - 50% of waking day. | |
| 3: Moderate | : 51 - 75% of waking day. | Total Hours Awake: |
| 4: Severe: | > 75% of waking day. | 2. Total Hours OFF: |
| | | 3. % OFF = ((2/1)*100): |

July 1, 2008 Copyright © 2008 International Parkinson and Movement Disorder Society. All rights reserved Page 29
This scale may not be copied, distributed or otherwise used in whole or in part without prior written consent of the International Parkinson and Movement Disorder Society

| 4.4 FUNCTIONAL I | MPACT OF FLUCTUATIONS | SCORE |
|---|---|---|
| Instructions to examiner: Determine the degree to which motor fluctuations impact on the patient's daily function in terms of activities and social interactions. This question concentrates on the difference between the ON state and the OFF state. If the patient has no OFF time, the rating must be 0, but if patients have very mild fluctuations, it is still possible to be rated 0 on this item if no impact on activities occurs. Use the patient's and caregiver's response to your question and your own observations during the office visit to arrive at the best answer. | | |
| the past week. Do y<br>the rest of the day w | nt <u>fand caregiver</u> ]. Think about when those low or "OFF" periods have occurred over<br>you usually have more problems doing things or being with people than compared to<br>hen you feel your medications working? Are there some things you usually do<br>I that you have trouble with or stop doing during a low period? | |
| 0: Normal: | No fluctuations or No impact by fluctuations on performance of activities or social interactions. | |
| 1: Slight: | Fluctuations impact on a few activities, but during OFF, the patient usually performs all activities and participates in all social interactions that typically occur during the ON state | |
| 2: Mild: | Fluctuations impact many activities, but during OFF, the patient still usually performs all activities and participates in all social interactions that typically occur during the ON state. | |
| 3: Moderate: | Fluctuations impact on the performance of activities during OFF to the point that the patient usually does not perform some activities or participate in some social interactions that are performed during ON periods. | |
| 4: Severe: | Fluctuations impact on function to the point that, during OFF, the patient usually does not perform most activities or participate in most social interactions that are performed during ON periods. | |
| 4.5 COMPLEXITY | OF MOTOR FLUCTUATIONS | |
| of day, food intake of<br>supplement with you<br>a special time, most<br>from mild), only som | iner: Determine the usual predictability of OFF function whether due to dose, time rother factors. Use the information provided by the patients and caregiver and ir own observations. You will ask if the patient can count on them always coming at y coming at a special time (in which case you will probe further to separate slight etimes coming at a special time or are they totally unpredictable? Narrowing down allow you to find the correct answer. | |
| times during day or w<br>know when your low | at [and caregiver]: For some patients, the low or "OFF" periods happen at certain when they do activities like eating or exercising. Over the past week, do you usually periods will occur? In other words, do your low periods <u>allways</u> come at a certain ty come at a certain time? Do they <u>only sometimes</u> come at a certain time? Are ally unpredictable?" | |
| 0: Normal: | No motor fluctuations. | |
| 1: Slight: | OFF times are predictable all or almost all of the time (> 75%). | |
| 2; Mild; | OFF times are predictable most of the time (51-75%). | |
| 3: Moderate: | OFF times are predictable some of the time (26-50%). | |
| 4: Severe: | OFF episodes are rarely predictable (≤ 25%). | |

July 1, 2008 Copyright © 2008 International Parkinson and Movement Disorder Society. All rights reserved. Page 3
This scale may not be copied, distributed or otherwise used in whole or in part without prior written consent of the International Parkinson and Movement Disorder Novatje

| C. "OFF" DYSTONIA | |
|---|---|
| 4.6 PAINFUL OFF-STATE DYSTONIA Instructions to examiner: For patients who have motor fluctuations, determine what proportion of the OFF episodes usually includes painful dystonia? You have already determined the number of hours of "OFF" time (4.3). Of these hours, determine how many are associated with dystonia and calculate the percentage. If there is no OFF time, mark 0. Instructions to patient fand caregiver! In one of the questions I asked earlier, you said you generally have hours of low or "OFF" time when your Parkinson's disease is under poor control. During these low or "OFF" periods, do you usually have painful cramps or spasms? Out of the total hrs of this low time, if you add up all the time in a day when these painful cramps come, how many hours would this make? □: Normal: No dystonia OR NO OFF TIME. 1: Slight: ≤ 25% of time in OFF state. 2: Mild: 26-50% of time in OFF state. 3: Moderate: 51-75% of time in OFF state. | |
| | Total Hours Off: Total Off Hours w/Dystonia: W Off Dystonia = ((2/1)*100): |
| Summary statement to patient: READ TO PATIENT This completes my rating of your Parkinson's disease. I know the questions and tasks have taken several minutes, but I wanted to be complete and cover all possibilities. In doing so, I may have asked about problems you do not even have, and I may have mentioned problems that you may never develop at all. Not all patients develop all these problems, but because they can occur, it is important to ask all the questions to every patient. Thank you for your time and attention in completing this scale with me. | |

July 1, 2008 Copyright © 2008 International Parkinson and Movement Disorder Society. All rights reserved. Page 3
This scale may not be copied, distributed or otherwise used in whole or in part without prior written consent of the International Parkinson and Movement Disorder Novatje

## MDS UPDRS Score Sheet

| MIDS | OPDRS Score Sheet | | | | |
|---|---|---|---|---|---|
| 1.A | Course of information | Patient | | Rigidity- RUE | |
| 1.A | Source of information | Caregiver Patient + Caregiver | 3.3c | Rigidity- LUE | |
| Part I | | | 3.3d | Rigidity- RLE | |
| 1.1 | Cognitive impairment | | 3.3e | Rigidity- LLE | |
| 1.2 | Hallucinations and psychosis | | 3.4a | Finger tapping- Right hand | |
| 1.3 | Depressed mood | | 3.4b | Finger tapping- Left hand | |
| 1.4 | Anxious mood | | 3.5a | Hand movements- Right hand | |
| 1.5 | Apathy | | 3.5b | Hand movements- Left hand | |
| 1.6 | Features of DDS | | 3.6a | Pronation- supination movements— Right hand | |
| 1.6a | Who is filling out questionnaire | Patient Caregiver | 3.6b<br>3.7a | Pronation- supination movements- Left hand | |
| | | Patient + Caregiver | | Toe tapping- Right foot | |
| 1.7 | Sleep problems | | 3.7b | Toe tapping - Left foot | |
| 1.8 | Daytime sleepiness | | 3.8a | Leg agility- Right leg | |
| 1.9 | Pain and other sensations | | 3.8b | Leg agility– Left leg | |
| 1.10 | Urinary problems | | 3.9 | Arising from chair | |
| 1.11 | Constipation problems | | 3.10 | Gait | |
| 1.12 | Light headedness on standing | | 3,11 | Freezing of gait | |
| 1.13 | Fatigue | | 3.12 | Postural stability | |
| Part II | | | 3.13 | Posture | |
| 2.1 | Speech | | 3.14 | Global spontaneity of movement | |
| 2.2 | Saliva and drooling | | 3.15a | Postural tremor– Right hand | |
| 2.3 | Chewing and swallowing | | 3.15b | Postural tremor– Left hand | |
| 2.4 | Eating tasks | | 3.16a | Kinetic tremor- Right hand | |
| 2.5 | Dressing | | 3.1 <b>6</b> b | Kinetic tremor- Left hand | |
| 2.6 | Hygiene | | 3.17a | Rest tremor amplitude- RUE | |
| 2.7 | Handwriting | | 3.17b | Rest tremor amplitude- LUE | |
| 2.8 | Doing hobbies and other activities | | 3.17c | Rest tremor amplitude- RLE | |
| 2.9 | Turning in bed | | 3.17d | Rest tremor amplitude- LLE | |
| 2.10 | Tremor | | 3.17e | Rest tremor amplitude– Lip/jaw | |
| 2.11 | Getting out of bed | | 3.18 | Constancy of rest | |
| 2.12 | Walking and balance | | | Were dyskinesias present? | □No □Yes |
| 2.13 | Freezing | | | Did these movements interfere with ratings? | □No□Yes |
| 3a | Is the patient on medication? | □ No □ Yes | | Hoehn and Yahr Stage | |
| 3b | Patient's clinical state | □off □on | Part IV | <u> </u> | |
| Зс | Is the patient on Levodopa? | □No □Yes | 4.1 | Time spent with dyskinesias | |
| 3.01 | If yes, minutes since last dose: | | 4.2 | Functional impact of dyskinesias | |
| Part III | | | 4.3 | Time spent in the OFF state | |
| 3.1 | Speech | | 4.4 | Functional impact of fluctuations | |
| 3.2 | Facial expression | | 4.5 | Complexity of motor fluctuations | |
| 3.3a | Rigidity- Neck | | 4.6 | Painful OFF-state dystonia | |

July 1, 2008

Councied © 2008 International Parkinger and Managed Disorder Society, All sights recognish

Copyright © 2008 International Parkinson and Minement Disorder Society. All rights reserved.
This scale may not be copied, distributed or otherwise used in whole or in part without prior written consent of the International Parkinson and Movement Disorder Society

# APPENDIX F. PATIENT GLOBAL IMPRESSION OF CHANGE (PGI-C)

The subject will independently rate the following question of Patient Global Impression of Change (PGI-C) based on his/her overall impression at Visit 5 (Week 10), Visit 6 (Week 15), and Visit 7 (Week 20) or early discontinuation.

# **Patient Global Impression of Change:**

Compared to your condition prior to your starting on this study, how much has your condition changed with your current treatment?

| <b>1</b> | <b>2</b> | <b>3</b> | <b>4</b> | <b>5</b> | <b>G</b> 6 | <b>1</b> 7 |
|---|---|---|---|---|---|---|
| Very<br>Much<br>Worse | Much<br>Worse | Minimally<br>Worse | No<br>Change | Minimally<br>Improved | Much<br>Improved | Very<br>Much<br>Improved |

















# APPENDIX K. GASTROPARESIS CARDINAL SYMPTOM INDEX (GCSI)

## **GCSI**

This questionnaire asks you about the severity of symptoms you may have related to your gastrointestinal problem. There are no right or wrong answers. Please answer each question as accurately as possible.

For each symptom, please <u>circle the number</u> that best describes how <u>severe</u> the symptom has been during the past 2 weeks. If you have not experienced this symptom, circle 0. If the symptom has been very mild, circle 1. If the symptom has been mild, circle 2. If it has been moderate, circle 3. If it has been severe, circle 4. If it has been very severe, circle 5. Please be sure to answer every question.

Please rate the severity of the following symptoms during the past 2 weeks.

| | None | Very<br>Mild | Mild | Moderate | Severe | VerySevere |
|---|---|---|---|---|---|---|
| nausea (feeling sick to your stomach<br>as if you were going to vomit or<br>throw up) | 0 | 1 | 2 | 3 | 4 | 5 |
| retching (heaving as if to vomit, but<br>nothing comes up) | 0 | 1 | 2 | 3 | 4 | 5 |
| 3. vomiting | 0 | 1 | 2 | 3 | 4 | 5 |
| 4. stomach fullness | 0 | l | 2 | 3 | 4 | 5 |
| 5. not able to finish a normal-sized meal | 0 | 1 | 2 | 3 | 4 | 5 |
| <ol><li>feeling excessively full after meals</li></ol> | 0 | 1 | 2 | 3 | 4 | 5 |
| 7. loss of appetite | 0 | 1 | 2 | 3 | 4 | 5 |
| bloating (feeling like you need to loosen your clothes) | 0 | 1 | 2 | 3 | 4 | 5 |
| 9. stomach or belly visibly larger | 0 | 1 | 2 | 3 | 4 | 5 |

Revicki DA, Rentz AM, Dubois D, Kahrilas P, Stanghellini V, Talley NJ, Tack J. Gastroparesis Cardinal Symptom Index (GCSI): development and validation of a patient reported assessment of seventy of gastroparesis symptoms. Qual Life Res. 2004;13(4):833-44

Revicki DA, Rentz AM, Dubois D, Kahrilas P, Stanghellini V, Talley NJ, Tack J. Development and validation of a patient-assessed gastroparesis symptom severity measure: the Gastroparesis Cardinal Symptom Index. Aliment Pharmacol Ther. 2003;18(1):141-50

GCSI © 2001 Mapi Research Trust, All rights reserved

The Questionnaire contact information and permission to use: Mapi Research Trust, Lyon, France – Internet: <a href="https://eorovide.mapi-trust.org">https://eorovide.mapi-trust.org</a>

Impax\_IPX203-B16-02\_GCSI\_English (US)\_Version 1.1\_09AUG2018 CONFIDENTIAL

Page 1 of 1












# APPENDIX O. COLUMBIA-SUICIDE SEVERITY RATING SCALE (C-SSRS)

# COLUMBIA-SUICIDE SEVERITY RATING SCALE (C-SSRS)

Baseline/Screening Version

Version 1/14/09

Posner, K.; Brent, D.; Lucas, C.; Gould, M.; Stanley, B.; Brown, G.; Fisher, P.; Zelazny, J.; Burke, A.; Oquendo, M.; Mann, J.

#### Disclaimer:

This scale is intended to be used by individuals who have received training in its administration. The questions contained in the Columbia-Suicide Severity Rating Scale are suggested probes. Ultimately, the determination of the presence of suicidal ideation or behavior depends on the judgment of the individual administering the scale.

Definitions of behavioral suicidal events in this scale are based on those used in <u>The Columbia Suicide History Form</u>, developed by John Mann, MD and Maria Oquendo, MD, Conte Center for the Neuroscience of Mental Disorders (CCNMD), New York State Psychiatric Institute, 1051 Riverside Drive, New York, NY, 10032. (Oquendo M. A., Halberstam B. & Mann J. J., Risk factors for suicidal behavior: utility and limitations of research instruments. In M.B. First [Ed.] Standardized Evaluation in Clinical Practice, pp. 103-130, 2003.)

For reprints of the C-SSRS contact Kelly Posner, Ph.D., New York State Psychiatric Institute, 1051 Riverside Drive, New York, New York, 10032; inquiries and training requirements contact posnerk@nyspi.columbia.edu

© 2008 The Research Foundation for Mental Hygiene, Inc.

| SUICIDAL IDEATION | | and the | | | |
|---|---|---|---|---|---|
| Ask questions 1 and 2. If both are negative, proceed to question 2 is "yes", ask questions 3, 4 and 5. If the ans "Intensity of Ideation" section below. | | He/SI | e: Time<br>be Felt<br>Suicidal | Pas<br>Moi | |
| 1. Wish to be Dead Subject endorses thoughts about a wish to be dead or not alive anym. Have you wished you were dead or wished you could go to sleep an | | Yes | No | Yes | No 🗆 |
| If yes, describe: | | | | | |
| 2. Non-Specific Active Suicidal Thoughts General non-specific thoughts of wanting to end one's life/commit so of ways to kill onesel?associated methods, intent, or plan during the Have you actually had any thoughts of killing yoursel?? | | Yes | No | Yes | No |
| If yes, describe: | | | | | |
| 3. Active Suicidal Ideation with Any Methods (Not Pla Subject endorses thoughts of suicide and has thought of at least one r specific plan with time, place or method details worked out (e.g. tho who would say, "I thought about taking an overdose but I never madit and I would never go through with it." Have you been thinking about how you might do this? If yes, describe: | nethod during the assessment period. This is different than a<br>ught of method to kill self but not a specific plan). Includes person | Yes | No | Yes | No |
| 4. Active Suicidal Ideation with Some Intent to Act, we Active suicidal thoughts of killing oneself and subject reports having thoughts but I definitely will not do anything about them." Have you had these thoughts and had some intention of acting on the second secon | some intent to act on such thoughts, as opposed to "I have the | Yes | No<br>□ | Yes | No |
| If yes, describe: | | | | | |
| 5. Active Suicidal Ideation with Specific Plan and Inte Thoughts of killing oneself with details of plan fully or partially worl Have you started to work out or worked out the details of how to kill If yes, describe: | ked out and subject has some intent to carry it out. | Yes | No | Yes | No |
| 1,74,444 | | | | | |
| The following features should be rated with respect to the mo the least severe and 5 being the most severe). Ask about time Lifetime - Most Severe Ideation: Type # (1-5) Pest X Months - Most Severe Ideation: | | | lost<br>vere | EDWC9C9ANS | ost<br>⁄ere |
| Type # (1-5) | Description of Ideation | | | | |
| Frequency How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in | week (4) Daily or almost daily (5) Many times each day | | | _ | |
| Duration When you have the thoughts how long do they last? (1) Fleeting - few seconds or minutes (2) Less than 1 hour/some of the time (3) 1-4 hours/a lot of time | (4) 4-8 hours/most of day<br>(5) More than 8 hours/persistent or continuous | | | - | - |
| Controllability Could/can you stop thinking about killing yourself or wa (1) Easily able to control thoughts (2) Can control thoughts with little difficulty (3) Can control thoughts with some difficulty | (4) Can control thoughts with a lot of difficulty (5) Unable to control thoughts (0) Does not attempt to control thoughts | 4110<br>1111<br>1111<br>1111<br>1111 | | - | -<br>- |
| Deterrents Are there things - anyone or anything (e.g., family, religited or acting on thoughts of committing suicide? (1) Deterrents definitely stopped you from attempting suicide (2) Deterrents probably stopped you (3) Uncertain that deterrents stopped you | (4) Deterrents most likely did not stop you (5) Deterrents definitely did not stop you (0) Does not apply | | | _ | |
| Reasons for Ideation What sort of reasons did you have for thinking about wa or stop the way you were feeling (in other words you cou feeling) or was it to get attention, revenge or a reaction from others (2) Mostly to get attention, revenge or a reaction from others (3) Equally to get attention, revenge or a reaction from others and to end/stop the pain | nting to die or killing yourself? Was it to end the pain<br>Idn't go on living with this pain or how you were<br>from others? Or both? | _ | | | |
| © 2008 Research Foundation for Mental Hygiene, Inc. | C-SSRS—Baseline/Screening (Version 1/14/09) | | | Page | l of 2 |

| SUICIDAL BEHAVIOR (Check all that apply, so long as these are separate events; must ask about all types) | | Life | time | | ars |
|---|---|---|---|---|---|
| Actual Attempt: A potentially self-injurious act committed with at least some wish to die, as a result of act. Behavior was in part thought of as roneself. Intent does not have to be 100%. If there is any intent/desire to die associated with the act, then it can be considered a attempt. There does not have to be any injury or harm, just the potential for injury or harm. If person pulls trigger wh mouth but gun is broken so no injury results, this is considered an attempt. Inferring Intent: Even if an individual denies intent/wish to die, it may be inferred clinically from the behavior or circumstance highly lethal act that is clearly not an accident so no other intent but suicide can be inferred (e.g., gunshot to head, jumping fror high floor/story). Also, if someone denies intent to die, but they thought that what they did could be lethal, intent may be inferred. | in actual suicide<br>ile gun is in<br>s. For example, a<br>n window of a | Yes | No<br>□ | ∜ Yes | No |
| Have you made a suicide attempt? Have you done anything to harm yourself? Have you done anything dangerous where you could have died? What did you do? Did you as a way to end your life? Did you want to die (even a little) when you ? Were you trying to end your life when you ? Or Did you think it was possible you could have died from ? Or did you do it purely for other reasons / without ANY intention of killing yourself (like to relieve stress get sympathy, or get something else to happen)? (Self-Injurious Behavior without suicidal intent) | , feel better, | | l # of<br>empts | | l # of<br>mpts |
| If yes, describe: | | Yes | No | Yes | No |
| Has subject engaged in Non-Suicidal Self-Injurious Behavior? | | Yes | No | Yes | No |
| Interrupted Attempt: When the person is interrupted (by an outside circumstance) from starting the potentially self-injurious act (if not for that, actual have occurred). Overdose: Person has pills in hand but is stopped from ingesting. Once they ingest any pills, this becomes an attempt rather the attempt. Shooting: Person has gun pointed toward self, gun is taken away by someone else, or is somehow prevented from pulli they pull the trigger, even if the gun fails to fire, it is an attempt. Jumping: Person is poised to jump, is grabbed and taken down Hanging: Person has noose around neck but has not yet started to hang - is stopped from doing so. Has there been a time when you started to do something to end your life but someone or something stoppy you actually dld anything? If yes, describe: | an an interrupted<br>ing trigger, Once<br>from ledge. | Tota | I # of | Total | l# of |
| Aborted Attempt: When person begins to take steps toward making a suicide attempt, but stops themselves before they actually have engaged in a destructive behavior. Examples are similar to interrupted attempts, except that the individual stops him/herself, instead of being something else. Has there been a time when you started to do something to try to end your life but you stopped yourself be actually did anything? If yes, describe. | stopped by | | No U # of orted | | No I # of orted |
| Preparatory Acts or Behavior: Acts or preparation towards imminently making a suicide attempt. This can include anything beyond a verbalization or thought assembling a specific method (e.g., buying pills, purchasing a gun) or preparing for one's death by suicide (e.g., giving things a suicide note). Have you taken any steps towards making a suicide attempt or preparing to kill yourself (such as collecting a gun, giving valuables away or writing a suicide note)? If yes, describe: | way, writing a | Yes | No | Yes | No |
| Suicidal Behavior: Suicidal behavior was present during the assessment period? | | Yes | No | Yes | No |
| Answer for Actual Attempts Only | Attempt | Most Leth<br>Attempt<br>Date: | nal | Initial/Fi<br>Attempt<br>Date: | 755-030 |
| Actual Lethality/Medical Damage: 0. No physical damage or very minor physical damage (e.g., surface scratches). 1. Minor physical damage (e.g., lethargic speech; first-degree burns; mild bleeding; sprains). 2. Moderate physical damage; medical attention needed (e.g., conscious but sleepy, somewhat responsive; second-degree burns; bleeding of major vessel). 3. Moderately severe physical damage, medical hospitalization and likely intensive care required (e.g., comatose with reflexes intact; third-degree burns less than 20% of body; extensive blood loss but can recover; major fractures). 4. Severe physical damage; medical hospitalization with intensive care required (e.g., comatose without reflexes; third-degree burns over 20% of body; extensive blood loss with unstable vital signs; major damage to a vital area). 5. Death | Enter Code | Enter C | | Enter | Code |
| Potential Lethality: Only Answer if Actual Lethality=0 Likely lethality of actual attempt if no medical damage (the following examples, while having no actual medical damage, had potential for very serious lethality: put gun in mouth and pulled the trigger but gun fails to fire so no medical damage; laying on train tracks with oncoming train but pulled away before run over). 0 = Behavior not likely to result in injury | Enter Code | Enter ( | Tode | Enter | Code |
| 1 = Behavior likely to result in injury but not likely to cause death 2 = Behavior likely to result in death despite available medical care | | | _ | | |

# COLUMBIA-SUICIDE SEVERITY RATING SCALE (C-SSRS)

Since Last Visit

Version 1/14/09

Posner, K.; Brent, D.; Lucas, C.; Gould, M.; Stanley, B.; Brown, G.; Fisher, P.; Zelazny, J.; Burke, A.; Oquendo, M.; Mann, J.

#### Disclaimer:

This scale is intended to be used by individuals who have received training in its administration. The questions contained in the Columbia-Suicide Severity Rating Scale are suggested probes. Ultimately, the determination of the presence of suicidal ideation or behavior depends on the judgment of the individual administering the scale.

Definitions of behavioral suicidal events in this scale are based on those used in <u>The Columbia Suicide History Form</u>, developed by John Mann, MD and Maria Oquendo, MD, Conte Center for the Neuroscience of Mental Disorders (CCNMD), New York State Psychiatric Institute, 1051 Riverside Drive, New York, NY, 10032. (Oquendo M. A., Halberstam B. & Mann J. J., Risk factors for suicidal behavior: utility and limitations of research instruments. In M.B. First [Ed.] Standardized Evaluation in Clinical Practice, pp. 103-130, 2003.)

For reprints of the C-SSRS contact Kelly Posner, Ph.D., New York State Psychiatric Institute, 1051 Riverside Drive, New York, New York, 10032; inquiries and training requirements contact posnerk@nyspi.columbia.edu

© 2008 The Research Foundation for Mental Hygiene, Inc.

| SUICIDAL IDEATION | | | WEST TO |
|---|---|---|---|
| | Suicidal Behavior" section. If the answer to question 2 is "yes",<br>for 2 is "yes", complete "Intensity of Ideation" section below. | | e Last<br>isit |
| 1. Wish to be Dead Subject endorses thoughts about a wish to be dead or not alive anymore Have you wished you were dead or wished you could go to sleep and n | | Yes | No |
| If yes, describe: | | | |
| 2. Non-Specific Active Suicidal Thoughts General, non-specific thoughts of wanting to end one's life/commit suic oneself/associated methods, intent, or plan during the assessment period Have you actually had any thoughts of killing yourself? | cide (e.g., "I've thought about killing myself") without thoughts of ways to kill i. | Yes | No |
| If yes, describe: | | | |
| | thod during the assessment period. This is different than a specific plan with time, but not a specific plan). Includes person who would say, "I thought about taking an | Yes | No |
| If yes, describe: | | | |
| 4. Active Suicidal Ideation with Some Intent to Act, with Active suicidal thoughts of killing oneself and subject reports having so definitely will not do anything about them." Have you had these thoughts and had some Intention of acting on the | eme intent to act on such thoughts, as opposed to "I have the thoughts but I | Yes | No |
| If yes, describe: | | | |
| <ol> <li>Active Suicidal Ideation with Specific Plan and Intent<br/>Thoughts of killing oneself with details of plan fully or partially worked<br/>Have you started to work out or worked out the details of how to kill yo</li> </ol> | I out and subject has some intent to carry it out. | Yes | No |
| If yes, describe: | | | |
| INTENSITY OF IDEATION | | | |
| The following features should be rated with respect to the most and 5 being the most severe). | severe type of ideation (i.e., 1-5 from above, with 1 being the least severe | | ost |
| Most Severe Ideation: | D. J. C. of H. C. | Sey | vere |
| Type # (1-5) | Description of Ideation | - | |
| How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in we | cek (4) Daily or almost daily (5) Many times each day | _ | _ |
| Duration When you have the thoughts, how long do they last? | | 10 | |
| (1) Fleeting - few seconds or minutes (2) Less than 1 hour/some of the time (3) 1-4 hours/a lot of time | (4) 4-8 hours/most of day (5) More than 8 hours/persistent or continuous | _ | _ |
| Controllability Could/can you stop thinking about killing yourself or want (1) Easily able to control thoughts (2) Can control thoughts with little difficulty (3) Can control thoughts with some difficulty | ing to die if you want to? (4) Can control thoughts with a lot of difficulty (5) Unable to control thoughts (0) Does not attempt to control thoughts | _ | _ |
| Deterrents Are there things - anyone or anything (e.g., family, religion thoughts of committing suicide? (1) Deterrents definitely stopped you from attempting suicide (2) Deterrents probably stopped you (3) Uncertain that deterrents stopped you | (4) Deterrents most likely did not stop you (5) Deterrents definitely did not stop you (0) Does not apply | _ | |
| Reasons for Ideation What sort of reasons did you have for thinking about wanti | ing to die or killing yourself? Was it to end the pain or stop the way with this pain or how you were feeling) or was it to get attention, (4) Mostly to end or stop the pain (you couldn't go on living with the pain or how you were feeling) (5) Completely to end or stop the pain (you couldn't go on living with the pain or how you were feeling) | | |

© 2008 Research Foundation for Mental Hygiene, Inc.

C-SSRS—Since Last Visit (Version 1/14/09)

Page 1 of 2

| Actual Attempt: Appendixly sold injurious act committed with at least some with 10 die, ar a result of act. Behavior was in part thought of an method to kill oncored. Intent does not have to be 100%. If there is any intentification to die associated with the act, thus it can be considered an actual studied attempt. There does not have to be 100%. If there is any intentification to die, it may be inferred clinically from the behavior or circumstance. For example, a highly letter of the control of | SUICIDAL BEHAVIOR | Since | e Last |
|---|---|---|---|
| A potentially self-injentious act committed with a closus areas when the disk, are resulted placed. Behavior was in part thought of an embod to kill owned: Intenditure of the contribution to the construction of the contribution of the contribution of the part player or harm. Intenditure of the player or harm. It presents the player or harm. It presents that the contribution are committed to the contribution of the contribu | (Check all that apply, so long as these are separate events; must ask about all types) | V | isit |
| Intent at that is clearly not an accident so no other intent but saictic can be interrued (e.g., granted to bead, jumping from window of a high floor/fiery). Alon, if smoone demie inserts to die, but when they did could be lethal, intent may be inferred. Have you done anything to that may courself? Have you done anything dangerous where you could have died? What did you | A potentially self-injurious act committed with at least some wish to die, as a result of act. Behavior was in part thought of as method to kill oneself. Intent does not have to be 100%. If there is any intent/desire to die associated with the act, then it can be considered an actual suicide attempt. There does not have to be any injury or harm, just the potential for injury or harm. If person pulls trigger while gun is in mouth but gun is broken so no injury results, | 100 800 | |
| Have you done anything dangerous where you could have died? What did you do? Did you are a lattle; when you? Were you trying to end your life when you? Were you trying to end your life when you? Or did you do it purely for other reasons' without ANY Instention of killing yourself (like to relieve stress, feel better, get sympathy, or get something else to happen)? (Self-injurious Behavior without suicidal intent) If ye, describe Yes No Has subject engaged in Non-Suicidal Self-Injurious Behavior? Interrupted Attempt: When the prose is interrupted (by an outside circumstance) from starting the potentially self-injuriou act (if not for that, actual attempt would have Overdose. Person has pills in hand be is stopped from ingesting. Once they night to the sent and the trying of the trying | lethal act that is clearly not an accident so no other intent but suicide can be inferred (e.g., gunshot to head, jumping from window of a high floor/story). Also, if someone denies intent to die, but they thought that what they did could be lethal, intent may be inferred. Have you made a suicide attempt? | B | |
| What did you do? Did you want to die (even a little) when you? Were you trying to end your life when you? Or did you think it was possible you could have died from? Or did you think it was possible you could have died from? Or did you do think it was possible you could have died from? Or did you do think it was possible you could have died from? Or did you do think it was possible you could have died from? Or did you do think it was possible you could have died from? Or did you do the purely for other reasons /without AIV intention of killing yourself dike to relieve stress, feel better, get ymputly, or get something else to happen? (Self-injurious Behavior? Interrupted Attempt: When the person is interrupted (by an outside circumstance) from starting the potentially self-injurious axt (if not for the a national divided of the person is interrupted (by an outside circumstance) from starting the potentially self-injurious axt (if not for the a national divided of the person is interrupted (by an outside circumstance) from starting the potentially self-injurious axt (if not for the a national divided of the person is interrupted (by an outside circumstance) from starting the potentially self-injurious axt (if not for the a national divided of the person is interrupted (by an outside circumstance) from starting the person is interrupted (by an outside of the person is interrupted (by an outside of the person is interrupted (by an outside of the person is interrupted (by an outside statemy) and the person is not an outside person is the start of the person is not a start of the person is not a start of the person is the start of the person is not a | | Tota | l#of |
| Did you want to die (even a little) when you? Were you trying to end your life when you? Or did you do it purely for other reasons' without ANY Intention of killing yourself (like to relieve stress, feel better, get sympathy, or get something else to happen)? (Self-injurious Behavior without suicidal intent) If yes, describe Yes No Has subject engaged in Non-Suicidal Self-Injurious Behavior? Interrupted Attempt: When the penes is interrupted (by an outside circumstance) from starting the potentially self-injurious act (if not for that, actual attempt would have When the penes is interrupted (by an outside circumstance) from starting the potentially self-injurious act (if not for that, actual attempt would have Overdone-Penon has pills in hand but is stopped from lingesting. Once they night self-injurious act (if not for that, actual attempt would have Overdone-Penon has pills in hand but is stopped from lingesting. Once they night to tigger, were if the gan fails to fire, it is an attempt. Jumping-Person is poised to jump, is grabbed and taken down from ledge. Hanging-Person has noose around note but has not yet stated to hange, is larged. Once they night to tigger. Has there been a time when you started to do something to end your life but someone or something stopped you before you actually did around the interrupted attempt, except that the individual stops him/farent(i, instead of being stopped by something else. Has there been a time when you started to do something to try to end your life but you stopped yourself before you actually did anything? If yes, describe. Preparatory Acts or Behavior: Acts or preparation towards imminently making a suicide attempt, except that the individual stops themselves before they actually have engaged in any self-destructive behavior. But you taken my steps towards making a suicide attempt, or you actually did anything? If yes, describe. Preparatory Acts or Behavior: Suicidal Behavior: Suicidal Behavior: Actual Lethality/Medical Damage: No hybrid dian | | | |
| Did you want to die (even a little) when you ? Were you tring to end you could have died from ? Or did you think it was possible you could have died from ? Or did you think it was possible you could have died from ? Or did you to the purefy for other reasons / without ANY intention of killing yourself (like to relieve stress, feel better, get sympathy, or get something else to happen)? (Scif-injurious Behavior? Interrupted Attempt: When the person is interrupted (by an outside circumstance) from starting the potentially self-injurious act (if not for that, actual attempt would have cocurred). One courred. One courred. One was a strengt table than he gis in hand but is stopped from ingesting. Once they ingest any pills, this becomes an attempt rather than an interrupted attempt. Shooting-Person has gun pointed toward self, pus is takes away by someone else, or is comelow prevented from puling trigger. Once they pull the trigger entire than the pull to trigger. I strength of the pull than not yet started to hang. is stopped from doing so. Has there been at time when you started to do something to end your life but someone or something stopped you before you actually did anything? If yet, describe. Aborted Attempt: When the person is in the trigger toward making a suicide attempt, but stops themselves before they actually have engaged in any self-destructive behavior. Preparatory Acts or Buhavior: Acts or preparation towards handleng as suicide attempt, but stops themselves before they actually have engaged in any self-destructive behavior. Acts or preparation towards handleng as suicide attempt, but stops themselves before they actually have engaged in any self-destructive behavior. Acts or preparation towards handleng as suicide attempt, but stops themselves before they actually have engaged in any self-destructive behavior. Acts or preparation cowards handleng as suicide attempt, this can include anything beyond a weblication or though, such as assembling a destructive propersion of the self-destructive | | | |
| Or did you do thank it was possible you could have died from | | | |
| Or did you do it purely for other reasons / without ANY intention of killing yourself (like to relieve stress, feel better, get sympathy, or get something else to huppen)? (Self-Injurious Behavior without suicidal intent) If yes, describe: Yes No Interrupted Attempt: When the person is interrupted (by an outside circumstance) from starting the potentially self-injurious act (if not for inat, actual attempt would have occurred). Overdonce Person has pills in hand but is stopped from ingesting. Once they ingest any pills, this becomes an attempt rather than an interrupted attempt. Shooting: Person has pills in hand but is stopped from onling so, bed to jump, is grabed and taken to down from liegh intaging. From his moore round neck but has not ye started to have a stopped from doing so, bed to jump, is grabed and taken town from liegh intaging. From his moore round reactually did anything? If yes, describe. Has there been a time when you started to do something to end your life but someone or something stopped you before you actually did anything? If yes, describe. Aborted Attempt: When person begins to take steps toward making a suicide attempt, but stops themselves before they actually have engaged in any self-destructive behavior. Esamples are similar to interrupted attempts, except that the individual stops him/nersoft, instead of being stopped by something gets actually did anything? If yes, describe Preparatory Acts or Behavior: Acts or preparation towards imminently making a suicide attempt or preparing to kill yourself (such as collecting pills, getting a gun, pill getting a gun, getting and gun, | Were you trying to end your life when you? | | |
| If yes, describe. Yes No Has subject engaged in Non-Suicidal Self-Injurious Behavior? Interrupted Attempt: When the person is interrupted dry an outside circumstance) from starting the potentially self-injurious act (if not for ital, actual attempt would have occurred). Overdose: Person has pills in hand but is stopped from ingesting. Once they ingest any pills, this becomes an attempt rather than an interrupted attempts. Overdose: Person has pills in hand but is stopped from ingesting. Once they ingest any pills, this becomes an attempt rather than an interrupted attempt, cover if the gan fails to fire, it is an attempt. Jumping: Person is poised to jump, is grabbed and taken down from ledge. Hanging: Person has none around that she have not a dine when you started to do something to end your life but someone or something stopped you before you actually did anything? If you, describe: When person begins to take steps toward making a suicide attempt, but stops themselves before they actually have engaged in any self-destructive behavior. Aborted Attempt: When person begins to take steps toward making a suicide attempt, but stops him/herself, instead of being stopped by something else. Has there been a time when you started to do something to try to end your life but you stopped yourself before you actually did anything? If yes, describe: Preparatory Acts or Behavior: Area or preparation bounds inminently making a suicide attempt or preparing for one's death by suicide (e.g., giving things away, writing a suicide note)? If yes, describe: Preparatory Acts or Behavior: Alway ou taken any steps towards making a suicide attempt or preparing to kill yourself (such as collecting pills, getting a gun, giving valuables away or writing a suicide note)? If yes, describe: Answer for Actual Attempts Only Actual Lethality/Medical Damage: No physical damage or yellow preparation and likely intensive care required (e.g., comainse with reflexes; third-degree burns over 20% of body; extensive blood loss with | | | |
| Laterrupted Attempt: When the person is interrupted (by an outside circumstance) from starting the potentially self-injurious act (if not for ibat, actual attempt would have concurred). Overdose: Person has pills in hand but is stopped from ingesting. Once they ingest any pills, this becomes an attempt rather than an interrupted attempt. Overdose: Person has pills in hand but is stopped from ingesting. Once they ingest any pills, this becomes an attempt rather than an interrupted attempt, even if the gam fails to fire, it is an attempt. Jumping: Person is pointed to jump, is grabbed and daten down from ledge. Hanging: Person has noose around neck but has not yet started to has; is stopped from oling so. **Has there been a time when you started to do something to end your life but someone or something stopped you before you actually did anything?** If yes, doscribe: **Aborted Attempt:** **When person begins to take steps toward making a suicide attempt, but stops themselves before they actually have engaged in any self-destructive behavior. **Businjeas are similar to interrupted attempts, except that the individual stops him/hersoft, instead of being stopped by something eige. **Preparatory Acts or Behavior:** **Are so repravation towards imminently making a suicide attempt, but any of end your life but you stopped yourself before you actually did anything?* If yes, describe: **Preparatory Acts or Behavior:** **Are you taken any steps towards making a suicide attempt or preparing to one's death by suicide (e.g., giving things away, writing a suicide not)? **If you disches away or writing a suicide attempt or preparing to one's death by suicide (e.g., giving things away, writing a suicide not)? **If yes, describe:** **Suicidal Behavior:** **Suicidal Behavior:** **Suicidal Behavior:** **Suicidal Behavior:** **Actual Lethality/Medical Damage:** **O Popisial damage or very minor physical damage (e.g., surface semethes). **O Popisial damage or very minor physical damage (e.g., onesions but st | sympathy, or get something else to happen)? (Self-Injurious Behavior without suicidal intent) | | |
| Has subject engaged in Non-Suicidal Self-Injurious Behavior? Interrupted Attempt: When the person is interrupted (by an outside circumstance) from starting the potentially self-injurious act (if not for that, actual attempt would have occurred). Overdoose: Person has gills in hand but is stepped from ingesting. Once they ingest any pills, this becomes an attempt rather than an interrupted attempt. Shooting: Person has gill so in hand but is stepped from ingesting. Once they ingest any pills, this becomes an attempt rather than an interrupted attempt. Shooting: Person has gill so in hand but is stepped from ingesting. Once they ingest any pills, this becomes an attempt rather than an interrupted attempt. Shooting: Person has gill so in the step in th | n yes, destrice. | V. | No |
| This study let diagraph of Non-Suttengtic When the person is interrupted (by an outside circumstance) from starting the potentially self-injurious act (if not for that, actual attemps would have occurred). When the person is interrupted (by an outside circumstance) from starting the potentially self-injurious act (if not for that, actual attemps would have occurred). Sociolog: Person has plin in hand but is stopped from injusting. Once they injust the trigger, concerned, but has post yet started to hang, is stopped from doing, so. Has there been at time when you started to do something to end your life but someone or something stopped you before you actually did anything? If yes, describe: **No Aborted Attempt:** When person begins to take steps toward making a suicide attempt, but stops themselves before they actually have engaged in any self-destructive behavior. **Has there been at time when you started to do something to try to end your life but you stopped yourself before you actually did anything? If yes, describe: **Preparatory Acts or Behavior:** Acts or preparation towards imminently making a suicide attempt, this can include anything beyond a verbalization or thought, such as assembling a specific method (e.g., buying pills, purchasing a pun) or preparing for one's death by suicide (e.g., giving things away, writing a suicide note)? If yes, describe: **Preparatory Acts or Behavior:** Suicidal Behavior:** Answer for Actual Attempts Only Actual Lethality/Medical Damage: No physical damage or very minor physical damage (e.g., surface scratches). More physical damage, medical hospitalization and likely intensive care required (e.g., comatose with reflexes intact, third-degree bums less than 20% of body; extensive blood loss but unclassed vial sign; major damage to a vial area). Society of body of the proper should be repaired to more). | | 14000 | |
| When the person is interrupted (by an outside circumstance) from starting the potentially self-injurious at (if nex for hint, actual attempt with here occurred). Overdose: Person has pills in hand but is stopped from ingesting. Once they pills, this becomes an attempt rather than an inventible attempt, shouling Person has pills in hand but is stopped from doing so. Has there been a time when you started to do something to end your life but someone or something stopped you before you actually did anything? If yes, describe: Aborted Attempt: When person begins to take steps toward making a suicide attempt, but stops themselves before they actually did anything? If yes, describe: Preparatory Acts or Behavior: Acts or preparation towards imminently making a suicide attempt, the special possible of the preparation towards imminently making a suicide attempt, or preparing for one's death by suicide (e.g., buying things away, writing a suicide note)? If yes, describe: Preparation towards imminently making a suicide attempt or preparing to kill yourself (such as collecting pills, getting a gun, giving valuables away or writing a suicide note)? If yes, describe: Salicidal Behavior: Suicidal Ebavior: Suicidal Ebavior: Suicidal Cattal Attempts Only Actual Lethality/Medical Damage: No physical damage or very minor physical damage (e.g., surface scratches). No physical damage or very minor physical damage, (e.g., surface scratches). No physical damage red on the or physical damage, medical hospitalization and likely intensive care required (e.g., comatose with reflexes intact, third-degree burns less than 20% of body; extensive blood loss but necessary and family and family of making a vivil a reductive of the physical damage, medical hospitalization with intensive care required (e.g., comatose with reflexes intact, third-degree burns beet for no reducted damage, medical hospitalization with intensive care required (e.g., comatose without reflexes; third-degree burns over 20% of body; Severe physical dam | Has subject engaged in Non-Suicidal Self-Injurious Behavior? | | |
| Overdose: Person has pills in hand but is stopped from ingesting. Once they ingest any pills, this becomes an attempt rather than an interrupted attempt, shooting. Person has guan pointed toward self, guin is taken away by someone else, or is somehow prevented from pulling trigger. Once they pull the trigger, even if the gun fails to fire, it is an attempt. Jumping: Person is poised to jump, is grabbed and taken down from ledge. Hanging. Person has noose around nock but has not yet starde to hang, is stopped from doing so. **Has there been a time when you started to do something to end your life but someone or something stopped you before you actually did anything? If yes, describe: **New person begins to take steps toward making a suicide attempt, but stops themselves before they actually have engaged in any self-destructive behavior. **Examples are similar to interrupted attempts, except that the individual stops him/herself, instead of being stopped yourself before you actually did anything? If yes, describe: **Preparatory Acts or Behavior:** **Preparatory Acts or Behavior:** **Acts or preparation towards imminently making a suicide attempt for preparing to kill yourself (such as collecting pills, getting a gun, giving valuables away or writing a suicide attempt or preparing to kill yourself (such as collecting pills, getting a gun, giving valuables away or writing a suicide attempt or preparing for one's death by suicide (e.g., giving things away, writing a suicide note)? **Suicidal Behavior:** **Suicidal Behavior:** **Suicidal Behavior was present during the assessment period?** **Actual Lethality/Medical Damage:** **Actual Lethality/Medical Damage:** **Actual Lethality/Medical Damage:** **Actual Lethality/Medical Damage:** **Actual Lethality-index damage, reside hospitalization and likely intensive care required (e.g., comatose with reflexes intact; third-degree bums less than 20% of body, extensive blood loss but miscry to blood loss with unstable valua larges, mayind damage or very minor | | Yes | No |
| Shooting. Person has gun pointed toward self, gun is taken away by someone else, or is somehow prevented from putiling trigger. Once they put the trigger, even if the gun fails to fire, it is an attempt. Jumping: Person is posited to jump, is grabbed and taken down from ledge. Hanging Person has noos around neck but has not yet started to hang is stopped from doing so. Has there been a time when you started to do something to end your life but someone or something stopped you before you actually did anything? If yes, describe: Meen person begins to take steps toward making a suicide attempt, but stops themselves before they actually have engaged in any self-destructive behavior. Examples are similar to interrupted attempts, except that the individual stops him/tenself, instead of being stopped yourself before you actually did anything? If yes, describe. Has there been a time when you started to do something to try to end your life but you stopped yourself before you actually did anything? If yes, describe. Preparatory Acts or Behavior: Acts or preparation towards imminently making a suicide attempt. This can include anything beyond a verbalization or thought, such as assembling a properific method (e.g., buying pills, purchasing a gun) or preparing for one's death by suicide (e.g., giving things away, writing a suicide note). Have you taken any steps towards making a suicide attempt or preparing to kill yourself (such as collecting pills, getting a gun, giving valuables away or writing a suicide antempt on preparing to kill yourself (such as collecting pills, getting a gun, giving valuables away or writing as suicide antempt on preparing to kill yourself (such as collecting pills, getting a gun, giving valuables away or writing as suicide attempt or preparing to kill yourself (such as collecting pills, getting a gun, giving dunings away, writing a suicide note). Suicide: Answer for Actual Lethality/Medical Damage: No physical damage, medical attention needle (e.g., comotions with networks intact, thi | | | |
| Total # of interrupted attempts Total # of interrupted attempt Total # of interrupted Total # of interrupted attempts, except that the individual stops him/herself, instead of being stopped by something else. Total # of aborted To | Shooting: Person has gun pointed toward self, gun is taken away by someone else, or is somehow prevented from pulling trigger. Once they pull the trigger, even if the gun fails to fire, it is an attempt. Jumping: Person is poised to jump, is grabbed and taken down from ledge. Hanging: Person has noose around | | |
| If yes, describe: When person begins to take steps toward making a suicide attempt, but stops themselves before they actually have engaged in any self-destructive behavior. Examples are similar to interrupted attempts, except that the individual stops him/herself, instead of being stopped by something else. Has there been a time when pour started to do something to try to end your life but you stopped yourself before you actually did anything? If yes, describe: Preparatory Acts or Behavior: Acts or preparation towards imminently making a suicide attempt, This can include anything beyond a verbalization or thought, such as assembling a specific method (e.g., toying pills, purchasing a gun) or preparing for one's death by suicide (e.g., giving things away, writing a suicide note). Have you taken any steps towards making a suicide attempt or preparing to kill yourself (such as collecting pills, getting a gun, giving valuables away or writing a suicide note)? If yes, describe: Suicidal Behavior: Suicidal Behavior: Suicidal Behavior Suicidal subary or very minor physical damage (e.g., surface scratches). Answer for Actual Attempts Only Answer for Actual Attempts Only Actual Lethality/Medical Damage: On physical damage (e.g., lathagic speech, first-degree burns, mild bleeding, sprains). In Minor physical damage, medical attention needed (e.g., conscious but sleepy, somewhat responsive, second-degree burns, bleeding of major vessel). Moderately severe physical damage, medical attention needed (e.g., conscious but sleepy, somewhat responsive, second-degree burns over 20% of body; extensive blood loss with unstable vital signs, major fractures) Severe physical damage, medical absopilization and likely intensive care required (e.g., comatose without reflexes; third-degree burns over 20% of body; extensive blood loss with unstable vital signs, major fandange (e.g., conscious but sleepy, somewhat responsive, second-degree burns over 20% of body; extensive blood loss with unstable vital signs, major damag | | | |
| When person begins to take steps toward making a suicide attempt, but stops themselves before they actually have engaged in any self-destructive behavior. Examples are similar to interrupted attempts, except that the individual stops him/threstle, instead of being stopped by something else. Has there been a time when you started to do something to try to end your life but you stopped yourself before you actually did anything? If yes, describe: Preparatory Acts or Behavior: Acts or preparation towards imminently making a suicide attempt. This can include anything beyond a verbalization or thought, such as assembling a specific method (e.g., buying pills, purchasing a gun) or preparing for one's death by suicide (e.g., giving things away, writing a suicide note) If yes, describe: Suicidal Behavior: Suicidal Behavior: Suicidal Behavior: Suicidal Behavior: Suicidal Behavior was present during the assessment period? Answer for Actual Attempts Only Actual Lethality/Medical Damage: On ophysical damage or very minor physical damage (e.g., lethargis speech, first-degree burns, mild bleeding; sprains). Actual Lethality/Medical Damage: On ophysical damage or very minor physical damage, medical attention needed (e.g., conscious but steppy, somewhat responsive, second-degree burns, bleeding of major vessel). Moderately severe physical damage, medical hospitalization and likely intensive care required (e.g., comatose without reflexes; third-degree burns over 20% of body; extensive blood loss but can recover, major fractures) Death: Potential Lethality: Only Answer if Actual Lethality=0 Likely lethality of actual attempt if no medical damage (the following examples, while having no actual medical damage, had potential for very serious lethality; put gun in moth and pulled the trigger but gun fails to fire so no medical damage, laying on train tracks with oncoming train but pulled away before run over). Enter Code Enter C | actually did anything? | inten | rupted |
| Examples are similar to interrupted attempts, except that the individual stops him/herself, instead of being stopped by something else. Has there been a time when you started to do something to try to end your life but you stopped yourself before you actually did anything? If yes, describe: Preparatory Acts or Behavior: Acts or preparation towards imminently making a suicide attempt. This can include anything beyond a verbalization or thought, such as assembling a specific method (e.g., buying pills, purchasing a gun) or preparing for one's death by suicide (e.g., giving things away, writing a suicide note). Have you taken any steps towards making a suicide attempt or preparing to kill yourself (such as collecting pills, getting a gun, giving valuables away or writing a suicide note)? If yes, describe: Suicidal Behavior: Suicidal Behavior: Suicidal Behavior was present during the assessment period? Answer for Actual Attempts Only Answer for Actual Attempts Only Actual Lethality/Medical Damage: 0. No physical damage or very minor physical damage (e.g., surface scratches). 1. Minor physical damage, medical attention needed (e.g., conscious but sleepy, somewhat responsive, second-degree burns; bleeding of major vessel). 3. Moderately severe physical damage, medical hospitalization and likely intensive care required (e.g., comatose with out reflexes; third-degree burns over 20% of body; exertisely blood loss but can recover, major fractures). 4. Severe physical damage, medical hospitalization with intensive care required (e.g., comatose without reflexes; third-degree burns over 20% of body; exertisely blood loss with unstable vital signs; major damage to a vital area). 5. Death Potential Lethality: Only Answer if Actual Lethality=0 Likely lethality of actual attempt; if no medical damage (the following examples, while having no actual medical damage, had potential for very serious lethality; put gun in mouth and pulled the trigger but gun fails to fire so no medical damage, laying on train tracks | | Yes | No |
| Total of of aborted | | | |
| If yes, describe: Preparatory Acts or Behavior: Acts or preparation towards imminently making a suicide attempt. This can include anything beyond a verbalization or thought, such as assembling a specific method (e.g., buying pills, purchasing a gun) or preparing for one's death by suicide (e.g., giving things away, writing a suicide note). | Has there been a time when you started to do something to try to end your life but you stopped yourself before you | | |
| Preparatory Acts or Behavior: Acts or preparation towards imminently making a suicide attempt. This can include anything beyond a verbalization or thought, such as assembling a specific method (e.g., buying pills, purchasing a gun) or preparing for one's death by suicide (e.g., giving things away, writing a suicide note). Have you taken any steps towards making a suicide attempt or preparing to kill yourself (such as collecting pills, getting a gun, giving valuables away or writing a suicide note)? If yes, describe: Suicidal Behavior: Suicidal Behavior Suicidal Behavior was present during the assessment period? Yes No Answer for Actual Attempts Only Answer for Actual Attempts Only Actual Lethality/Medical Damage: 0. No physical damage or very minor physical damage (e.g., surface scratches). 1. Minor physical damage (e.g., lethargic speech, first-degree burns; mild bleeding; sprains). 2. Moderate physical damage, medical attention needed (e.g., conscious but sleeppy, somewhat responsive; second-degree burns; bleeding of major vessel). 3. Moderately severe physical damage, medical hospitalization and likely intensive care required (e.g., comatose with reflexes intact, third-degree burns less than 20% of body; extensive blood loss with unstable vital signs; major damage to a vital area). 5. Death Potential Lethality: Only Answer if Actual Lethality=0 Likely lethality of actual attempt if no medical damage (the following examples, while having no actual medical damage, had potential for very serious lethality; put gun in mouth and pulled the trigger but gun fails to fire so no medical damage, laying on train tracks with oncoming train but pulled away before run over). Behavior likely to result in injury but not likely to cause death 2 - Behavior likely to result in injury but not likely to cause death 2 - Behavior likely to result in injury but not likely to cause death 2 - Behavior likely to result in death despite available medical care | | | |
| Action preparation towards imminently making a suicide attempt. This can include anything beyond a verbalization or thought, such as assembling a period preparing for one's death by suicide (e.g., giving things away, writing a suicide note). Have you taken any steps towards making a suicide note)? If yes, describe: Suicidal Behavior: Suicidal Behavior was present during the assessment period? Suicidal Behavior was present during the assessment period? Suicidal Behavior was present during the assessment period? Answer for Actual Attempts Only Answer for Actual Attempts Only Answer for Actual Attempts Only Most Lethal Attempt Date: Actual Lethality/Medical Damage: 0. No physical damage or very minor physical damage (e.g., tethagic speech, first-degree burns; mild bleeding; sprains). 2. Moderate physical damage; medical attention needed (e.g., conscious but sleepy, somewhat responsive; second-degree burns; bleeding of major vessel). 3. Moderate physical damage; medical attention needed (e.g., conscious but sleepy, somewhat responsive; second-degree burns; bleeding of major vessel). 4. Severe physical damage; medical attention needed (e.g., conscious but sleepy, somewhat responsive; second-degree burns; bleeding of major vessel). 5. Death Potential Lethality: Only Answer if Actual Lethality=0 Likely lethality: Only Answer if Actual Lethality=0 Likely lethality: Only Answer if Actual Lethality=0 Likely lethality or essult in injury 1 = Behavior likely to result in injury 2 = Behavior likely to result in injury but not likely to cause death 2 = Behavior likely to result in indeath despite available medical care | If yes, describe: | abo | nteu |
| specific method (e.g., buying pills, purchasing a gun) or preparing for one's death by suicide (e.g., giving things away, writing a suicide note). Have you taken any steps towards making a suicide attempt or preparing to kill yourself (such as collecting pills, getting a gun, giving valuables away or writing a suicide note)? If yes, describe: Suicidal Behavior: Suicidal Behavior was present during the assessment period? Yes No Guicidal Behavior was present during the assessment period? Answer for Actual Attempts Only Most Lethal Attempts Actual Lethality/Medical Damage: 0. No physical damage or very minor physical damage (e.g., surface scratches). 1. Minor physical damage (e.g., telhargic speech, first-degree burns; mild bleeding; sprains). 2. Moderate physical damage, medical attention needed (e.g., conscious but sleepy, somewhat responsive; second-degree burns; bleeding of major vessel). 3. Moderately severe physical damage, medical hospitalization and likely intensive care required (e.g., comatose with reflexes intact, third-degree burns less than 20% of body; extensive blood loss but can recover, major fractures). 4. Severe physical damage, medical hospitalization with intensive care required (e.g., comatose without reflexes; third-degree burns over 20% of body; extensive blood loss with unstable vital signs; major damage to a vital area). 5. Death Potential Lethality: Only Answer if Actual Lethality=0 Likely lethality of actual attempt if no medical damage (the following examples, while having no actual medical damage, had potential for very serious lethality; put gun in mouth and pulled the trigger but gun fails to fire so no medical damage, laying on train tracks with oncoming train but pulled away before run over). Behavior likely to result in injury 1 = Behavior likely to result in injury but not likely to cause death 2 2 = Behavior not likely to result in death despite available medical care | | - | _ |
| Have you taken any steps towards making a suicide attempt or preparing to kill yourself (such as collecting pills, getting a gun, giving valuables away or writing a suicide note)? If yes, describe: Suicidal Behavior: Suicidal Behavior was present during the assessment period? Suicide: Yes No Answer for Actual Attempts Only Most Lethal Attempt Date: Actual Lethality/Medical Damage: 0. No physical damage or very minor physical damage (e.g., surface scratches). 1. Minor physical damage or very minor physical damage (e.g., surface scratches). 3. Moderately severe physical damage; medical attention needed (e.g., conscious but sleepy, somewhat responsive, second-degree burns; bleeding of major vessel). 3. Moderately severe physical damage; medical hospitalization and likely intensive care required (e.g., comatose with reflexes intact; third-degree burns less than 20% of body; extensive blood loss but can recover; major fractures). 4. Severe physical damage; medical hospitalization with intensive care required (e.g., comatose without reflexes; third-degree burns over 20% of body; extensive blood loss but can recover; major fractures). 5. Death Potential Lethality: Only Answer if Actual Lethality=0 Likely lethality of actual attempt if no medical damage (the following examples, while having no actual medical damage, had potential for very serious tethality; put gun in mouth and pulled the trigger but gun fails to fire so no medical damage; laying on train tracks with oncoming train but pulled away before run over). Behavior not likely to result in injury but not likely to cause death 2 Behavior likely to result in injury but not likely to cause death 2 Behavior likely to result in injury but not likely to cause death 2 Behavior likely to result in injury but not likely to cause death | | Yes | No |
| Suicidal Behavior: Suicidal Behavior was present during the assessment period? Yes No Suicidal Behavior was present during the assessment period? Yes No Suicidal Behavior was present during the assessment period? Period | | | |
| Suicidal Behavior: Suicidal Behavior: Suicidal Behavior was present during the assessment period? Suicide: Answer for Actual Attempts Only Most Lethal Attempt Date: Actual Lethality/Medical Damage: 0. No physical damage or very minor physical damage (e.g., surface scratches). 1. Minor physical damage (e.g., letharige speech, first-degree burns; mild bleeding; sprains). 2. Moderately severe physical damage, medical attention needed (e.g., conscious but sleepy, somewhat responsive; second-degree burns; bleeding of major vessel). 3. Moderately severe physical damage, medical hospitalization and likely intensive care required (e.g., comatose with reflexes intact; third-degree burns less than 20% of body; extensive blood loss but can recover, major fractures). 4. Severe physical damage; medical hospitalization with intensive care required (e.g., comatose without reflexes; third-degree burns over 20% of body; extensive blood loss with unstable vital signs; major damage to a vital area). 5. Death Potential Lethality: Only Answer if Actual Lethality=0 Likely lethality of actual attempt if no medical damage (the following examples, while having no actual medical damage, had potential for very serious tethality; put gun in mouth and pulled the trigger but gun fails to fire so no medical damage, laying on train tracks with oncoming train but pulled away before run over). De Behavior not likely to result in injury but not likely to cause death 2 Behavior likely to result in indeath despite available medical care | | 87948 | |
| Suicide: Suicide: No plants | | | |
| Suicide: Answer for Actual Attempts Only Actual Lethality/Medical Damage: Only Actual Lethality/Medical Megica expressions with oncoming than but publied away before run over). Only Actual Lethality/Medical Megica expressions with intensive | | Yes | No |
| Answer for Actual Attempts Only Actual Lethality/Medical Damage: Only No physical damage or very minor physical damage (e.g., surface scratches). Moderate physical damage (e.g., lethargic speech; first-degree burns; mild bleeding; sprains). Moderate physical damage; medical hospitalization and likely intensive care required (e.g., comatose with reflexes intact; third-degree burns less than 20% of body; extensive blood loss but can recover; major fractures). Severe physical damage; medical hospitalization with intensive care required (e.g., comatose without reflexes; third-degree burns over 20% of body; extensive blood loss with unstable vital signs; major damage to a vital area). Death Potential Lethality: Only Answer if Actual Lethality=0 Likely lethality of actual attempt if no medical damage (the following examples, while having no actual medical damage, had potential for very serious lethality: put gun in mouth and pulled the trigger but gun fails to fire so no medical damage; laying on train tracks with oncoming train but pulled away before run over). De Behavior not likely to result in injury 1 = Behavior not likely to result in injury but not likely to cause death 2 = Behavior likely to result in death despite available medical care | Suicidal denaylor was present during the assessment period? | | |
| Actual Lethality/Medical Damage: O. No physical damage or very minor physical damage (e.g., surface scratches). I. Minor physical damage (e.g., lethargic speech, first-degree burns; mild bleeding; sprains). O. Moderatel physical damage; medical tention needed (e.g., conscious but sleepy, somewhat responsive; second-degree burns; bleeding of major vessel). Moderately severe physical damage; medical hospitalization and likely intensive care required (e.g., comatose with reflexes intact; third-degree burns less than 20% of body; extensive blood loss but can recover; major fractures). Severe physical damage; medical hospitalization with intensive care required (e.g., comatose without reflexes; third-degree burns over 20% of body; extensive blood loss with unstable vital signs; major damage to a vital area). Death Potential Lethality: Only Answer if Actual Lethality=0 Likely lethality of actual attempt if no medical damage (the following examples, while having no actual medical damage, had potential for very serious lethality: put gun in mouth and pulled the trigger but gun fails to fire so no medical damage; laying on train tracks with oncoming train but pulled away before run over). De Behavior not likely to result in injury 1 = Behavior likely to result in injury 1 = Behavior likely to result in death despite available medical care | Suicide: | Yes | No |
| Attempt Date: Actual Lethality/Medical Damage: 0. No physical damage or very minor physical damage (e.g., surface scratches). 1. Minor physical damage (e.g., lethargic speech; first-degree burns; mild bleeding; sprains). 2. Moderate physical damage; medical attention needed (e.g., conscious but sleepy, somewhat responsive; second-degree burns; bleeding of major vessel). 3. Moderately severe physical damage; medical hospitalization and likely intensive care required (e.g., comatose with reflexes intact; third-degree burns less than 20% of body; extensive blood loss but can recover; major fractures). 4. Severe physical damage; medical hospitalization with intensive care required (e.g., comatose without reflexes; third-degree burns over 20% of body; extensive blood loss with unstable vital signs; major damage to a vital area). 5. Death Potential Lethality: Only Answer if Actual Lethality=0 Likely lethality; of actual attempt if no medical damage (the following examples, while having no actual medical damage, had potential for very serious lethality: put gun in mouth and pulled the trigger but gun fails to fire so no medical damage; laying on train tracks with oncoming train but pulled away before run over). 0 = Behavior not likely to result in injury 1 = Behavior likely to result in indeath despite available medical care | | | |
| Actual Lethality/Medical Damage: 0. No physical damage or very minor physical damage (e.g., surface scratches). 1. Minor physical damage (e.g., lethargic speech; first-degree burns; mild bleeding; sprains). 2. Moderate physical damage; medical attention needed (e.g., conscious but sleepy, somewhat responsive; second-degree burns; bleeding of major vessel). 3. Moderately severe physical damage; medical hospitalization and likely intensive care required (e.g., conatose with reflexes intact; third-degree burns less than 20% of body; extensive blood loss but can recover; major fractures). 4. Severe physical damage; medical hospitalization with intensive care required (e.g., comatose without reflexes; third-degree burns over 20% of body; extensive blood loss with unstable vital signs; major damage to a vital area). 5. Death Potential Lethality: Only Answer if Actual Lethality=0 Likely lethality of actual attempt if no medical damage (the following examples, while having no actual medical damage, had potential for very serious lethality: put gun in mouth and pulled the trigger but gun fails to fire so no medical damage; laying on train tracks with oncoming train but pulled away before run over). 6. Behavior likely to result in injury 1 = Behavior likely to result in injury 1 = Behavior likely to result in death despite available medical care Enter Code | Answer for Actual Attempts Only | Attempt | |
| Minor physical damage; medical attention needed (e.g., conscious but sleepy, somewhat responsive; second-degree burns; bleeding of major vessel). Moderately severe physical damage; medical hospitalization and likely intensive care required (e.g., comatose with reflexes intact; third-degree burns less than 20% of body; extensive blood loss but can recover; major fractures). Severe physical damage; medical hospitalization with intensive care required (e.g., comatose with reflexes intact; third-degree burns over 20% of body; extensive blood loss with unstable vital signs; major damage to a vital area). Death Potential Lethality: Only Answer if Actual Lethality=0 Likely lethality of actual attempt if no medical damage (the following examples, while having no actual medical damage, had potential for very serious lethality; put gun in mouth and pulled the trigger but gun fails to fire so no medical damage, laying on train tracks with oncoming train but pulled away before run over). Behavior not likely to result in injury Behavior not likely to result in injury but not likely to cause death Behavior likely to result in death despite available medical care | | | Code |
| 2. Moderate physical damage; medical attention needed (e.g., conscious but sleepy, somewhat responsive; second-degree burns; bleeding of major vessel). 3. Moderately severe physical damage; medical hospitalization and likely intensive care required (e.g., comatose with reflexes intact; third-degree burns less than 20% of body; extensive blood loss but can recover; major fractures). 4. Severe physical damage; medical hospitalization with intensive care required (e.g., comatose without reflexes; third-degree burns over 20% of body; extensive blood loss with unstable vital signs; major damage to a vital area). 5. Death Potential Lethality: Only Answer if Actual Lethality=0 Likely lethality of actual attempt if no medical damage (the following examples, while having no actual medical damage, had potential for very serious lethality; put gun in mouth and pulled the trigger but gun fails to fire so no medical damage; laying on train tracks with oncoming train but pulled away before run over). 0 = Behavior not likely to result in injury 1 = Behavior likely to result in injury but not likely to cause death 2 = Behavior likely to result in death despite available medical care | | | |
| 3. Moderately severe physical damage; medical hospitalization and likely intensive care required (e.g., comatose with reflexes intact; third-degree bums less than 20% of body; extensive blood loss but can recover; major fractures). 4. Severe physical damage; medical hospitalization with intensive care required (e.g., comatose without reflexes; third-degree bums over 20% of body; extensive blood loss with unstable vital signs; major damage to a vital area). 5. Death Potential Lethality: Only Answer if Actual Lethality=0 Likely lethality of actual attempt if no medical damage (the following examples, while having no actual medical damage, had potential for very serious lethality: put gun in mouth and pulled the trigger but gun fails to fire so no medical damage; laying on train tracks with oncoming train but pulled away before run over). 6. Behavior likely to result in injury 1 = Behavior likely to result in injury but not likely to cause death 2 = Behavior likely to result in death despite available medical care | | | |
| 4. Severe physical damage; medical hospitalization with intensive care required (e.g., comatose without reflexes; third-degree burns over 20% of body; extensive blood loss with unstable vital signs; major damage to a vital area). 5. Death Potential Lethality: Only Answer if Actual Lethality=0 Likely lethality put gun in mouth and pulled the trigger but gun fails to fire so no medical damage; laying on train tracks with oncoming train but pulled away before run over). 6. Behavior not likely to result in injury 1. Behavior likely to result in injury but not likely to cause death 2. Behavior likely to result in death despite available medical care | | l | |
| extensive blood loss with unstable vital signs; major damage to a vital area). 5. Death Potential Lethality: Only Answer if Actual Lethality=0 Likely lethality of actual attempt if no medical damage (the following examples, while having no actual medical damage, had potential for very serious lethality: put gun in mouth and pulled the trigger but gun fails to fire so no medical damage; laying on train tracks with oncoming train but pulled away before run over). 0 = Behavior likely to result in injury 1 = Behavior likely to result in injury but not likely to cause death 2 = Behavior likely to result in death despite available medical care | | | |
| 5. Death Potential Lethality: Only Answer if Actual Lethality=0 Likely lethality of actual attempt if no medical damage (the following examples, while having no actual medical damage, had potential for very serious lethality: put gun in mouth and pulled the trigger but gun fails to fire so no medical damage, laying on train tracks with oncoming train but pulled away before run over). 0 = Behavior not likely to result in injury but not likely to cause death 1 = Behavior likely to result in death despite available medical care | extensive blood loss with unstable vital signs; major damage to a vital area). | l | |
| Likely lethality of actual attempt if no medical damage (the following examples, while having no actual medical damage, had potential for very serious lethality: put gun in mouth and pulled the trigger but gun fails to fire so no medical damage; laying on train tracks with oncoming train but pulled away before run over). 0 = Behavior not likely to result in injury 1 = Behavior likely to result in injury but not likely to cause death 2 = Behavior likely to result in death despite available medical care | 5. Death | <u> </u> | |
| lethality: put gun in mouth and pulled the trigger but gun fails to fire so no medical damage; laying on train tracks with oncoming train but pulled away before run over). 0 = Behavior not likely to result in injury 1 = Behavior likely to result in injury but not likely to cause death 2 = Behavior likely to result in death despite available medical care | | Enter | r Code |
| before run over). 0 = Behavior net likely to result in injury 1 = Behavior likely to result in injury but not likely to cause death 2 = Behavior likely to result in death despite available medical care | | l | |
| 1 = Behavior likely to result in injury but not likely to cause death 2 = Behavior likely to result in death despite available medical care | | | |
| 1 = Behavior likely to result in injury but not likely to cause death 2 = Behavior likely to result in death despite available medical care | 0 = Behavior not likely to result in injury | | |
| | 1 = Behavior likely to result in injury but not likely to cause death | - | |
| © 2008 Research Foundation for Mental Hygiene, Inc. C-SSRS—Since Last Visit (Version 1/14/09) Page 2 of 2 | | Page | 2 of 2 |

### APPENDIX P. PARKINSON'S DISEASE DIARY

#### PARKINSON'S DISEASE DIARY, IPX203-B16-02

#### INSTRUCTIONS FOR COMPLETING PARKINSON'S DISEASE DIARY

For each half-hour time period place <u>one</u> check mark to indicate your predominant states during most of that period.

ON = Time when medication is providing benefit with regard to mobility, slowness, and stiffness.

OFF = Time when medication has worn off and is no longer providing benefit with regard to mobility, slowness, and stiffness.

**Dyskinesia** = Involuntary twisting, turning movements. These movements are an effect of medication and occur during ON time.

Non-troublesome dyskinesia does not interfere with function or cause meaningful discomfort.

Troublesome dyskinesia interferes with function or causes meaningful discomfort.

Tremor is shaking back and forth and is not considered dyskinesia.

| Table of Contents | |
|-----------------------------------------------------|--------|
| Parkinson's Disease Diary for First 24-hour Period | Page 2 |
| Parkinson's Disease Diary for Second 24-hour Period | Page 3 |
| Parkinson's Disease Diary for Third 24-hour Period | Page 4 |

#### EXAMPLE OF DIARY COMPLETION

| Time | Asleep | OFF | ON without dyskinesia | ON with <u>non</u> -<br>troublesome<br>dyskinesia | ON with troublesome dyskinesia |
|---|---|---|---|---|---|
| 6:00 AM | <b>√</b> | | | | |
| :30 | V | V | | | |
| 7:00 AM | | V | | | |
| :30 | | V | | | |
| 8:00 AM | | | | | |
| :30 | | V | | | V |
| 9:00 AM | | | V | | |

| Correct |
|-----------|
| Incorrect |
| Correct |
| Correct |
| Incorrect |
| Incorrect |
| Correct |

#### Start Date DD-MMM-YYYY:

Instructions: For each half-hour time period place one check mark to indicate your predominant status during most of that period.

ON = Time when medication is providing benefit with regard to mobility, slowness, and stiffness.

OFF = Time when medication is not providing benefit with regard to mobility, slowness, and stiffness

Dyskinesia = Involuntary twisting, turning movements. These movements are an effect of medication and occur during ON time.

Non-troublesome dyskinesia does not interfere with function or cause meaningful discomfort.

Troublesome dyskinesia interferes with function or causes meaningful discomfort.

Tremor is shaking back and forth and is not considered dyskinesia.

| t | ime | asleep | OFF | ON<br>without<br>dyskinesia | ON with non- troublesome dyskinesia | ON with troublesome dyskinesia |
|---|---|---|---|---|---|---|
| 6:0 | MA OO | | | | , | |
| | :30 | | | | | |
| 7:0 | MA OC | | | | | |
| | :30 | | | | | |
| 8:0 | MA OC | | | | | |
| | :30 | | | | | |
| 9:0 | MA OC | | | | | |
| | :30 | | | | | |
| 10: | 00 AM | | | | | |
| | :30 | | | | | |
| 11: | 00 AM | | | | | |
| | :30 | | | | | |
| 12: | 00 PM | | | | | |
| | :30 | | | | | |
| 1:0 | 00 PM | | | | | |
| | :30 | | | | | |
| 2:0 | M9 00 | | | | | |
| | :30 | | | | | |
| 3:0 | 00 PM | | | | | |
| | :30 | | | | | |
| 4:0 | 00 PM | | | | | |
| | :30 | | | | | |
| 5:0 | M9 OC | | | | | |
| | :30 | | | | | |

| time | asleep | OFF | ON<br>without<br>dyskinesia | ON with<br>non-<br>troublesome<br>dyskinesia | ON with troublesome dyskinesia |
|---|---|---|---|---|---|
| 6:00 PM | | | | | |
| :30 | | | | | |
| 7:00 PM | | | | | |
| :30 | | | | | |
| 8:00 PM | | | | | |
| :30 | | | | | |
| 9:00 PM | | | | | |
| :30 | | | | | |
| 10:00 PM | | | | | |
| :30 | | | | | |
| 11:00 PM | | | | | |
| :30 | | | | | |
| 12:00 AM | | | | | |
| :30 | | | | | |
| 1:00 AM | | | | | |
| :30 | | | | | |
| 2:00 AM | | | | | |
| :30 | | | | | |
| 3:00 AM | | | | | |
| :30 | | | | | |
| 4:00 AM | | | | | |
| :30 | | | | | |
| 5:00 AM | | | | | |
| :30 | | | | | |

Copyright © The University of South Florida, 2000. All rights reserved

Hauser et al. J Clin Neurophar 2000; 23:75-81 Impax\_IPX203-816-02\_PD Diary\_English (US)\_Version 1.2\_14Sep2018


#### Start Date DD-MMM-YYYY:

Instructions: For each half-hour time period place one check mark to indicate your predominant status during most of that period.

ON = Time when medication is providing benefit with regard to mobility, slowness, and stiffness.

OFF = Time when medication is not providing benefit with regard to mobility, slowness, and stiffness

Dyskinesia = Involuntary twisting, turning movements. These movements are an effect of medication and occur during ON time.

Non-troublesome dyskinesia does not interfere with function or cause meaningful discomfort.

Troublesome dyskinesia interferes with function or causes meaningful discomfort.

Tremor is shaking back and forth and is not considered dyskinesia.

| time | asleep | OFF | ON<br>without<br>dyskinesia | ON with ron- troublesome dyskinesia | ON with troublesome dyskinesia |
|---|---|---|---|---|---|
| 6:00 AM | | | | | |
| :30 | | | | | |
| 7:00 AM | | | | | |
| :30 | | | | | |
| 8:00 AM | | | | | |
| :30 | | | | | |
| 9:00 AM | | | | | |
| :30 | | | | | |
| 10:00 AM | | | | | |
| :30 | | | | | |
| 11:00 AM | | | | | |
| :30 | | | | | |
| 12:00 PM | | | | | |
| :30 | | | | | |
| 1:00 PM | | | | | |
| :30 | | | | | |
| 2:00 PM | | | | | |
| :30 | | | | | |
| 3:00 PM | | | | | |
| :30 | | | | | |
| 4:00 PM | | | | | |
| :30 | | | | | |
| 5:00 PM | | | | | |
| :30 | | | | | |

| time | asleep | OFF | ON<br>without<br>dyskinesia | ON with<br>non-<br>troublesome<br>dyskinesia | ON with<br>troublesome<br>dyskinesia |
|---|---|---|---|---|---|
| 6:00 PM | | | | | |
| :30 | | | | | |
| 7:00 PM | | | | | |
| :30 | | | | | |
| 8:00 PM | | | | | |
| :30 | | | | | |
| 9:00 PM | | | | | |
| :30 | | | | | |
| 10:00 PM | | | | | |
| :30 | | | | | |
| 11:00 PM | | | | | |
| :30 | | | | | |
| 12:00 AM | | | | | |
| :30 | | | | | |
| 1:00 AM | | | | | |
| :30 | | | | | |
| 2:00 AM | | | | | |
| :30 | | | | | |
| 3:00 AM | | | | | |
| :30 | | | | | |
| 4:00 AM | | | | | |
| :30 | | | | | |
| 5:00 AM | | | | | |
| :30 | | | | | |

Copyright @ The University of South Florida, 2000. All rights reserved

Hauser et al. J Clin Neurophar 2000; 23:75-81 Impax\_IPX203-B16-02\_PD Diary\_English (US)\_Version 1.2\_14Sep2018


#### Start Date DD-MMM-YYYY:

Instructions: For each half-hour time period place one check mark to indicate your predominant status during most of that period.

**ON =** Time when medication is providing benefit with regard to mobility, slowness, and stiffness.

OFF = Time when medication is not providing benefit with regard to mobility, slowness, and stiffness

Dyskinesia = Involuntary twisting, turning movements. These movements are an effect of medication and occur during ON time.

Non-troublesome dyskinesia does not interfere with function or cause meaningful discomfort.

Troublesome dyskinesia interferes with function or causes meaningful discomfort.

Tremor is shaking back and forth and is not considered dyskinesia.

| timo | asloop | OFF | ON<br>without<br>dyskinesia | ON with<br>non-<br>troublesome<br>dyskinesia | ON with<br>troublesome<br>dyskinesia | timo | asloop | OFF | ON<br>without<br>dyskinesia | ON with<br>non-<br>troublesome<br>dyskinesia | ON with<br>troublesome<br>dyskinesia |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 6:00 AM | | | | | | 6:00 PM | | | | | |
| :30 | | | | | | :30 | | | | | |
| 7:00 AM | | | | | | 7:00 PM | | | | | |
| :30 | | | | | | :30 | | | | | |
| 8:00 AM | | | | | | 8:00 PM | | | | | |
| :30 | | | | | | :30 | | | | | |
| 9:00 AM | | | | | | 9:00 PM | | | | | |
| :30 | | | | | | :30 | | | | | |
| 10:00 AM | | | | | | 10:00 PM | | | | | |
| :30 | | | | | | :30 | | | | | |
| 11:00 AM | | | | | | 11:00 PM | | | | | |
| :30 | | | | | | :30 | | | | | |
| 12:00 PM | | | | | | 12:00 AM | | | | | |
| :30 | | | | | | :30 | | | | | |
| 1:00 PM | | | | | | 1:00 AM | | | | | |
| :30 | | | | | | :30 | | | | | |
| 2:00 PM | | | | | | 2:00 AM | | | | | |
| :30 | | | | | | :30 | | | | | |
| 3:00 PM | | | | | | 3:00 AM | | | | | |
| :30 | | | | | | :30 | | | | | |
| 4:00 PM | | | | | | 4:00 AM | | | | | |
| :30 | | | | | | :30 | | | | | |
| 5:00 PM | | | | | | 5:00 AM | | | | | |
| :30 | | | | | | :30 | | | | | |

Copyright © The University of South Florida, 2000. All rights reserved

Hauser et al. J Clin Neurophar 2000; 23:75-81 |mpax\_IPX203-B16-02\_PD Diary\_English (US)\_Version 1.2\_14Sep2018


# APPENDIX Q. EXCIPIENTS IN IPX203, IPX203 PLACEBO, IR CD-LD, AND IR PLACEBO

| IPX203<br>(Various Strengths) | IPX203 Placebo | IR CD-LD<br>(25-100 mg) | IR Placebo |
|---|---|---|---|
| Microcrystalline Cellulose,<br>NF | Microcrystalline Cellulose,<br>NF | Crospovidone | Microcrystalline cellulose,<br>NF |
| Croscarmellose Sodium, NF | Tale, USP | Hydroxypropyl Cellulose | Magnesium Stearate, NF |
| Magnesium Stearate, NF | Magnesium Stearate, NF | Magnesium Stearate | Quinoline yellow E104 |
| Mannitol, USP | Sugar Spheres, NF | Microcrystalline cellulose | |
| Sodium Lauryl Sulfate, NF | Methacrylic acid copolymer<br>Type A, NF | Starch (corn) | |
| Povidone, USP | Triethyl citrate, NF | D&C Yellow No. 10 | |
| Cellulose Acetate | Hard gelatin capsules | Aluminum Oxide | |
| Copovidone, NF | | | |
| Amino Methacrylate<br>Copolymer, NF | | | |
| Methacrylic acid copolymer<br>Type A, NF | | | |
| Triethyl Citrate, NF | | | |
| Talc, USP | | | |
| Hard gelatin capsules | | | |

### APPENDIX R. CLINICAL LABORATORY STUDIES

HEMATOLOGY

hemoglobin % lymphocytes absolute lymphocytes
hematocrit % monocytes absolute monocytes
red blood cell count % basophils absolute basophils
white blood cell count % eosinophils absolute eosinophils

% neutrophils absolute neutrophils platelet count

**CHEMISTRY** 

sodium calcium indirect bilirubin
potassium phosphorous alkaline phosphatase
chloride albumin alanine aminotransferase

carbon dioxide total protein (ALT, SGPT)

blood urea nitrogen (BUN) uric acid aspartate aminotransferase

creatinine (AST, SGOT)

glucose direct bilirubin creatine phosphokinase lactate dehydrogenase

**URINALYSIS** 

pH ketones leukocyte esterase

specific gravity microscopic exam (RBC protein and WBC, only when

blood indicated)

glucose

URINE DRUG TEST

amphetamines benzodiazepines

barbiturates cannabinoids

cocaine metabolites

opiates

phencyclidines

## ALCOHOL BREATH TEST

## PREGNANCY TEST

Urine pregnancy test (to be completed on site) for female subjects of childbearing potential.